## **Statistical Analysis Plan**

**Official Title of Study:** A randomized, double blind (sponsor open), comparative, multi-center study to evaluate the safety and efficacy of subcutaneous belimumab (GSK1550188) and intravenous rituximab co-administration in subjects with primary Sjögren's syndrome.

**NCT ID:** NCT02631538

**Other Identifiers**: 2015-000400-26

**Date of Document**: 15Sep2020

The GlaxoSmithKline group of companies

201842

| Information Type | : Reporting and Analysis Plan (RAP) |
|------------------|-------------------------------------|

| Title | : | Reporting and Analysis Plan for a randomized, double blind (sponsor open), comparative, multi-center study to evaluate the safety and efficacy of subcutaneous belimumab (GSK1550188) and intravenous rituximab co-administration in subjects with primary Sjögren's syndrome. |
|---|---|---|
| <b>Compound Number</b> | : | GSK1550188 |
| <b>Effective Date</b> | : | 18-AUG-2020 |

#### **Description:**

The purpose of this RAP is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol 201842.

This RAP is intended to describe the planned safety & tolerability, efficacy, biomarker/pharmacodynamic, pharmacokinetic and health outcomes analyses required for the study.

This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverables.

RAP Section 3.3 (Final Analyses) outlined the intended purpose of the RAP was for the planned analyses for Primary and End of Study (EoS) SAC deliverables. However, in the event that the Primary Analysis reporting does not identify treatment benefit, an abridged set of analysis may be conducted for EoS analysis, which will be detailed in a RAP amendment or addendum. Therefore, this RAP amendment includes updates to the approved version for the Primary Analysis. As the milestone (Last Subject Last Visit) for RAP approval as per SOP\_54838 has been achieved, agreement and approval steps allow confirmation of any planned changes outside the steps outlined in the RAP SOP.

#### RAP Author(s)

| Author | Date |
|----------------------------------------------------------|--------------|
| PPD | 23-OCT-2019 |
| Senior Statistician (Immuno-Inflammation, Biostatistics) | 25 001 2017 |
| PPD | 10 ALIC 2020 |
| Statistical Leader (Biostatistics, Development, GSK) | 18-AUG-2020 |
| PPD | 14 CED 2020 |
| Statistical Leader (Biostatistics, Development, GSK) | 14-SEP-2020 |

Copyright 2020 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

2020N437857\_00

The GlaxoSmithKline group of companies

201842

## **RAP Team Review Confirmations**

(Method: E-mail)

| Reviewer | Date |
|--------------------------------------------------------------|-------------|
| Clinical Development Director Immuno-Inflammation, GSK | 23-OCT-2019 |
| PPD Discovery Medicine Group Leader, GSK | 23-OCT-2019 |
| Programming Manager, Immuno-Inflammation, Biostatistics, GSK | 24-OCT-2019 |
| Global Clinical Development Manager, GSK | 23-OCT-2019 |
| Research Manager in Clinical Biomarker Group, GSK | 23-OCT-2019 |
| SERM Physician, Development Global Medical, GSK | 23-OCT-2019 |

## **Clinical Statistics & Clinical Programming Line Approvals**

(Method: Pharma TMF eSignature)

| Approver | Date |
|---------------------------------------------------------------|-------------|
| Statistical Leader, Immuno-Inflammation, Biostatistics, GSK | 25-OCT-2019 |
| Director Programming, Immuno-Inflammation, Biostatistics, GSK | 25-OCT-2019 |

2020N437857\_00

The GlaxoSmithKline group of companies

201842

## **RAP Team Review Confirmations: RAP Addendum**

(Method: E-mail)

| Reviewer | Date |
|---|---|
| Clinical Development Director, Clinical Science Lupus, GSK | 14-SEP-20 |
| Clinical Development Director, Clinical Science (II and Fibrosis), GSK | 14-SEP-20 |
| Programming Manager, Biostatistics, Development, GSK | 14-SEP-20 |
| Global Clinical Development Manager, R&D GCSD, GSK | 14-SEP-20 |
| Clinical Biomarker Director, Group, Clinical Biomarkers One, GSK | 14-SEP-20 |
| SERM Physician, Development Global Medical, GSK | 14-SEP-20 |

# Clinical Statistics & Clinical Programming Line Approvals: RAP Addendum (Method: Pharma TMF eSignature)

| Approver | Date |
|------------------------------------------------------------|-----------|
| Head - Statistics, Biostatistics (India), Development, GSK | 15-SEP-20 |
| PPD | |
| Programming Leader, Biostatistics, Development, GSK | 15-SEP-20 |
| On behalf of PPD (Line Manager, Director Programming, | 13-3E1-20 |
| Biostatistics, Development, GSK) | |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | REPO | ORTING & ANALYSIS PLAN SYNOPSIS | 7 |
| 2. | SLIMI | MARY OF KEY PROTOCOL INFORMATION | 10 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | Changes to the Final RAP for End of Study Reporting | |
| | 2.3. | Study Objective(s) and Endpoint(s) | |
| | 2.4. | Study Design | |
| | 2.4. | Statistical Hypotheses | |
| | 2.5. | Statistical Hypotheses | 10 |
| 3. | | INED ANALYSES | |
| | 3.1. | Regular Data Reviews | 15 |
| | 3.2. | Interim Analyses | 16 |
| | 3.3. | Final Analyses | 17 |
| 4. | ANAL | YSIS POPULATIONS | 18 |
| • | 4.1. | Protocol Deviations | |
| | 4.2. | Per-Protocol Population | |
| | | · | |
| 5. | | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | VENTIONS | 20 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3. | Multi-center Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | 23 |
| | | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | 23 |
| | 5.6. | Other Considerations for Data Analysis and Data Handling | |
| | | Conventions | 23 |
| 6. | STUE | DY POPULATION ANALYSES | 24 |
| | 6.1. | Overview of Planned Analyses | 24 |
| | | • | |
| 7. | | ARY STATISTICAL ANALYSES | |
| | 7.1. | Safety Analyses | |
| | | 7.1.1. Overview of Planned Analyses | |
| | | 7.1.2. Immunogenicity | |
| | | 7.1.3. Immunoglobulin | |
| | | 7.1.4. Adverse Events of Special Interest | 28 |
| 8. | SECONDARY STATISTICAL ANALYSES | | |
| | 8.1. | Efficacy and Biomarker Analyses | 31 |
| | | 8.1.1. Overview of Planned Efficacy and Biomarker Analyses | |
| | | 8.1.2. Planned Efficacy and Biomarker Statistical Analyses | |
| | 8.2. | Pharmacokinetic Analyses | |
| | | 8.2.1. Overview of Planned Pharmacokinetic Analyses | |
| | | 8.2.2. Drug Concentration Measures | |
| | 8.3. | Pharmacokinetic / Pharmacodynamic Analyses | |

| 9. | OTHE | | TICAL ANALYSES | |
|---|---|---|---|---|
| | 9.1. | Explorato | ory | |
| | | 9.1.1. | Overview of Exploratory Analysis | 39 |
| | | 9.1.2. | Planned Exploratory Analyses | |
| | 9.2. | | utcomes | |
| | | 9.2.1. | Overview of Health Outcome Analysis | |
| | | 9.2.2. | Planned Health Outcomes Statistical Analyses | |
| | | 9.2.3. | Planned Health Outcomes Psychometric Analyses | 45 |
| 10. | REFE | RENCES | | 46 |
| 11. | APPEI | NDICES | | 47 |
| | 11.1. | <b>Appendix</b> | 1: Protocol Deviation Management and Definitions for Per | |
| | | Protocol | Population | |
| | | 11.1.1. | Exclusions from Per-Protocol Population | 47 |
| | 11.2. | <b>Appendix</b> | 2: Schedule of Activities | 49 |
| | | 11.2.1. | Protocol Defined Schedule of Events | 49 |
| | 11.3. | <b>Appendix</b> | 3: Treatment States and Phases | 53 |
| | | 11.3.1. | Treatment Phases | 53 |
| | | 11.3.2. | Treatment States | 53 |
| | 11.4. | <b>Appendix</b> | 4: Data Display Standards & Handling Conventions | 54 |
| | | | Reporting Process & Standards | |
| | 11.5. | <b>Appendix</b> | 5: Derived and Transformed Data | 56 |
| | | 11.5.1. | General | 56 |
| | | 11.5.2. | Study Population | 59 |
| | | 11.5.3. | Safety | 60 |
| | | 11.5.4. | Efficacy | 71 |
| | | 11.5.5. | Health Outcomes | |
| | | 11.5.6. | Biomarkers | |
| | 11.6. | | 6: Reporting Standards for Missing Data | |
| | | 11.6.1. | Premature Withdrawals | |
| | | 11.6.2. | Handling of Missing Data | |
| | 11.7. | | 7: Values of Potential Clinical Importance | |
| | | 11.7.1. | Laboratory Values | |
| | | 11.7.2. | Vital Signs | 86 |
| | 11.8. | | 8: Laboratory Parameters & Toxicity Grading Tables | |
| | | | Laboratory Parameters | |
| | | | Toxicity Grading Tables | 89 |
| | 11.9. | | 9: Model Checking and Diagnostics for Statistical | |
| | | Analyses | | 92 |
| | | | Statistical Analysis Assumptions | |
| | | | (10 – Abbreviations & Trade Marks | |
| | 11.11. | | (11: Questionnaires | 97 |
| | | 11.11.1. | Columbia Suicide severity rate scale (CSSRS) post | 0.7 |
| | | 44.44.0 | baseline | |
| | | | Columbia Suicide severity rate scale (CSSRS) at baseline | |
| | | | Eular Sjögren's syndrome disease activity index (ESSDAI) | |
| | | | Neurological Symptoms | |
| | | | Oral and Ocular dryness | |
| | | 11.11.6. | Physician global assessment of disease activity (PGA) | 116 |
| | | 11.11.7. | Eular Sjögren's syndrome patient reported index | 447 |
| | | | (ESSPRI) | 117 |

2020N437857\_00

| 201842 |
|--------|
|--------|

| | 11.11.8. | Profile of fatigue and discomfort - SICCA symptoms | |
|---|---|---|---|
| | | inventory short form (PROFAD-SSI-SF) | |
| | | Patient global assessment of disease activity (PtGA) | |
| | 11.11.10. | .Sjogren's Allowable Medication Categories | 121 |
| | 11.11.11. | Prednisone Conversion Factors | 123 |
| | | Exit Interview | |
| 11.12. | <b>Appendix</b> | (12: Headline Results | 129 |
| | 11.12.1. | Headline Results Output | 129 |
| 11.13. | <b>Appendix</b> | (13: List of Data Displays | 130 |
| | 11.13.1. | Data Display Numbering | 130 |
| | 11.13.2. | Mock Example Shell Referencing | 131 |
| | 11.13.3. | Deliverables | 131 |
| | 11.13.4. | Study Population Tables | 132 |
| | 11.13.5. | Efficacy Tables | 135 |
| | 11.13.6. | Efficacy Figures | 142 |
| | 11.13.7. | Safety Tables | 146 |
| | 11.13.8. | Safety Figures | 156 |
| | 11.13.9. | Pharmacokinetic Tables | 157 |
| | 11.13.10. | .Pharmacokinetic Figures | 158 |
| | 11.13.11. | .Pharmacokinetic / Pharmacodynamic Figures | 159 |
| | 11.13.12. | .Health Outcomes Tables | 160 |
| | 11.13.13. | .Health Outcomes Figures | 164 |
| | 11.13.14. | Exploratory Tables | 165 |
| | 11.13.15. | Exploratory Figures | 172 |
| | | ICH Listings | |
| | 11.13.17. | Non-ICH Listings | 180 |
| 11.14. | <b>Appendix</b> | ( 14: Example Mock Ups | 184 |

## 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | This RAP details all planned analyses and outputs required for: |
| | Primary Analyses (post completion of all week 52 assessments) |
| | 2. End of Study (EoS) Analyses (Week 104) |
| Protocol | This RAP is based on the protocol amendment 06 (Dated 25/Jun/2019) of study 201842 (GSK Document Number 2014N220285_06 and eCRF Version 1.02). |
| Primary<br>Objective | <ul> <li>Investigate the safety and tolerability of anti-BLyS / anti-CD20 co-<br/>administration therapy and anti-BLyS and anti-CD20 monotherapies for<br/>subjects with active primary Sjögren's syndrome (pSS).</li> </ul> |
| Primary<br>Endpoint | Safety and tolerability; including incidence of SAEs and AESIs. |
| Study<br>Design | A randomized, double blind (sponsor open), comparative, multi-national, multi-center, placebo-controlled trial in subjects with active pSS. |
| | <ul> <li>Approximately 70 subjects will be recruited into the study initially. At Day 0, subjects will be randomized 1:2:2:2 into one of 4 treatment arms.</li> <li>Withdrawals may be replaced.</li> </ul> |
| | Study 201842 consisted of 3 phases: |
| | <ul> <li>A 52-week treatment phase during which subjects were randomized to<br/>one of four arms</li> </ul> |
| | <ul> <li>A 16-week general follow (GFU) up period focused on safety<br/>assessments</li> </ul> |
| | <ul> <li>An individualized follow (IFU) up period for subjects with persistently<br/>low B cell counts</li> </ul> |
| | NOTE: All subjects will enter a 16-week general follow-up period after the Week 52 visit or after discontinuation if a subject discontinues IP and withdraws from the treatment phase visits prior to Week 52. Assessments to be performed are included in protocol Time and Events Table. During the general follow up period subjects will remain off of investigational product, endeavor not to change concomitant medication regimen, receive monthly safety follow up phone calls, and will return to the clinic for asite visit at the end of the general follow up period |
| | Subjects entering IFU are assessed every 12 wks (± 7 days), with calls every 4 wks (±7 days) between visits. Subjects exit IFU when: CD19+ B-lymphocyte counts are within normal range or 10% of baseline levels (if baseline < LLN), OR at investigator's discretion starts receiving disease modifying therapy that may affect B-cell numbers OR for up to a maximum of 2 years (i.e., up to Week 104) – whichever comes first. Subjects exiting IFU period will attend a |

| Overview | Key Elements of the RAP |
|---|---|
| | final visit (within 28 days of decision) for final assessments (IFU Final Visit). |
| | Subjects who withdrew (WD) prematurely from investigational product (IP) during treatment phase & refused to attend further visits through wk 52, were encouraged to participate in the GFU & IFU for safety purposes. |
| Planned<br>Analyses | <ul> <li>Quarterly blinded safety data summaries for SRT.</li> <li>Quarterly un-blinded safety data summaries and secondary efficacy endpoint, ESSDAI for iSRC.</li> <li>Interim analyses occurring once approximately 35 subjects have completed their Week 24 assessments.</li> <li>Primary Analysis <ul> <li>The primary analyses will be conducted following completion of all Week 52 visits, with inclusion of the FU visit data which is available at this time. The analyses will be performed once the data from all visits up to and including this Week 52 cutoff have been collected, verified and validated. Week 68 data will also be included, if available.</li> </ul> </li> <li>End of Study <ul> <li>The follow-up (end of study) analyses will include all follow-up data (i.e. general follow-up data between Week 52 and Week 68 and individualized follow-up data from Week 68 through Week 104/IFU final visit). These analyses will be performed once data from Week 52 through Week 104/IFU final visit has been collected, verified and validated.</li> </ul> </li> </ul> |
| Analysis<br>Populations | <ul> <li>'Screened Population' will be used to evaluate selected study population.</li> <li>'Enrolled Population' will be used to evaluate selected study population.</li> <li>'Safety Population' will be used to evaluate study population, efficacy, safety, PD, exploratory and health outcomes data.</li> <li>'PK' populations will be used to evaluate belimumab and rituximab pharmacokinetics.</li> <li>'Per-protocol Population' may be used to evaluate a subset of Efficacy, PD, and biomarker data.</li> </ul> |
| Hypothesis | <ul> <li>The study is designed to investigate the safety and tolerability of the coadministration of belimumab with rituximab and belimumab monotherapy in subjects with pSS.</li> <li>No formal hypotheses will be tested.</li> <li>For secondary endpoints, an estimation approach will be adopted with derivation of estimates and 95% confidence interval (CI) for the comparisons of interest (see Section 2.5)</li> </ul> |
| Primary<br>Endpoint<br>Analysis | Safety data will be presented in a tabular and graphical format. |
| | Clinical interpretation will be based upon review of AEs, laboratory values and vital signs. |
| | No formal statistical testing will be performed on the safety data. |
| Secondary | Secondary endpoints will be analysed to provide point estimates and |

2020N437857\_00 201842

| Overview | Key Elements of the RAP |
|---|---|
| Endpoints | corresponding 95% CIs for the comparisons of interest. |
| Analysis | <ul> <li>In addition, probabilities of success of the co-administration therapy and<br/>belimumab monotherapy will be conducted.</li> </ul> |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the planned statistical analysis specified in the protocol amendment 06 [(Dated: 25/Jun/2019)].

Changes from the originally planned statistical analysis specified in the protocol are outlined:

| Protocol | Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| Section 9.3.1: Analysis Population | Section 4: Analysis Populations | <ul> <li>"Screened" and "Enrolled" populations<br/>were included to support data disclosure<br/>displays</li> <li>Per Protocol analysis population was also<br/>defined for sensitivity analysis</li> </ul> |
| Section 9.4.2 Primary<br>Analyses | Section 8.1.1.1 ESSDAI | A corrected ESSDAI score will also be calculated. ESSDAI scores disease activity in 12 domains. In 5 (renal, PNS, CNS, cutaneous and pulmonary) of the domains, ESSDAI requires that if activity has been present for greater than or equal to 12 months then it must be treated as irreversible damage and the activity should be scored as zero (Seror, 2015a). This is a problem for clinical trials of long duration such as study 201842 because it can result in misleading evidence of reduced activity. |

All data displays (Tables, Figures & Listings) will use the term "Subject" which reflects CDISC and GSK Data Display Standards terminology.

## 2.2. Changes to the Final RAP for End of Study Reporting

This section outlines key (not limited too) updates from the RAP version approved prior to the RAP SOP milestone (Last Subject Last Visit).

Additional updates post EoS Database Release (DBR) have also been included to clarify timepoints included for the general follow up period and individualised follow up period. Subjects who withdrew (WD) prematurely from investigational product (IP) during the treatment phase and refused to attend further visits through week 52, were encouraged to participate in the GFU period and the IFU period (if required) for safety purposes. For several subjects withdrawing early from IP, this resulted in a temporal misalignment of data such that data which were collected during their follow up calls and visits were allocated to visits which occurred much later in the study (i.e. in the post W52 general and individualized follow up periods). Additional analyses have been included to assess the response in the GFU and IFU.

| RAP Section | Summary of Change |
|---|---|
| 4.0 Study Population | |
| | 68/FU / IFU analyses. |
| 7.1 Safety Analyses | Primary Analysis: Implemented MedDRA V22.0. |
| 11.5.3 Safety | <b>EoS Analysis:</b> Implement MedDRA V23.0 which constitutes a major release and |
| Appendix 13: List of | relevant sections are updated. |
| Data Displays | Primary Analysis: Summarized safety data for all completed visits up to W68 |
| Bata Bioplayo | (where reported by visit) and up to W104 (where not reported by visit), with cut-off |
| | date of 09/09/19 (W52 LSLV). |
| | <b>EoS Analysis:</b> Will summarize (Tables, Figures and Listings) AE/AESI safety |
| | endpoints for all completed visits <u>up to Week 68 only.</u> Other safety endpoints will |
| 744 4 1 | be reported using scheduled visits, unless specified. |
| 7.1.4. Adverse | <b>EoS Analysis:</b> Specified additional AESI details for post-administration systemic |
| Events of Special | reactions by Rituximab/Placebo Infusion. |
| Interest | |
| 8. Secondary | <b>Primary Analysis:</b> Specified any formal model based statistical analyses included |
| Statistical Analyses | visits upto Week 52. |
| 9. Other Statistical | <b>EoS Analysis:</b> Additional ESSDAI statistical analyses included using the completer |
| Analyses | population. |
| Appendix 13: List of | |
| Data Displays | Driver Analysis (/ sharps from booting in No. of D.O. II. (ODOO)/r. O. |
| 8. Secondary | Primary Analysis: % change from baseline in No. of B Cells (CD20)/mm2 in |
| Statistical Analyses | salivary gland biopsy at Week 24 was reported. |
| Appendix 13: List of | <b>EoS Analysis:</b> Change from baseline will be reported instead of % change from |
| Data Displays | baseline. |
| 11.5.3 Appendices: | <b>EoS Analysis:</b> Added Section 11.5.3.2. Coronavirus Disease 2019 (COVID-19) |
| Safety | Environment Onset Date. |
| 11.5.6 Biomarker | <b>EoS Analysis:</b> Table 11 (Flow Cytometry Parameters) & Table 13 (Minor Salivary |
| Appendix 13: List of | Gland Parameters) updated to reflect final EoS delivery. Additional details included |
| Data Displays | for imputation of Flow Cytometry Parameters. |
| 11.8.1 Laboratory | |
| Parameters | FaC Analysia, Additional datable have been included to classify the proportion of |
| 11.5.6.1. | <b>EoS Analysis:</b> Additional details have been included to clarify the reporting of |
| Immunogenicity | Antibodies to Rituximab |
| Appendix 13: List of | <b>EoS Analysis:</b> Any selected Primary Analysis displays that has been identified for |
| Data Displays | generation for EoS has been allocated unique numbering. |
| | <b>EoS Analysis:</b> All figures will be displayed up to Week 68/FU only and a line break |
| | after Week 52 will be included, so as to indicate Week 68/FU timepoint is not |
| | sequential for all subjects. |
| | EoS Analysis: The following display will not be generated: |
| | T2.13: ESSDAI and ClinESSDAI Bland-Altman Plot at Week 24 (Corrected) T3.44: Contain Plot of Mile 24 Changes for Table FCCDAI Season of California |
| | T2.14: Scatter Plot of Wk 24 Changes for Total ESSDAI Score vs Salivary Cland B Calls |
| | Gland B Cells |
| | T2.15: Median Free Blys Vs Median CD19+ B cell by Treatment T3.0.0 |
| | T7.3: Summary Statistics: Lacrimal Gland Function (Schirmer's Test) T7.4: Summary Statistics: Lacrimal Gland Function (Schirmer's Test) |
| | T7.4: Summary Statistics of Change from Baseline: Lacrimal Gland Function |
| | (Schirmer's Test) |
| | T7.5: Summary Statistics of PGA |
| | T7.6: Summary Statistics of Change from Baseline: PGA |
| | T2.1009: Summary of Statistical Analysis Results of Change from Baseline: |
| | ESSDAI Total Score (Uncorrected) |

| RAP Section | Summary of Change |
|---|---|
| | T2.1010: Summary of Statistical Analysis Results of Change from Baseline: |
| | ESSDAI Total Score (Uncorrected) – Per Protocol Population |
| | T2.1011: Summary of Statistical Analysis Results of Change from Baseline: |
| | ESSDAI Total Score (Corrected) |
| | T2.1012: Summary of Statistical Analysis Results of Change from Baseline: |
| | ESSDAI Total Score (Corrected) - Per Protocol Population |
| | T2.1021: Summary of Statistical Analysis of Responder on Total ESSDAl Score (Corrected) |
| | • F2.1005: Adjusted Mean (95% CI) Change from Baseline: ESSDAI Total Score |
| | (Uncorrected) |
| | • F2.1006: Adjusted Mean (95% CI) Change from Baseline: ESSDAI Total Score (Corrected) |
| | T2.1029: Summary of Statistical Analysis Results of Change from Baseline: Stimulated Salivary Flow |
| | T2.1030: Summary of Statistical Analysis Results of Change from Baseline: |
| | Stimulated Salivary Flow - Per Protocol Population |
| | T2.1033: Summary of Statistical Analysis Results of Change from Baseline: |
| | Oral Dryness Numeric Response Scale |
| | T2.1034: Summary of Statistical Analysis Results of Change from Baseline: |
| | Oral Dryness Numeric Response Scale - Per Protocol Population |
| | T6.1006: Summary of Statistical Analysis of Responders on ESSPRI |
| | EoS Analysis: The following additional displays will be generated: |
| | Table 1.1006 Summary of Study Populations |
| | T1.1023: Summary of Overall Subject Status |
| | T.1.1025: Serious Acute Post-Injection Systemic Reactions per GSK |
| | Adjudication by PT, in First Six Doses of Belimumab/Placebo |
| | T.3.63: Post-IV Systemic Reactions per Anaphylactic Reactions CMQ Broad search by PT, in First Two 2 Infusions of Rituximab/Placebo |
| | T2.1040: Summary Statistics of ESSDAI Total Score (Corrected) - Completers |
| | T2.1041: Summary of Statistical Analysis Results of Change from Baseline: |
| | ESSDAI Total Score (Corrected) - Completers |
| | <ul> <li>T2.1042: Summary Statistics of Stimulated and Unstimulated Salivary Flow -<br/>Completers</li> </ul> |
| | T2.1043: Summary Statistics of Oral Dryness Numeric Response Scale - |
| | Completers |
| | T6.1015: Summary Statistics of ESSPRI Total Score and Domains - |
| | Completers |
| | T7.023: Summary Statistics of Flow Cytometry Flow Parameters- Completers I 1050: Listing of Overall Subject Status |
| | L1059: Listing of Overall Subject Status L1061: Listing of Protocol Devictions Related to Covid 10. |
| | L1061: Listing of Protocol Deviations Related to Covid-19 |

## 2.3. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary | |
| Safety and tolerability of anti-BLyS / anti-CD20 co-administration therapy and anti-BLyS and anti- CD20 monotherapies | <ul> <li>Safety and tolerability; including incidence of SAEs<br/>and AESIs.</li> </ul> |
| Secondary | |
| Clinical efficacy of anti-BLyS / anti-<br>CD20 co-administration therapy<br>and anti-BLyS and anti-CD20<br>monotherapies | <ul> <li>ESSDAI score over time</li> <li>Stimulated salivary flow over time</li> <li>Oral dryness numeric response scale over time</li> </ul> |
| Assessment of anti-BLyS / anti-<br>CD20 co-administration therapy<br>and anti-BLyS and anti-CD20<br>monotherapies on tissue B-cells. | B cell quantification within salivary gland biopsy at<br>Week 24 |
| Exploratory | |
| Assessment of mechanism and durability of effect of anti-BLyS/anti-CD20 co-administration therapy and anti-BLyS and anti-CD20 monotherapies. | <ul> <li>Clinical efficacy</li> <li>Ocular dryness numeric response scale over time</li> <li>Lacrimal gland function as measured by Schirmer's test</li> <li>Physician's Global Assessment (PGA) of disease activity over time</li> <li>Biomarkers</li> <li>Serologic markers over time</li> <li>Change in peripheral blood leukocytes including B cell subsets over time</li> <li>BLyS levels in blood</li> <li>Immunogenicity of rituximab and belimumab</li> <li>Pharmacokinetics of rituximab and belimumab</li> <li>Change from baseline in the cellular composition of the salivary gland</li> <li>Sustained efficacy of anti-BLyS/anti-CD20 coadministration at Week 52. Additional exploratory biomarkers may be evaluated [1]</li> <li>Transcriptomic analysis of blood and salivary gland</li> <li>B and T cell receptor clonal analysis in peripheral blood and salivary gland</li> <li>Proteomic assessment of the saliva</li> </ul> |
| Health Outcomes | <u></u> |
| Gather preliminary information on patient reported outcomes of anti-BLyS/anti-CD20 co-administration | <ul> <li>ESSPRI score (and individual scale sub-scores) over time</li> <li>Fatigue and Discomfort- SICCA Symptom Inventory</li> </ul> |

| Objectives | Endpoints |
|---|---|
| therapy and anti-BLyS and anti-CD20 | (PROFAD SSI SF) over time |
| monotherapies. | <ul> <li>Patient Global Assessment (PtGA) of disease activity<br/>over time.</li> </ul> |
| | Subject exit interviews. |
| NOTE: | |
| [1] Analysis will be implemented post week 52 primary analysis | |

## 2.4. Study Design



| Overview of Study Design and Key Features | |
|---|---|
| Interim | Formal planned interim analysis was performed once approximately 35 |
| Analysis | subjects had completed their Week 24 assessments. |

## 2.5. Statistical Hypotheses

The primary objective of the study is to investigate the safety and tolerability of the coadministration of belimumab with rituximab and belimumab monotherapy in subjects with pSS. No formal statistical comparisons will be conducted to assess this objective.

Secondary efficacy and mechanistic endpoints will be investigated. The following exploratory comparisons will be conducted:

- 1. Co-administration belimumab/rituximab treatment arm vs. Placebo arm
- 2. Co-administration belimumab/rituximab treatment arm vs. Rituximab monotherapy arm
- 3. Co-administration belimumab/rituximab treatment arm vs. Belimumab monotherapy arm
- 4. Belimumab monotherapy arm vs. Placebo arm
- 5. Belimumab monotherapy arm vs. Rituximab monotherapy arm

#### 3. PLANNED ANALYSES

## 3.1. Regular Data Reviews

Safety data will be reviewed on a quarterly basis in a blinded fashion by an internal safety review team (SRT). Summaries will be produced in order to describe the baseline demography and the following safety parameters:

- 1. Adverse events and serious adverse events including fatalities
- 2. Adverse events of special interest as defined in the belimumab PSAP
- 3. Withdrawals and reasons for withdrawal
- 4. Blood chemistry
- 5. Hematology
- 6. CD4 and CD8 as measured by flow cytometry
- 7. Immunoglobulin levels (IgG)

The displays for the SRT meetings will not include any laboratory data that could potentially un-blind the treatments. IgA, IgM and CD19 assessment are excluded.

Additionally, summaries of the above parameters plus IgA, IgM, vital signs and ESSDAI will be reviewed in an unblinded manner by the internal Safety Review Committee (iSRC) as outlined in protocol and in the iSRC charter. In order to protect the blinding status, these displays will be produced by a third party (Quanticate).

## 3.2. Interim Analyses

A formal interim analysis was planned to take place once half of the planned subjects (i.e.: approximately 35 subjects) have completed their Week 24 assessments. The interim analysis displays included the available data for all visits up to Week 68 as indicated in the table below. The interim analysis reviewed safety outputs produced for iSRC and additional summaries for efficacy, biomarkers and health outcomes parameters. The interim analysis summaries were produced by treatment group and reviewed by the TA-DAC and the iSRC. At the interim analysis, to aid internal decision making, predictive probabilities for ESSDAI effects were computed for comparison of combination (belimumab/rituximab) vs placebo at Week 24 and for comparison of belimumab monotherapy vs placebo at Week 24. The predictive probabilities for ESSDAI treatment differences greater than 3 and greater than 5, under varying assumptions for target sample size were assessed to support potential sample size re-estimation for the study. Access to interim outputs were restricted to individuals specified in the iSRC charter. There were no changes made to the sample size/study as a result of the interim analysis.

| Section | Interim Analysis |
|---|---|
| Study Population | Baseline demography |
| | Disease History |
| | Disposition |
| Safety | Adverse events and serious adverse events |
| (Primary study | Adverse events of special interest as defined in Belimumab PSAP |
| objective) | Withdrawals and reasons for withdrawal |
| | Immunoglobulin (IgG, IgA, IgM) |
| | Haematology |
| | Blood chemistry |
| | Vital Signs |
| | CD4 and CD8 |
| Clinical Efficacy | ESSDAI Total Score and Domains |
| Biomarkers | B cells (CD20) count/mm² in salivary gland biopsy (by histology) |
| | B cell (CD20) / T cell (CD3) ratio in salivary gland biopsy (by histology) |
| | Lymphocyte Focus Score (expressed per 4mm²) in salivary gland biopsy (by histology) |
| | Plasma cells (CD138+; both CD20pos and CD20neg) count/mm² in salivary gland tissue (by histology). |
| | Frequency of B cells <sup>1</sup> , naïve <sup>2</sup> , memory <sup>3</sup> , and plasmablast <sup>4</sup> in peripheral blood (by flow cytometry) |
| | Serum SS-A concentration |

| Section | Interim Analysis |
|---|---|
| Health Outcomes | ESSPRI (total score and the pain, fatigue and dryness domains) |

- 1. CD19+ B cells (CD3-CD19+)
- 2. Naïve B cells (CD19+CD20+CD27-)
- 3. Memory B cells (CD19+CD20+CD27+)
- 4. Plasmablast All (CD19+CD27+CD38+)

## 3.3. Final Analyses

There will be two database freezes for this study, corresponding to the Primary Analyses and the End of Study Analyses (Week 104).

## **Primary Analysis**

The cut-off date in the Primary Analysis datasets will be 09-Sep-2019 (i.e. the date the last subject completed their Week 52 visit). Data after 09-Sep-2019 will be removed from the extracted data after DBR based on the algorithms detailed in refer to Appendix 5: Derived and Transformed Data for details. The data cut off will be applied on DMDATA before generating any analysis datasets and outputs.

The primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed their Week 52 (or early withdrawal assessment for subjects withdrawing consent prior to Week 52).
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for un-blinding the randomization codes have been met:
  - AESI adjudication through Week 68/FU assessments.
  - Protocol deviation review as described in Protocol Deviation Management Plan (PDMP) is completed.
  - Exclusions from the per protocol population have been agreed and documented.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.
- 5. Database freeze (DBF) has been declared by Data Management.

All outputs as described in Section 6 to Section 9 of the RAP and detailed in Appendix 13 will be reported for the primary analyses:

- Summary tables reported by visit will include only data collected till Week 68/FU
- Summary tables not reported by visit will include all date collected based on the date-cut date, unless otherwise specified/ required.
- All collected data from the Individualized Follow Up (IFU) period will be listed.

#### **End of Study Analysis**

The end of study (after week 104) analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the 16-week generalized follow-up visit (Week 68) and individualized follow up visit (up to Week 104 or IFU final visit for subjects leaving the IFU prior to W104) or Early Withdrawal visit for those subjects who withdraw from the study prior to the Week 104 visit.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management as described in Steps 2, 3 and 5 above.

For the End of Study Analysis reporting, selected Primary Analysis displays (Appendix 13: List of Data Displays) have been identified and will be generated, using the final data.

The displays will be updated (as required) to capture the additional visits and to reflect the final data. If further details are required, a RAP amendment or addendum will be generated to specify the changes.

This RAP details the planned analysis for both database freezes, with the expectation of an observed treatment benefit being observed following the Primary Analysis. In the event that the Primary Analysis reporting does not identify treatment benefit, an abridged set of analysis may be conducted for the end of study analysis, which will be detailed in a RAP amendment or addendum.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | <ul> <li>Selected Study<br/>Population</li> </ul> |
| Enrolled | <ul> <li>All participants who passed screening and entered the study. Includes Randomized Participants.</li> <li>Note: Screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Selected Study Population |
| Safety | <ul> <li>Comprises all subjects who receive at least one dose of study treatment.</li> <li>This population will be based on the treatment the subject actually received.</li> </ul> | <ul> <li>Study Population</li> <li>Efficacy</li> <li>Safety/tolerability</li> <li>PD/Biomarker</li> <li>Exploratory</li> <li>Health Outcomes</li> </ul> |
| Belimumab<br>Pharmacokinetic<br>(PK-B) | Subjects in the "Safety" population for whom a post<br>treatment belimumab pharmacokinetic sample was<br>obtained and analysed. | Belimumab PK |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Rituximab<br>Pharmacokinetic<br>(PK-R) | Subjects in the "Safety" population for whom a post<br>treatment rituximab pharmacokinetic sample was<br>obtained and analysed | Rituximab PK |
| Per-Protocol (PP) | <ul> <li>All participants in the safety population who comply with the protocol.</li> <li>Protocol deviations that would exclude participants from the PP population are defined in Section 4.1 (Protocol Deviations) and Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population.</li> <li>The Per-Protocol set will not be analysed if this population comprises more than 85% of the safety population.</li> </ul> | Subset of<br>Efficacy/PD/<br>Biomarker |
| Completer | Subjects who completed the 52 Week treatment visits AND general follow up phase of the study including the visit at Week 68 NOTE: Definition as per protocol Section 5.5 Subject and Study Completion Does not include any subjects with a study treatment discontinuation flag. | <ul><li>Efficacy</li><li>Health Outcomes</li><li>PD/Biomarkers</li><li>Exploratory</li></ul> |

#### NOTES:

 Please refer to Appendix 13, List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarized and listed.

Separately, important deviations which result in exclusion from the per-protocol analysis population will also be summarized and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the current Protocol Deviation Management Plan. [Version 007 (18-Sep-2019 or higher)].

- Data related to the Primary Analysis will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which lead to the exclusion from the analyses are captured and categorized on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of the protocol deviations.

All deviations will be discussed and adjudicated as important or not important.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

## 4.2. Per-Protocol Population

Periodic review of the per-protocol population will be conducted during the course of the study, with the final assessment made prior to unblinding the data for Primary Analysis reporting.

The per-protocol population will be primarily based on an assessment of the important protocol deviations. However, non-important deviations or other study conduct issues may be identified during the study and warrant a subject's exclusion from the per-protocol population. This will be documented in the protocol deviation adjudication meeting minutes prior to database freeze. Only protocol deviations or study conduct issues that have the potential to impact a subset of Efficacy/PD/Biomarker evaluations will lead to a subject's exclusion from the per-protocol population.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| RandAll NG Data Displays for Reporting | | | |
| Code | Description | Description | Order [1] |
| Α | Co-administration therapy | Co-administration | 2 |
| В | Belimumab 200 mg SC injection | Belimumab | 3 |
| С | Rituximab 1,000 mg IV infusion | Rituximab | 4 |
| Р | Placebo | Placebo | 1 |

#### NOTES:

## Treatment Descriptors, Colors, Line Style and Symbols for Reporting

| Treatment Descriptor | Color | SAS Color | Line Style | Symbol |
|----------------------|--------|-----------|------------|-------------------|
| Co-administration | Green | CX228B22 | LongDash | Circle (filled) |
| Belimumab | Blue | CX0000FF | Dash | Triangle (filled) |
| Rituximab | Purple | CX800080 | ShortDash | Diamond (filled) |
| Placebo | Brown | CXA05000 | Solid | Square (filled) |

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 0 assessments are assumed to be taken prior to first dose and used as baseline.

| Parameter | Study Asse | essments Considere | Baseline Used in | |
|---|---|---|---|---|
| | Screening | Day 0 (Pre-Dose) | Week 8 | Data Display |
| Safety | | | | |
| Laboratory [1] | Х | Х | | Day 0 (Pre Dose) [3] |
| Vital Signs | Х | Х | | Day 0 (Pre Dose) [3] |
| CSSRS | | Х | | Day 0 (Pre Dose) |
| Neurological Assessment | | Х | | Day 0 (Pre Dose) |
| Immunogenicity (Rituximab) | | | Χ | Week 8 |

| Parameter | Study Asse | Study Assessments Considered as Baseline | | |
|---|---|---|---|---|
| | Screening | Day 0 (Pre-Dose) | Week 8 | Data Display |
| Efficacy | | | | |
| ESSDAI/ClinESSDAI | Х | | | Screening |
| Salivary Flow | Х | | | Screening |
| Oral Dryness | Х | | | Screening |
| Salivary Gland B Cell<br>Quantification | Х | | | Screening |
| Exploratory | | | | |
| Ocular Dryness | Х | | | Screening |
| Lacrimal Gland Function | Х | | | Screening |
| PGA | Х | | | Screening |
| Unstimulated Salivary Flow | Х | | | Screening |
| BLyS | | X | | Day 0 (Pre Dose) |
| Serologic Markers | Х | X | | Day 0 (Pre Dose) [3] |
| Flow Cytometry | Х | Х | | Day 0 (Pre Dose) [3] |
| Minor Salivary Gland<br>Histology Assessments [2] | Х | | | Screening |
| Health Outcomes | | | | |
| ESSPRI | Х | | | Screening |
| PRO FAD SSI SF | Х | | | Screening |
| PtGA | Х | | | Screening |

#### Notes:

- 1. Includes Clinical Chemistry, Hematology, Urinalysis and Other Screening Tests
- 2. Salivary gland biopsy may be conducted at any time during screening up to day 0
- 3. If day 0 pre dose assessment is missing, the screening assessment will be used as baseline.
- Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.
- Unless otherwise stated, if baseline data are missing no derivation will be performed and baseline will be set to missing.

Changes from baseline will be derived as follows.

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 5.2 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 5.3. Multi-center Studies

In this multicenter global study, enrolment will be presented by country and site.

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

Independent variables to be included in efficacy and exploratory analyses are described in Section 8 and Section 9, respectively.

## 5.4.2. Examination of Subgroups

Subgroup analysis based on following Randomization Stratum ESSDAI categories may be analysed as a post SAC analysis.

## ESSDAI groups:

- Low (<5)
- Moderate (>=5 & <=12)
- Severe (>12)
- High Activity (>=14)

## 5.5. Multiple Comparisons and Multiplicity

No adjustments for multiple comparisons are planned.

# 5.6. Other Considerations for Data Analysis and Data Handling Conventions

Other considerations for Data Analysis are described in the appendices;

| Section | Component |
|---------|-------------------------------------------------------------|
| 11.3 | Appendix 3: Treatment States and Phases |
| 11.4 | Appendix 4: Data Display Standards and Handling Conventions |
| 11.5 | Appendix 5: Derived and Transformed Data |
| 11.6 | Appendix 6: Reporting Standards for Missing Data |
| 11.7 | Appendix 7: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Table 1 provides an overview of the planned study population analyses for the primary analyses, and the specific data displays are captured in Appendix 13: List of Data Displays.

Table 1 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| Randomization | | | |
| Randomization and Actual Treatments | | | Υ |
| Subject Disposition | | | T |
| Subject Disposition | Υ [1] | | |
| Reasons for Screening Failures | Υ | | Y |
| Reasons for Withdrawals | Y | | Υ |
| Treatment Discontinuations | | | Y |
| Important Protocol Deviations | Y | | <b>Y</b> [2] |
| Enrolment | Y | | |
| Exclusions from Study Populations | Y | | Y |
| Demographic and Baseline Characteristics | • | | • |
| Demographic Characteristics | Y | | Y |
| Race & Racial Combinations | Y | | Y |
| Smoking Use | Y | | |
| Family History of Cardiovascular Risk Factors | Y | | |
| Physical Examination | | | Y |
| Medical Condition & Concomitant Medications | 1 | • | |
| Medical Conditions (Sjögren specific) | Y | | Y |
| Medical Conditions (non-Sjögren specific) | Y | | Y |
| Concomitant Medication | Y | | Y |
| NOTES: | L. | | |

#### NOTES:

Selected Primary Analysis study population displays will also be generated for the End of Study Analysis and are identified in Appendix 13: List of Data Displays. Where required, programming notes (Appendix 13 or Mock Shell Examples) have been included for any specific changes based on the Primary Analysis displays.

Y = Yes display generated.

<sup>[1]</sup> For End of Study, a further subject disposition table will be generated to summarize subject's completion status upto Week 52 & W68, subjects withdrawn and who continued or discontinued study visits.

<sup>[2]</sup> For End of Study, a further listing will be generated to capture important PDs related to COVID-19.

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Safety Analyses

## 7.1.1. Overview of Planned Analyses

The safety analyses will be based on the "Safety" population, unless otherwise specified.

Table 2 provides an overview of the planned safety Primary Analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

Table 2 Overview of Planned Safety Analyses

| Endpoint | | Ab | solute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | | ridual | | mary | | <u>/idual</u> |
| | T | F | F | L | T | F | F | L |
| Exposure | | | | ı | 1 | | | 1 |
| Extent of Exposure | Υ | | | Y | | | | |
| Adverse Events | | | | ı | 1 | | | 1 |
| All AEs [1] | Υ | | | Y | | | | |
| All Drug-Related AEs | Υ | | | | | | | |
| AEs of Special Interest | Υ | | | Y | | | | |
| Serious AEs | Υ | | | | | | | |
| Withdrawal AEs | Υ | | | Υ | | | | |
| Fatal Adverse Events | Υ | | | Υ | | | | |
| Common AEs [2] | Υ | | | | | | | |
| Reasons for Considering as SAE | | | | Y | | | | |
| Laboratory Values | l l | | | | • | | | 1 |
| Immunoglobulins | Υ | Υ | | Υ | Υ | <b>Y</b> [3] | | |
| Clinical Chemistry | <b>Y</b> [4] | | | Y | Y [4] | | | |
| Hematology | Y [4] | Υ | | Υ | Υ [4] [5] | | | |
| Liver | Υ | | | | | | | Υ |
| Urinalysis (Dipstick) | Υ | | | Y | | | | |
| Other Screening Tests [6] [7] | | | | Υ | | | | |
| C-Reactive Protein | Υ | | | | Y | | | |
| CD4 and CD8 | Υ | Υ | | Υ | | | | |
| ECGs | | | | | | | | |
| ECG | Υ | | | | | | | |
| Abnormal ECG | | | | Υ | | | | |
| Vital Signs | | | | | | | | |
| Vital Signs | Υ [8] | | | Υ | Υ [8] | | | |

| Endpoint | | Ab | solute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sur | nmary | Individual | | Sum | mary | Individual | |
| | T | F | F | L | T | F | F | L |
| Neurological Symptoms | | | | | | | | |
| Neurological Symptoms | Υ | | | Υ | | | | |
| Columbia-Suicide Severity | Rating | Scale | | | | | | |
| C-SSRS | Υ | | | Υ | | | | |
| Immunogenicity | • | • | | | | | • | • |
| Belimumab | Υ | | | Υ | | | | |
| Immunogenicity | | | | | | | | |
| Rituximab Immunogenicity9 | Υ | | | Y | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Listing will include subject's numbers for individual AE's & AE system organ classes, preferred terms and verbatim text. A separate listing will be generated for Primary & EoS to capture with subjects with post Week 68/FU events.
- 2. Common AEs are adverse events occurring with a frequency > 5%.
- 3. IgG, IgA & IgM will be reported
- 4. Including summaries of Toxicity grading
- 5. Including evaluation of shifts from baseline.
- 6. Positive/abnormal findings
- 7. Other screening tests include HIV, Hepatitis B (HBsAg), HbcAb, Hepatitis C (Hep C antibody), FSH, estradiol and serum or urine hCG pregnancy test.
- 8. Including evaluation of PCI criteria
- 9. Reported only for End of Study (Baseline is defined as Week 8)

Selected Primary Analysis safety displays will also be generated for the End of Study Analysis and are identified in Appendix 13: List of Data Displays. Where required, programming notes (Appendix 13 or Mock Shell Examples) have been included for any specific changes based on the Primary Analysis displays.

**Primary Analysis:** Summarized safety data for all completed visits up to Week 68 (where reported by visit) and up to Week 104 (where not reported by visit), with a cut-off date of 9 September 2019 (Week 52 LSLV).

On completion of the Primary Analysis, it was noted that the safety data included 39 AEs (out of a total of 49) reported during the IFU phase that were not within the defined scope of the protocol for AE collection. The over-reported AEs included 2 SAEs reported by 2 subjects; both were assessed as unrelated to study treatment. An additional blinded listing of the 49 AEs reported during the IFU period was generated. Full details are included in the Primary Analysis CSR.

**End of Study Analysis:** Summarize AE/AESI safety data for all completed visits up to Week 68 only to include AEs collected in the defined protocol AE collection period. An unblinded listing of the AEs reported during the IFU period will be generated, which will also include information as to whether the AE occurred pre or during the COVID-19 pandemic.

Additional safety analyses may (if required) also be conducted to further assess the impact of the over-reported AEs in the FU or COVID-19 pandemic.

## 7.1.2. Immunogenicity

#### **Exploratory Analyses: Immunogenicity**

#### **Endpoints**

- Immunogenic Response to Belimumab
- Immunogenic response to Rituximab (will not be reported until all subjects have completed the follow-up phases of the study)

#### **Summary Results Presentation**

The method for calculation of belimumab & rituximab immunogenic response is given in Section 11.5.6.1.

The belimumab and rituximab immunogenicity response will be summarized for the binding antibody assay by treatment group and visit. The table will include the number and proportion of subjects in each result category for each visit. Binding confirmatory assay results will be categorized as Negative, Positive, or Unknown. Positive samples in the binding assay are further categorized as Transient Positive (i.e. single positive response that does not occur at the final assessment) or Persistent Positive (i.e. positive response that occurs at least 2 consecutive assessments or a single result at the final assessment)

Belimumab only: Presence of neutralizing antibodies and titre for samples confirming positive in the blinding assay will be listed.

Rituximab: Baseline is Week 8. Titre for samples confirming positive in the blinding assay will be listed.

## 7.1.3. Immunoglobulin

#### **Exploratory Analyses: Immunoglobulin**

#### **Endpoints**

The number and percentage of subjects with immunoglobulin values (IgG, IgA, and IgM) below the LLN at each visit will be presented

The number and percentage of subjects with immunoglobulin values (IgG, IgA, and IgM) above the ULN at each visit will be presented

#### Worst IqG toxicity grade

The number and percentage of subjects at each toxicity grade will be assessed at baseline and also for anytime post baseline.

#### IgG toxicity ≥ 2 grade shift post-baseline

The number and percentage of subjects with at least one  $\geq$  2 grade shift as well as the specific shift categories: Grade 0 to 2, Grade 0 to 3, Grade 0 to 4, Grade 1 to 3, Grade 1 to 4 and Grade 2 to 4 will be computed by treatment group.

#### 7.1.4. Adverse Events of Special Interest

The AESI definitions from Section 15 and Section 16 of the current belimumab PSAP (Note: Version 5 was used for the interim analysis and version 6 for the final analysis) will be followed to identify the program level AESI. Search terms based on the current version of MedDRA (Primary Analysis = 22.0 and End of Study = 23.0) at the time of database release will be utilized. The additional study specific AESI are:

**Severe skin reaction**: All events identified by Severe Cutaneous Adverse Reactions SMQ broad search will be adjudicated (Preferred terms corresponding to broad search from SMQ are given in the Section 11.5.3.1)

**Cardiac Disorders:** All events identified by applying Cardiac Arrhythmias SMQ, Cardiac Failure SMQ, Cardiomyopathy SMQ, and Ischaemic heart disease SMQ will be adjudicated (Preferred terms corresponding to broad search from SMQ are given in Section 11.5.3.1)

**Posterior Reversible Encephalopathy Syndrome (PRES):** Defined as all events identified in the preferred term "Posterior Reversible Encephalopathy Syndrome".

**Progressive Multifocal Leukoencephalopathy (PML):** Defined as all events identified in the preferred term "Progressive multifocal leukoencephalopathy"

**Adverse events related to the biopsy:** Preferred terms corresponding to adverse events related to biopsy will be reviewed and adjudicated.

Malignancies, serious post-administration systemic reactions, potential opportunistic infections, suicide/self-injury, fatalities, severe infections and skin reactions will be adjudicated at the subject level by the GSK blinded Safety Review Team (SRT). Additionally, the study specific AESI's will be adjudicated at the subject level by the study team. Adjudication will be conducted periodically with a final adjudication completed prior to the DBF for the primary analysis. Further adjudications (periodically and prior to End of Study DBF) will also be performed for the End of Study analysis. Only adjudicated study specific AESI's will be reported.

An overall summary of AESI will be presented and each specific category of AESI will be presented separately by PT. Infection AESIs will also be presented by PT for all infections leading to discontinuation. The number and percentage of subjects with at least one occurrence and the number of events for each AESI will be provided. The AESI categories are:

#### **Malignant Neoplasms**

- Malignancies Excluding non-melanoma skin cancer (NMSC)
- Malignancies Including NMSC
- Solid Tumor
- Hematologic
- Skin (All)
  - o NMSC

- Excluding NMSC
- Tumors of unspecified malignancy adjudicated as malignant per GSK adjudication

#### **Post-Administration Systemic Reactions**

- Post-Administration Systemic Reactions per Anaphylactic Reaction Customized MedDRA Query (CMQ) narrow search
- Post-Administration Systemic Reactions per Anaphylactic Reaction CMQ broad search
- Post-Administration Systemic Reactions per Anaphylactic Reaction CMQ algorithmic search
- Serious Anaphylaxis per Sampson Criteria
- Serious Acute Post-Administration Systemic Reactions/Hypersensitivity per GSK adjudication
  - Serious Acute Post-Administration Systemic Reactions Excluding Hypersensitivity per GSK adjudication
  - Serious Acute Hypersensitivity Reactions per GSK adjudication
- Serious Delayed Acute Hypersensitivity Reactions per GSK adjudication
- Serious Delayed Non-Acute Hypersensitivity Reactions per GSK adjudication

#### **All Infections of Special Interest**

- All opportunistic infections per GSK adjudication
- Opportunistic infections per GSK adjudication excluding Tuberculosis and Herpes Zoster
  - Serious opportunistic infections per GSK adjudication excluding Tuberculosis and Herpes Zoster
- Active Tuberculosis
  - o Non-Opportunistic
  - o Opportunistic
- Herpes Zoster
  - Non-Opportunistic
  - o Opportunistic
    - Recurrent
    - Disseminated
- Sepsis

#### Depression/suicide/self-injury

- Depression (Inc. mood disorders and anxiety)
- Suicide/self-injury
- Serious Suicide/Self-injury per GSK Adjudication
  - o Suicidal Behaviour per GSK Adjudication
    - Completed Suicide per GSK Adjudication
  - Suicidal Ideation per GSK Adjudication
  - Self-injurious Behaviour Without Suicidal Intent per GSK Adjudication

**Deaths** 

#### **Study Specific AESI**

- Severe skin reaction per GSK Adjudication
- Cardiac Disorders
- Posterior Reversible Encephalopathy Syndrome (PRES)
- Progressive multifocal leukoencephalopathy (PML)
- Adverse events related to the biopsy

# 7.1.4.1. Post-Administration systemic reactions by Belimumab/Placebo Injection

Summaries of post-injection systemic reactions will be presented by the first six injections (belimumab/placebo) in addition to overall injections for the following categories:

- Post-Injection Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the injection or within 3 days after the injection)
- Serious Post-Injection Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the injection or within 3 days after the injection)
- Serious Acute Post-Injection Systemic Reactions/Hypersensitivity per GSK adjudication
- Serious Delayed Acute Post-Injection Systemic Reactions per GSK adjudication
- Serious Delayed Non-Acute Post-Injection Systemic Reactions per GSK adjudication

# 7.1.4.2. Post-Administration Systemic Reactions by Rituximab/Placebo Infusion

Summaries of post-infusion systemic reactions will be presented by the first two infusions (rituximab/placebo):

• Post-Injection Systemic Reactions per Anaphylactic Reaction CMQ broad search (on the day of the infusion or within 3 days after the infusion)

## 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Efficacy and Biomarker Analyses

## 8.1.1. Overview of Planned Efficacy and Biomarker Analyses

The secondary efficacy analyses will be based on the "Safety" population, unless otherwise specified.

Table 3 provides an overview of the planned efficacy Primary Analyses, with further details of data displays being presented in Appendix 13: List of Data Displays.

 Table 3
 Overview of Planned Efficacy and Biomarker Analyses

| Endpoint | Absolute | | | | | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats | Anal | ysis | Summary Individual | | | Stats Analysis | | | Sum | mary | Individual | | |
| | T | F | L | T | F | F | L | T | F | L | Т | F | F | L |
| Clinical Efficacy | | | | | | | | | | | | | | |
| ESSDAI Score | | | | Υ | Υ | | Υ | Υ | Υ | | Υ | Υ | | |
| (Uncorrected & | | | | | | | | | [2] | | | | | |
| Corrected) | | | | | | | | | | | | | | |
| ESSDAI Domains | | | | Υ | Υ | | Υ | | | | Υ | | | |
| (Uncorrected & | | | | | | | | | | | | | | |
| Corrected) | | | | | | | | | | | | | | |
| ESSDAI Responder | Y [2] | | | Υ | Υ | | | | | | | | | |
| (Corrected) | | | | | | | | | | | | | | |
| ClinESSDAI | | | | Υ | | | Υ | Y [2] | | | Υ | | | |
| (Corrected) | | | | | | | | | | | | | | |
| ClinESSDAI | | | | Υ | | | | | | | | | | |
| Responder | | | | | | | | | | | | | | |
| (Corrected) | | | | | | | | | | | | | | |
| ESSDAI Corrected | | | | | | | | | | | | <b>Y</b> [2] | | |
| /ClinESSDAI | | | | | | | | | | | | | | |
| Corrected Correlations | | | | | | | | | | | | | | |
| Stimulated Salivary | | | | Υ | | | Υ | Y [2] | | | Υ | Υ | | |
| Flow | | | | | | | | | | | | | | |
| Oral Dryness NRS | | | | Υ | | | Υ | Y [2] | | | Υ | Υ | | |
| Biomarker | | | | | | | | | | | | | | |
| Number of B cells | | | | Υ | | | Υ | Y [1] | | | <b>Y</b> [1] | <b>Y</b> [1] | | Υ |
| (CD20) /mm <sup>2</sup> in | | | | | | | | | | | | | | |
| Salivary Gland Biopsy | | | | | | | | | | | | | | |
| NOTES: | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- NRS, Numeric Response Scale
- [1] Based on change from baseline
- [2] Will not be generated for EoS

Selected Primary Analysis efficacy displays will also be generated for the End of Study Analysis and are identified in Appendix 13: List of Data Displays. Where required, programming notes (Appendix 13 or Mock Shell Examples) have been included for any specific changes based on the Primary Analysis displays.

#### 8.1.1.1. ESSDAI

ESSDAI scores disease activity in 12 domains. In 5 (renal, PNS, CNS, cutaneous and pulmonary) of the domains, ESSDAI requires that if activity has been present for greater than or equal to 12 months then it must be treated as irreversible damage and the activity should be scored as zero (Seror, 2015a). This is a problem for clinical trials of long duration such as study 201842 because it can result in misleading evidence of reduced activity. For that reason, a corrected ESSDAI score will be calculated.

#### The ESSDAI Corrected score will be calculated as:

- For each damage eligible domain
  - where damage is scored as present for 1st time after screening THEN corrected activity score = damage score for that domain for that visit and the activity score for all subsequent visits should be changed to equal the corresponding damage domain score
  - Except in rare cases where the activity score for the visit concerned is already
    equal to or greater than the damage score, in which case no change should be
    made.
- If damage is scored as present at screening **AND** if the damage score increases in level of involvement (low to moderate or moderate to high) after the screening visit then the activity score for that domain for that visit and all subsequent visits should be changed to equal the corresponding damage domain score
  - Except in rare cases where the activity score for the visit concerned is already
    equal to or greater than the damage score, in which case no change should be
    made.
- If damage is scored at screening and remains constant across visits, then no programmed correction can or should be made to the activity scores.

Further details are included in Section 11.5.4 Efficacy.

The primary inference will be based on the corrected ESSDAI score, with the uncorrected score being used as a supporting sensitivity analysis to assess any impact.

For the Primary Analysis, the correction could not be applied for 1 subject (ID one domain of ESSDAI. The complexity of disease scoring in the PNS domain for this subject prevented the correction algorithm from appropriately recording low activity for this domain from Week 24 onwards. Consequently, the total corrected ESSDAI score for this subject is underestimated by 5 points for each visit from Week 24 onwards. Only a single domain of ESSDAI was affected and there is thought to be no impact on the interpretation of the overall corrected ESSDAI data. This subject will subsequently not be corrected for the End of Study Analysis.

#### 8.1.2. Planned Efficacy and Biomarker Statistical Analyses

#### Secondary Statistical Analyses – Efficacy (MMRM)

#### Endpoint(s)

- Change from Baseline in ESSDAI Total Score (Uncorrected & Corrected)
- ESSDAI Domain Scores (Corrected)
- ESSDAI Improvements (At Least 1 Category on Domain Score) (Corrected)
- ESSDAI Worsening (At Least 1 Category on Domain Score) (Corrected)
- Change from Baseline in Stimulated Salivary Flow
- Change from Baseline in Oral Dryness Numeric Response Scale

#### **Model Specification**

- Endpoints will be statistically analyzed using a mixed model repeated measures (MMRM)
- Terms fitted in MMRM models will include:

Fixed Categorical : Treatment, Visit, Treatment \* Visit Interaction
Fixed Continuous Covariates : Baseline (see Section 5.2 for baseline definition)

Repeated : Visit

 For the analysis of salivary flow and oral dryness numeric response, ESSDAI stratification (moderate or severe) will also be included as a fixed categorical term.

#### **Model Checking & Diagnostics**

• Refer to Appendix 9: Model Checking and Diagnostics for Statistical analyses.

#### **Model Results Presentation**

- Adjusted means and corresponding standard error of means (SEs) and 95% confidence intervals will be
  presented for changes from baseline on each treatment by Visit. together with estimates and the
  corresponding 95% confidence intervals for the comparisons of interest.
- If the model checking deems the above parametric analysis to be unsuitable, nonparametric rank Hodges-Lehmann's confidence intervals will be provided in order to assess the robustness of the parametric analysis. This will be carried out in addition to the parametric analyses
- For ESSDAI Total Score (Uncorrected and Corrected), plots of LS means and SE for changes from baseline for each treatment at all visits up to Week 52 as derived from the MMRM model will be presented.

#### **Summary Results Presentation**

- Summary statistics (n, mean, median, minimum and maximum), will be presented on the absolute values at each visit and the change from baseline at each visit.
- Plots of the mean and corresponding SE on changes from baseline over time for each treatment will also be presented.

#### Supportive Analyses

- For ESSDAI, additional statistical analysis using MMRM will be conducted for changes from baseline for each treatment at all visits up to Week 68/FU, using the completer population.
- The relationship between Scoring of ESSDAI (corrected) and Clinical ESSDAI (corrected) will be assessed graphically.
- ESSDAl domain scores (Corrected) will be summarized. The number and proportion of subjects reporting no, Low, moderate (and high response where applicable), will be computed for each of the 12 domains by treatment and visit.
- Improvements in ESSDAI Domain Scores (corrected) will be evaluated. For each domain, the number
  and proportion of improvers (i.e. higher to lower category) out of the subjects who had an activity score
  on the specific domain at baseline will be computed. The number and proportion of subjects with
  worsening will be assessed for each ESSDAI Domain (Corrected). The domain level denominator is
  the subset of subjects who do not have highest level of symptom at baseline.

#### Secondary Statistical Analyses – Efficacy (Bayesian)

#### Endpoint(s)

Change from baseline in Total ESSDAI Score (Corrected)

#### **Model Specification**

- A Bayesian repeated Measures model will be used to fit the change from baseline in Total ESSDAI Score (Corrected).
- A multivariate (MVN) normal distribution is assumed for the vector of changes from baseline for each subject (i.e. the change from baseline at weeks 12, 24, 36 & 52).
- Markov-Chain-Monte-Carlo (MCMC) method in SAS will be used to derive the posterior distributions of the endpoint.
- A linear model for Change from Baseline (CFB) in Total ESSDAI Score at each Week (visit) will be constructed to model the within-subject covariance structures:

CFB = Intercept + Treatment + Baseline + Week + Treatment\*Week

Terms fitted in the model will include:

Fixed Categorical: Week (Week 12 to Week 52), Treatment, Treatment\*Week Interaction

Fixed Continuous: Baseline

Random: Subject

- The prior for the variance covariance matrix will follow an Inverse Wishart Distribution.
- Set seed=123456 with simulation size of 100,000 (i.e. every 10<sup>th</sup> iteration will be kept which will form the final MCMC (thinned) sample of 10,000) & 10,000 burn-in iterations. The simulation size and number of burn-in iterations may be updated during the convergence check.
- Vague priors (normal (0, var=1e6)) will be used for regression parameters.

#### **Model Checking & Diagnostics**

Refer to Appendix 9: Model Checking and Diagnostics for Statistical analyses.

#### **Summary Results Presentation**

- The sample size n, mean, median, standard deviation and highest posterior density (HPD: smallest interval width among all credible intervals) interval will be presented from the posterior density function.
- The posterior distribution will be used to produce several probability statements (where  $\theta$  is the ESSDAI change from baseline), such as (but not limited to and maybe refined):
  - O Pr ( $\theta$  Co-administration, 24w  $\theta$  Placebo, 24w < 0 | 201842 data)
  - $\circ$  Pr ( $\theta$  Co-administration,  $52w \theta$  Placebo,  $52w < 0 \mid 201842$  data)
  - O Pr ( $\theta$  Co-administration,  $24w \theta$  Placebo,  $24w < 3 \mid 201842$  data)
  - O Pr ( $\theta$  Co-administration,  $52w \theta$  Placebo,  $52w < 3 \mid 201842$  data)
  - $\circ$  Pr ( $\theta$  Co-administration, 24w  $\theta$  Belimumah, 24w < 0 | 201842 data)
  - O Pr ( $\theta$  Co-administration,  $52w \theta$  Belimumab,  $52w < 0 \mid 201842$  data)
  - $\circ$  Pr ( $\theta$  Co-administration,  $24w \theta$  Rituximab,  $24w < 0 \mid 201842$  data)
  - $\circ$  Pr ( $\theta$  Co-administration,  $52w \theta$  Rituximab, 52w < 0 | 201842 data)
  - $\circ$  Pr ( $\theta_{\text{Belimumab}}$ , 24w  $\theta_{\text{Placebo}}$ , 24w < 0 | 201842 data)
  - $\circ$  Pr ( $\theta$  Belimumab,  $52w \theta$  Placebo,  $52w < 0 \mid 201842$  data)
  - $\circ$  Pr ( $\theta$  Belimumab, 24w  $\theta$  Placebo, 24w < 3 | 201842 data)
  - $\circ$  Pr ( $\theta_{\text{Belimumab}}$ , 52w  $\theta_{\text{Placebo}}$ , 52w < 3 | 201842 data)

#### Secondary Statistical Analyses – Efficacy

#### **Endpoints**

ESSDAI Responders (Corrected)

#### **Summary Results Presentation**

- The proportion of ESSDAI responders based on corrected total ESSDAI score will be summarized descriptively using counts and percentages by treatment and visit. Responders are defined as below
  - Responders 1 Subjects with a reduction in total ESSDAI of at least 5 points over baseline
  - Responders 2 Subjects with a reduction in total ESSDAI of at least 3 points over baseline
  - Responders 3 Subjects with a reduction in total ESSDAI of at least 3 points over baseline, and ESSDAI Total Score <5</li>
  - Responders 4 ESSDAI Total Score < 5
- The proportion of ESSDAI responders will be presented as a bar chart grouped by treatment for each visit.

#### **Model Specification**

- Responder endpoints will be statistically analysed using a Generalised Estimating Equations (GEE) model
- The model will be fitted using an unstructured covariance structure of the correlated responses.
- Terms fitted in GEE models will include:

Fixed Categorical : Treatment, Visit, Treatment\*Visit Interaction

Fixed Continuous Covariate: Baseline Total ESSDAI Score

Repeated : Visit

#### **Model Checking & Diagnostics**

Refer to Appendix 9: Model Checking and Diagnostics for Statistical analyses.

#### **Model Results Presentation**

- The Binary endpoints will be summarized using counts and proportions of subjects achieving a response by treatment group.
- Differences in the proportions of subjects achieving response between treatment groups will be summarized by Visit (up to Week 52). 95% CI for the differences will be constructed using their asymptotic standard errors (asymptotic Wald confidence limits) without continuity correction.
- Point estimates and corresponding 95% confidence intervals will be constructed using contrasts for the treatment by day interactions.

#### Secondary Statistical Analyses – Efficacy

#### Endpoint(s)

ClinESSDAI Responders (Corrected)

#### **Summary Results Presentation**

 The proportion of ESSDAI responders based on corrected total ESSDAI score will be summarized descriptively using counts and percentages by treatment and visit. Responders are defined as subjects with a reduction in total ClinESSDAI of at least 3 points over baseline

## Secondary Statistical Analyses – Biomarker

#### Endpoint(s)

Absolute change from baseline in Number of B Cells (CD20)/mm<sup>2</sup> in salivary gland biopsy at Week 24

#### **Model Specification**

The absolute change at Week 24 will be analysed using the Hodges-Lehmann method to provide a
#### 201842 | Statistical Analysis Plan EoS RAP 15 Sep 2020 | TMF-2108787 | 4.0

#### CONFIDENTIAL

2020N437857\_00 201842

#### Secondary Statistical Analyses – Biomarker

95% confidence interval for the contrasts of interest specified in Section 2.5 at Week 24

#### **Model Result Presentation**

 Along with the number of subjects (n) and median of absolute change from baseline of each treatment group, median difference with 95% Confidence intervals estimated from the H-L method will be presented at week 24 for the contrasts of interest.

#### **Summary Results Presentation**

• Summary statistics (n, mean, median, minimum and maximum) will be presented on the absolute values and the absolute change from baseline at Week 24.

## 8.2. Pharmacokinetic Analyses

#### 8.2.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the Pharmacokinetic (PK-B and PK-R) populations, unless otherwise specified.

Table 4 provides an overview of the planned primary analyses, with full details being presented in Appendix 13: List of Data Displays.

Table 4 Overview of Planned Pharmacokinetic Analyses

| Endpoint | | | Untr | ansfo | rmed | | | Log-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Individual | |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Serum Drug<br>Concentrations | | | | Υ | Υ | <b>Y</b> [1] | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modeling) conducted.
- o Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- o Individual = Represents FL related to any displays of individual subject observed raw data.
- 1. Linear and Semi-Log plots will be created on the same display.

## 8.2.2. Drug Concentration Measures

Refer to Appendix 4: Data Display Standards & Handling Conventions (Section 11.4.1 Reporting Process & Standards).

Serum belimumab concentrations will be listed and summarized by visit and nominal time. Standard summary statistics will be calculated (i.e. mean, standard deviation, and 95% confidence interval of mean, geometric mean, 95% confidence interval for geometric mean, % coefficient of variation (CV), median, minimum and maximum). Individual subject and median PK concentrations profiles will be graphically presented.

#### 8.2.2.1. Statistical Analysis of Pharmacokinetic Parameters

No formal statistical analyses will be performed.

## 8.3. Pharmacokinetic / Pharmacodynamic Analyses

The Pharmacokinetic / Pharmacodynamic analyses will be based on the "Safety" and "PK-B" populations, unless otherwise specified.

The primary goal of this analysis is to characterize the pharmacokinetic/pharmacodynamic relationship of belimumab administered through injection in subjects with Primary Sjogren's syndrome.

1. No formal population pharmacokinetic/pharmacodynamics analyses are planned. The relationships will be explored using descriptive methods only.

Table 5 provides an overview of the pharmacokinetic/pharmacodynamics analyses, with details being presented in Appendix 13: List of Data Displays.

Table 5 Overview of Pharmacokinetic / Pharmacodynamic Analyses

| Endpoint | | | | Absolu | ıte | | | | Cł | nange | from | Baseli | ne | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | alysis | Sum | mary | Indiv | /idual | Stat | s Ana | lysis | Sum | mary | Individual | |
| | T | F | L | T | F | F | L | Т | F | L | Т | F | F | L |
| Flow cytometry B cells (CD19+) /serum Belimumab concentration Comparison | | | | | | Y<br>[1] | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] For Belimumab and Combination Treatment Groups

## 9. OTHER STATISTICAL ANALYSES

## 9.1. Exploratory

## 9.1.1. Overview of Exploratory Analysis

The exploratory analyses will be based on the "Safety" population, unless otherwise specified.

Table 6 provides an overview of the planned exploratory Primary Analyses, with full details of data displays being presented in Appendix 13: List of Data Displays.

Table 6 Overview of Exploratory Analyses

| Endpoint | | | | Absol | ute | | | | Cł | nang | e fron | n Basel | line | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Α | Stat<br>naly | - | Sumi | mary | Indiv | ridual | _ | tats<br>alysi | s | Sun | nmary | Indiv | vidual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Clinical Efficacy | | | | • | | | | | | | | | • | |
| Ocular Dryness NRS | | | | Υ | | | Υ | | | | Υ | Υ | | |
| Lacrimal Gland | | | | Υ | | | Υ | | | | Υ | Υ | | |
| Function | | | | | | | | | | | | | | |
| PGA | | | | Υ | | | Υ | | | | Υ | Υ | | |
| Unstimulated Salivary | | | | Υ | | | Υ | | | | Υ | Υ | | |
| Flow | | | | | | | | | | | | | | |
| ESSDAI | | | | Υ | | | Υ | | | | | | | |
| Supplementary | | | | | | | | | | | | | | |
| Damage Assessments | | | | | | | | | | | | | | |
| Biomarkers | | | | | | | | | | | | | | |
| BLyS levels in blood | | | | | | | | | | | | | | |
| Free BLyS | | | | Υ | | | Υ | | | | Y[1] | Υ[1] | | |
| Total BLyS[4] | | | | | | | | | | | | | | |
| Flow | | | | Υ | <b>Y</b> [3] | | Υ | <b>Y</b> [1, | | | Y[1] | <b>Y</b> [1,3] | | |
| CytometryParameters <sup>2</sup> | | | | ' | 1 | | ' | 3, 5] | | | 1 | 1 | | |
| Serologic Markers <sup>2</sup> | | | | Y | | | Υ | | | | Υ[1] | Y[1] | | |
| Complement Factors <sup>2</sup> | | | | Υ | | | Υ | | | | Υ[1] | Υ[1] | | |
| Exploratory Minor<br>Salivary Gland<br>Histology<br>Assessments <sup>2</sup> | | | | Υ | Υ[3] | | Υ | Y[1,3,<br>5] | | | Y[1] | Υ[1,3] | | |
| Serum Chemokines - CXCL13 | | | | Υ | | | | | | | Υ[1] | <b>Y</b> [1] | | |
| ESSDAI/Salivary<br>Gland CD20+ B cell<br>Evaluation | | | | | <b>Y</b> [5] | | | | | | | | | |
| Flow cytometry B<br>Cells (CD19+) /serum<br>BLyS Evaluation | | | | | Y | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- NRS; Numeric Response Scale
- 1. Only Percentage Change from Baseline will be presented
- 2. See Section 11.5.6 for parameters.
- 3. Subset of the parameters as defined in Section 9.1.2
- 4. Total BLyS concentration only for End of Study analyses
- 5. Will not be reported for End of Study

Selected Primary Analysis exploratory displays will also be generated for the End of Study Analysis and are identified in Appendix 13: List of Data Displays. Where required, programming notes (Appendix 13 or Mock Shell Examples) have been included for any specific changes based on the Primary Analysis displays.

## 9.1.2. Planned Exploratory Analyses

#### **Exploratory Analyses: Clinical Efficacy and Biomarkers**

#### **Endpoints**

#### **Salivary Gland Assessments**

- Absolute values
- Change from Baseline
- Percentage Change from Baseline

Refer to Table 13 for parameters to be included in the summary table

#### **Summary Results Presentation**

• Descriptive statistics (N, n, arithmetic mean, standard deviation, median, minimum and maximum) will be calculated and summarized by treatment group and visit for the above endpoints. Absolute values and changes from baseline will be assessed.

#### **Model Results Presentation**

The absolute change from baseline for selected parameters: Lymphocyte Focus Score (in 4mm²), B (CD20) / T (CD3) cell ratio and Plasma cell (CD138+; both - CD20pos and CD20neg) count/mm²) at Week 24 will be analysed using Hodges-Lehmann method to provide a non-parametric 95% confidence interval for the contrasts of interest at Week 24 specified in Section 2.5.

#### **Endpoints**

- Ocular Dryness NRS
- Lacrimal gland function (Schirmers test see Section 11.5.4)
- PGA
- Unstimulated Salivary flow
- Free BLvS
- Total BLyS (NOTE: Total BLyS concentration only for End of Study analysis)
- Serologic Markers: SS-A, SS-B, Rheumatoid factor, Lambda and kappa free light chains Beta 2 microglobulins
- Complement Factors (C3, C4, CH50)
- Exploratory Minor Salivary Gland histology assessments (see Section 11.5.6)
- Serum chemokine CXCL13

Refer to Table 12 for further parameter details

#### **Exploratory Analyses: Clinical Efficacy and Biomarkers**

#### **Summary Results Presentation**

- Descriptive statistics (N, n, arithmetic mean, standard deviation, median, minimum maximum) will be calculated and summarized by treatment group and visit for the above endpoints.
- Absolute values and changes from baseline will be assessed.

#### **Exploratory Analyses: Damage Scoring**

Damage Scores for Cutaneous, pulmonary, renal, PNS and CNS domains of ESSDAI

#### **Summary Results Presentation**

- The number and percentage of subjects who report damage will be summarized for each of these 5 domains by treatment and visit.
- For the subset of subjects who report damage, a listing will be produced to display damage scoring
  alongside ESSDAI domain scores. The listing will include only the subject/domain combinations where
  there is damage reported, and in each case assessments from all visits to be presented.

#### **Exploratory Analyses: Flow Cytometry**

Refer to Table 11 for further details on parameters

#### **Model Results Presentation**

 The absolute change from baseline in cell count for each parameter at Week 24 will be analysed using Hodges-Lehmann method to provide a non-parametric 95% confidence interval for the contrasts of interest at Week 24 specified in Section 2.5. Similarly, this analysis will be repeated for the absolute changes in cell counts for each parameter at Week 52

#### **Summary Results Presentation**

- The cell counts and percentage change from baseline in cell counts will be summarized (n, mean, median, sd, min, max). Median (± IQR) will be presented by treatment and visit.
- B cells (CD19+) will be summarized by treatment and visit
- In addition, Naïve B Cells, Memory, Plasmablasts (all), Plasmablast (CD20+), Plasmablast (CD20-), Transitional and Activated B Cells, will all be additionally expressed as % of CD19+ cells and summarized by treatment and visit.

#### Sensitivity and Supportive Statistical Analyses

The relationship between the change in salivary gland B cell quantification from baseline and ESSDAI scores will be explored:

• Scatter plots of changes from baseline to Week 24 for Total ESSDAI score vs Change from baseline to Week 24 in salivary gland B cells will be produced.

#### 9.2. Health Outcomes

#### 9.2.1. Overview of Health Outcome Analysis

Table 7 provides an overview of the planned health outcomes, with full details of data displays being presented in Appendix 13: List of Data Displays

Table 7 Overview of Health Outcome Analyses

| Endpoint | | | A | bsolu | te | | | Change from Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sta | ts Ana | lysis | Sum | mary | Indiv | /idual | | Stats | | Sum | mary | Indiv | /idual |
| | | | - | | - | | | Α | nalys | is | | | | |
| | Т | F | L | T | F | F | L | Τ | F | L | Т | F | F | L |
| Patient reported health | outc | omes | | | | | | | | | | | | |
| ESSPRI Score | | | | Υ | | | Υ | | | | Υ | Υ | | |
| ESSPRI Domains - | | | | Υ | | | Υ | | | | Υ | Υ | | |
| Dryness, Fatigue, Pain | | | | | | | | | | | | | | |
| ESSPRI Responders | Υ | | | Υ | Υ | | | | | | | | | |
| | [1] | | | | | | | | | | | | | |
| PtGA | | | | Υ | | | Υ | | | | Υ | | | |
| PROFAD-SSI-SF | | | | Υ | | | Υ | | | | Υ | | | |
| Subscores – PROF, | | | | | | | | | | | | | | |
| PROFAD and SSI | | | | | | | | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modeling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data. [1] Will not be generated for EoS

Selected Primary Analysis health outcomes displays will also be generated for the End of Study Analysis and are identified in Appendix 13: List of Data Displays. Where required, programming notes (Appendix 13 or Mock Shell Examples) have been included for any specific changes based on the Primary Analysis displays.

Exploratory analyses of the EXIT Interview Data will be conducted in a separate report under the direction of the VEO/PRO Department after the study is reported and once EXIT Interview data has been delivered by ICON.

## 9.2.2. Planned Health Outcomes Statistical Analyses

#### **Secondary Statistical Analyses**

#### Endpoint(s)

- Change from Baseline in Total ESSPRI Score
- Change from Baseline in ESSPRI Dryness Domain
- Change from Baseline in ESSPRI Fatigue Domain
- Change from Baseline in ESSPRI Pain Domain
- Change from baseline in PROF Subscore

#### **Secondary Statistical Analyses**

- Change from baseline in PROFAD Subscore
- Change from baseline in SSI Subscore (assessed for female subjects only)

#### **Summary Results Presentation**

- Summary statistics for observed values and change from baseline (i.e. screening) will be presented by treatment group and visit, for the dryness domain, fatigue domain, pain domain, and total ESSPRI score
- Summary statistics for observed values and change from baseline will be presented by treatment group for the total PROF, PROFAD and SSI Subscore at each time point.

#### Endpoint(s)

ESSPRI Responders

#### **Summary Results Presentation**

- The proportion of ESSPRI responders will be summarized descriptively using counts and percentages by treatment and visit. The ESSPRI responders are defined as below
  - Responders 1 Decrease of Total ESSPRI score of at least 1 point or at least 15% relative to baseline
  - Responders 2 Subjects with baseline score of ≥ 5 and Total ESSPRI score of < 5
- The proportion of subjects with an ESSPRI response will be presented as bar chart grouped by treatment for each visit.

#### **Model Specification**

- Responder endpoints will be statistically analysed using a Generalised Estimating Equations (GEE) model using visits up to Week 52
- The model will be fitted using an unstructured covariance structure of the correlated responses.
- Terms fitted in GEE models will include:

Fixed Categorical : Treatment, Visit, Treatment\*Visit Interaction

Fixed Continuous Covariate: Baseline ESSPRI Score

Repeated : Visit

#### **Model Checking & Diagnostics**

Refer to Appendix 9: Model Checking and Diagnostics for Statistical analyses.

#### **Model Results Presentation**

- The Binary endpoints will be summarized using counts and proportions of subjects achieving a response by treatment group.
- Differences in the proportions of subjects achieving response between treatment groups will be summarized by Visit. 95% CI for the differences will be constructed using their asymptotic standard errors (asymptotic Wald confidence limits) without continuity correction.
- Point estimates and corresponding 95% confidence intervals will be constructed using contrasts for the treatment by day interactions.

#### **Endpoints**

PtGA

#### **Summary Results Presentation**

 Summary statistics for actual PtGA scores as well as changes from baseline will be presented for each time-point by treatment group.

#### Secondary Statistical Analyses (Bayesian)

#### Endpoint(s)

• Change from Baseline in Total ESSPRI Score

#### **Model Specification**

- A Bayesian repeated Measures model will be used to fit the change from baseline in Total ESSPRI Score.
- A multivariate (MVN) normal distribution is assumed for the vector of changes from baseline for each subject (i.e. the change from baseline at weeks 12, 24, 36 & 52).
- Markov-Chain-Monte-Carlo (MCMC) method in SAS will be used to derive the posterior distributions of the endpoint.
- A linear model for Change from Baseline (CFB) at each Week (visit) will be constructed to model the within-subject covariance structures:

CFB = Intercept + Treatment + Baseline + Week + Treatment\*Week

Terms fitted in the model will include:

Fixed Categorical: Week (Week 12 to Week 52), Treatment, Treatment\*Week Interaction

Fixed Continuous: Baseline

Random: Subject

- The prior for the variance covariance matrix will follow an Inverse Wishart Distribution.
- Set seed=123456 with simulation size of 100,000 (i.e. every 10<sup>th</sup> iteration will be kept which will form the final MCMC (thinned) sample of 10,000) & 10,000 burn-in iterations. The simulation size and number of burn-in iterations may be updated during the convergence check.
- Vague priors (normal (0, var=1e6)) will be used for regression parameters.

## **Model Checking & Diagnostics**

• Refer to Appendix 9: Model Checking and Diagnostics for Statistical analyses.

#### **Summary Results Presentation**

- The sample size N, mean, standard deviation and highest posterior density (HPD: smallest interval width among all credible intervals) interval will be presented from the posterior density function.
- The posterior distribution will be used to produce several probability statements (where θ is the Total ESSPRI change from baseline), such as (but not limited to and maybe refined):

```
O Pr (\theta co-administration, 24w – \theta Placebo, 24w < 0 | 201842 data)
```

- $\circ$  Pr (θ co-administration, 52w θ Placebo, 52w < 0 | 201842 data)
- $\circ$  Pr ( $\theta$  co-administration,  $24w \theta$  Placebo,  $24w < 0.67 \mid 201842$  data)
- $\circ$  Pr ( $\theta_{\text{Co-administration}}$ , 52w  $\theta_{\text{Placebo}}$ , 52w < 0.67 | 201842 data)

```
\circ Pr (\theta Co-administration, 24w - \theta Belimumab, 24w < 0 \mid 201842 data)
```

- $\circ$  Pr ( $\theta$  co-administration,  $52w \theta$  Belimumab,  $52w < 0 \mid 201842$  data)
- Pr ( $\theta$  co-administration, 24w  $\theta$  Rituximab, 24w < 0 | 201842data) Pr ( $\theta$  co-administration, 52w –  $\theta$  Rituximab, 52w < 0 | 201842data)

```
\circ Pr (\theta Belimumab, 24w - \theta Placebo, 24w < 0 \mid 201842 data)
```

- $\circ$  Pr ( $\theta$  Belimumab,  $52w \theta$  Placebo,  $52w < 0 \mid 201842$  data)
- $\circ$  Pr ( $\theta_{\text{Belimumab}}$ , 24w  $\theta_{\text{Placebo}}$ , 24w < 0.67 | 201842 data)
- O Pr ( $\theta$  Belimumab,  $52w \theta$  Placebo,  $52w < 0.67 \mid 201842$  data)

201842 | Statistical Analysis Plan EoS RAP 15 Sep 2020 | TMF-2108787 | 4.0

CONFIDENTIAL

2020N437857\_00 201842

## 9.2.3. Planned Health Outcomes Psychometric Analyses

As the original validation of ESSPRI demonstrated a fairly low sensitivity to change, validation analyses will be repeated to support interpretation of the data (including the ESSPRI responder analysis). The analyses will be conducted by a PRO external vendor, following unblinding for the Primary Analyses have been completed. The analysis will be done under the direction of the VEO-PCO Department.

10. REFERENCES

GlaxoSmithKline Document Number 2014N220285\_06 Protocol Amendment 06: A randomized, double blind (sponsor open), comparative, multi-center study to evaluate the safety and efficacy of subcutaneous belimumab (GSK1550188) and intravenous rituximab co-administration in subjects with primary Sjögren's syndrome. Effective date 25-JUN-2019.

Seror R, Bowman SJ, Brito-Zeron P, Theander E, Bootsma H, Tzioufas A, et al. EULAR Sjögren's syndrome disease activity index (ESSDAI): a user guide. RMD Open. 2015a;1(1):e000022.

Seror R, Meiners P, Baron G, Bootsma H, Bowman SJ, Vitali C, et al. Development of the ClinESSDAI: a clinical score without biological domain. A tool for biological studies. Ann Rheum Dis. 2016 Nov;75(11):1945–50.

Seror R, Theander E, Brun JG, Ramos-Casals M, Valim V, Dörner T, et al. Validation of EULAR primary Sjögren's syndrome disease activity (ESSDAI) and patient indexes (ESSPRI). Ann Rheum Dis. 2015b May;74(5):859–66.

#### 11. APPENDICES

# 11.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

#### 11.1.1. Exclusions from Per-Protocol Population

Subjects will be excluded from the per-protocol population if any of the following criteria apply. The outputs for the per-protocol population will not be produced if the per-protocol population comprises >85% of the safety population subjects.

- Received wrong treatment most of the time (>50% of the time).
- Did not receive treatment most of the time (>50% of the time).
- Did not have a clinical diagnosis of Primary Sjögren's Syndrome according to Inclusion Criterion #2.
- Did not have baseline unstimulated salivary flow >0.0 mL/min or stimulated baseline salivary flow >0.05 mL/min) as defined by inclusion criterion #3.
- Did not have symptomatic oral dryness (≥5/10 on subject completed Numeric Response Scale) as defined by inclusion criterion #4.
- Did not have systemically active disease defined as an ESSDAI score ≥5 at screening (Inclusion Criterion 5).
- Received an excluded systemically administered immunosuppressive or immunomodulatory medication prior to screening (see Exclusion Criteria 17-22).
- Received a prohibited systemically administered immunosuppressive or immunomodulatory medication prior to Week 52.
- Deviation from study blind/unblind procedures: Investigator/site staff did not remain blinded to one or both treatment assignments through Week 52/Early Withdrawal Visit.
- Other, a deviation that does not satisfy the above criteria, however, in the judgment of the clinical team, including the medical monitor, constitutes an exclusion from the Per-Protocol population.

A participant meeting any of the following criteria will be excluded from the Per-Protocol population:

| Exclusion Criteria | Protocol Deviation<br>Category | Protocol Deviation<br>Subcategory |
|---|---|---|
| Received wrong treatment most of the time (>50% of the time). | Wrong study treatment/<br>administration/ dose | Wrong study treatment or assignment administered |
| Did not receive treatment most of the time (>50% of the time). | N/A | N/A |
| Did not have a clinical diagnosis of Primary Sjögren's according to Inclusion Criterion #2. | Eligibility criteria not met | Documented Primary Sjögren's Syndrome by American European Consensus Group criteria including: either SS-A or SS-B positive. |
| Did not have baseline unstimulated salivary flow >0.0 mL/min or stimulated baseline salivary flow >0.05 mL/min) as defined by inclusion criterion #3. | Eligibility criteria not met | Baseline unstimulated salivary flow >0.0 mL/min or evidence of glandular reserve function (stimulated baseline salivary flow >0.05 mL/min). |
| Did not have symptomatic oral dryness (≥5/10 on subject completed Numeric Response Scale) as defined by inclusion criterion #4. | Eligibility criteria not met | Symptomatic oral dryness<br>(≥5/10 on subject completed<br>Numeric Response Scale) |
| Did not have systemically active disease defined as an ESSDAI score ≥5 at screening (Inclusion Criterion 5). | Eligibility criteria not met | Systemically active disease,<br>ESSDAI ≥5 points OR (for sites<br>in ITALY ONLY) Systemically<br>active disease, ESSDAI≥5<br>points and with at least: a) 1<br>extraglandular domain<br>moderate, OR b) 2<br>extraglandular domains low. |
| Received an excluded medication prior to screening (per Exclusion Criteria 17-22). | Eligibility criteria not met | Check the Protocol Section 5.2 |
| Received a prohibited medication prior to Week 52. | Excluded medication, vaccine or device | Medication, excluded by the protocol, was administered |
| Study blind/unblind procedures: Investigator/site staff did not remain blinded to one or both treatment assignments through Week 68/Exit visit efficacy evaluation. | Study Procedures | Study blinding/unblinding procedures |
| Other, a deviation that does not satisfy the above criteria, however, in the judgment of the clinical team, including the medical monitor, constitutes an exclusion from the Per Protocol population. | N/A | N/A |

2020N437857\_00 201842

## 11.2. Appendix 2: Schedule of Activities

## 11.2.1. Protocol Defined Schedule of Events

| | p<br>or | | | | | | Dοι | ıble B | lind T | reatme | ent Pe | riod | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | Screening (up to 35 days prior to Day 0) | Day 0 | 7 ± 1 days | 28 ± 7days | 56 ± 7days | 70 ± 7 days | 84 ± 7 days | 112 ± 7days | 140 ± 7days | 168 ± 7days | 196± 7days | 224 ± 7days | 252 ± 7days | 280 ± 7days | 308 ± 7days | 336 ± 7days | 364 ± 7days | General<br>follow<br>up<br>period <sup>1</sup> | Individualized<br>follow up<br>period (IFU) <sup>6</sup> | l IFU<br>Final<br>Visit |
| Study Week | W -5 | | W1 | W4 | W8 | W10 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44 | W48 | W52 | W68 | | |
| Informed consent | Χ | | | | | | | | | | | | | | | | | | | |
| Inclusion and exclusion criteria | Χ | | | | | | | | | | | | | | | | | | | |
| Demography | Х | | | | | | | | | | | | | | | | | | | |
| Full physical exam | Х | X3 | | | | | | | | | | | | | | | Χ | Х | | Х |
| Abbreviated physical exam symptom directed | | | Х | Х | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | | Х | |
| Past & current medical conditions [including AECG criteria & CV medical history] | Х | | | | | | | | | | | | | | | | | | | |
| Urine pregnancy test (WCBP) in clinic9 | Χ | Х3 | | Χ | Χ | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Х | Х |
| Concomitant medication review | X10 | Хз | Χ | Χ | Χ | Χ | Χ10 | Χ | Χ | Χ10 | Χ | Χ | Χ10 | Χ | Χ | Χ | Χ10 | X10 | Х | X10 |
| Study Treatments | | | | | | | | | | | | | | | | | | | | |
| Randomization | | Χ | | | | | | | | | | | | | | | | | | |
| Belimumab/placebo.(weekly, home, except 1st & 2nd dose), last dose wk 51 | | X <sup>11</sup> | χ11 | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | | | | |
| Monitor in clinic after dosing for 3hrs (1st & 2nd dose of belimumab/pbo) | | Х | Χ | | | | | | | | | | | | | | | | | |
| Rituximab/placebo (at site) | | | | | Χ8 | Χ8 | | | | | | | | | | | | | | |

2020N437857\_00 201842

| | o o | | | | | | Dοι | ıble Bl | lind Tr | reatme | ent Pe | riod | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | Screening (up to 35 days prior to Day 0) | Day 0 | 7 ± 1 days | 28 ± 7days | 56 ± 7 days | 70 ± 7 days | 84 ± 7 days | 112 ± 7days | 140 ± 7days | 168 ± 7days | 196± 7days | 224 ± 7days | 252 ± 7days | 280 ± 7days | 308 ± 7days | 336 ± 7days | 364 ± 7days | General<br>follow<br>up<br>period <sup>1</sup> | Individualized<br>follow up<br>period (IFU) <sup>6</sup> | l IFU<br>Final<br>Visit |
| Study Week | W -5 | | W1 | W4 | W8 | W10 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44 | W48 | W52 | W68 | | |
| Monitor in clinic after dosing for 1h post rituximab/placebo | | | | | Χ | Χ | | | | | | | | | | | | | | |
| Efficacy, pharmacokinetics and p | harmac | odyna | mics | | | | | | | | | | | | | | | | | |
| ESSDAI <sup>16</sup> | Х | | | | | | Χ | | | Χ | | | Χ | | | | Χ | Χ | | Х |
| ESSPRI | Х | | | | | | Χ | | | Χ | | | Χ | | | | Χ | Χ | | Х |
| Oral Dryness numerical resp. scale | Х | | | | | | Χ | | | Χ | | | Χ | | | | Χ | Χ | | Х |
| Ocular Dryness numerical resp. scale | Х | | | | | | Χ | | | Χ | | | Χ | | | | Χ | Χ | | Х |
| Salivary gland biopsy | χ5 | | | | | | | | | X12 | | | | | | | X13 | | | |
| Lacrimal function (Schirmer's) test | Х | | | | | | Χ | | | Χ | | | Χ | | | | Χ | | | |
| Fatigue- (PROFAD SSI SF) | Х | | | | | | | | | Χ | | | Χ | | | | Χ | | | |
| Patient Global Assessment (PtGA) | Х | | | | | | | | | Χ | | | Χ | | | | Χ | | | |
| Physicians Global Assessment (PGA) | Х | | | | | | | | | Χ | | | Χ | | | | Χ | | | |
| Exit interview | | | | | | | | | | | | | | | | | Χ | | | |
| Stimulated Salivary Flow | Χ | | | | | | Χ | | | Χ | | | Χ | | | | Χ | Χ | | Х |
| Unstimulated Salivary Flow | Χ | | | | | | Χ | | | Χ | | | Χ | | | | Χ | Χ | | Х |
| Blood: Leukocyte population <sup>2</sup> | Χ | X <sub>3</sub> | Χ | Χ | Χ | | Χ | | | Χ | Χ | | Χ | | Χ | | Χ | Χ | Χ | Χ |
| Serological biomarkers | Χ | X3 | | | Χ | | Χ | Χ | | Χ | Χ | | Χ | | Χ | | Χ | Χ | Χ | Χ |
| Saliva sample for proteomics | Χ | | | | | | Χ | | | Χ | | | Χ | | | | Χ | | | |
| Blood: BLyS levels <sup>2</sup> | | Χ3 | | Χ | Χ | | Χ | Χ | | Χ | Χ | | Χ | | Χ | | Χ | Χ | | Х |
| Blood: Transcriptomics | | Хз | | | Χ | | | | | Χ | | | Χ | | | | Χ | | | |
| Salivary gland: Transcriptomics | Χ | | | | | | | | | Χ | | | | | | | Χ13 | | | |
| Blood: PBMC exploratory endpoints | | Хз | | | Χ | | | | | Χ | | | | | | | | | | |

2020N437857\_00 201842

| | or<br>or | | | | | | Dοι | ıble B | lind Ti | reatme | ent Pei | riod | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day | Screening (up to 35 days prior to Day 0) | Day 0 | 7 ± 1 days | 28 ± 7days | 56 ± 7 days | 70 ± 7 days | 84 ± 7 days | 112 ± 7days | 140 ± 7days | 168 ± 7days | 196± 7days | 224 ± 7days | 252 ± 7days | 280 ± 7days | 308 ± 7days | 336 ± 7days | 364 ± 7days | General<br>follow<br>up<br>period <sup>1</sup> | Individualized<br>follow up<br>period (IFU) <sup>6</sup> | I IFU<br>Final<br>Visit |
| Study Week | W -5 | | W1 | W4 | W8 | W10 | W12 | W16 | W20 | W24 | W28 | W32 | W36 | W40 | W44 | W48 | W52 | W68 | | |
| Blood: Belimumab PK <sup>2</sup> | | | | | | | | | | Χ | | | Х | | Χ | | Χ | | | |
| Blood: Rituximab PK <sup>2</sup> | | | | | Χ7 | Χ7 | Χ | | | Х | | | Х | | | | | | | |
| Safety & Laboratory Assessments | | | | | | | | | | | | | | | | | | | | |
| AE/SAE review | X <sup>17</sup> | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | X18 | Χ |
| Vital signs | Χ | X3,4 | X <sup>4</sup> | Χ | X <sup>4</sup> | X <sup>4</sup> | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х |
| 12-lead ECG | Χ | | | | | | | | | | | | | | | | | | | |
| CSSRS (suicidality assessment) | | X <sub>3</sub> | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | |
| Neurological assessment | | X <sub>3</sub> | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ |
| Urinalysis | Χ | X3 | | | | | Χ | | | Χ | | | Χ | | | | Χ | Х | | Х |
| Blood: Immunoglobulin levels (IgG, IgA², IgM²) | Χ | Х3 | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Х | Χ | Х | X | Х |
| Blood: Cryoglobulins | Χ | | | | | | Χ | | | Χ | | | Χ | | | | Χ | Χ | | Х |
| Blood chemistry | Χ | X3 | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х |
| Hematology | Χ | X <sub>3</sub> | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х |
| HIV, Hep B and Hep C screen | X14 | | | | | | | | | | | | | | | | | Χ | | |
| Pharmacogenetics blood sample <sup>15</sup> | | Χ | | | | | | | | | | | | | | | | | | |
| Blood: Belimumab Immunogenicity <sup>2</sup> | | Хз | | | Χ | | | | | Χ | | | | | | | Χ | Χ | | |
| Blood: Rituximab Immunogenicity² | | | | | X <sub>3</sub> | | | | | Χ | | | | | | | Χ | | | |

<sup>1.</sup> All subjects, including subjects who are withdrawn from the study and decline to complete the treatment phase visits through Week 52, are required to enter the general follow up period. During this 16-week general follow up period, subjects will receive calls every 4 weeks (±7 days) to evaluate AEs, to check concomitant medications and to complete the neurological assessment.

<sup>2.</sup> In order to maintain the blind, sites will be blinded to these data following screening - including B-cell flow cytometry panels and IgA, IgM levels.

2020N437857\_00 201842

- 3. To be measured or collected pre-dose.
- 4. Subjects will be monitored post study treatment as detailed in protocol.
- 5. Biopsy can occur on Day 0 or at any time during the screening period provided the subject has met all other entry criteria prior to the biopsy.
- 6. Subjects will enter the IFU if, following the general follow up period, their CD19+ B-cell levels remain below the lower limit of normal (or less than 90% of baseline, if baseline value was below LLN). During the IFU, subjects will be seen in the clinic every 12 weeks (± 7 days), with calls every 4 weeks (±7 days) between visits to evaluate subjects for AEs & concomitant medications. Subjects will exit the IFU when: CD19+ B-lymphocyte counts are within normal range or 10% of baseline levels (if baseline < LLN), OR at the investigator's discretion the subject starts receiving disease modifying therapy that may affect B-cell numbers OR or for up to a maximum of 2 years (i.e., up to Week 104) whichever comes first. Subjects exiting IFU period will attend a final visit (within 28 days of that decision) for final assessments (IFU Final Visit) as detailed in the Table.
- 7. Obtain samples post-dose only, within 10 minutes after end of infusion.
- 8. Both doses of rituximab/placebo will be administered in the clinic. Approximately 60 minutes prior to rituximab/placebo, subjects will receive orally an antipyretic and an antihistamine. At least 30 minutes prior to administration of rituximab/placebo, subjects will receive IV 100mg methylprednisilone. The 2nd rituximab/placebo administration at the Week10 visit must be given 14 days (13-18 days, see SRM) after the first administration (given at the Week 8 visit). A patient alert card should be sent home with the subject following each dose of rituximab/placebo.
- 9. If urine test is positive, confirm with serum test. Pregnancy testing & contraception are required until 16 weeks post last administration of study treatment for those subjects who complete Weeks 46- 52 or withdraw from treatment prior to Week 8 dosing. Pregnancy testing and contraception are required for approximately 12 months after the administration of the final rituximab/placebo dose for the subset of subjects who discontinue treatment from Week 8 up to Week 46.
- 10. Subjects will receive a reminder phone call 48 hours prior to efficacy assessment visits to remind them that they should not be using certain symptomatic therapies prior to visit (see Section 4.1 of Study Reference Manual for details); in addition subjects should document their last use of symptomatic therapies in their self injection log book.
- 11. First & second dose of belimumab will be administered in clinic by subject or caregiver. A patient alert card will be sent home with the subject each time belimumab is dispensed for home administration.
- 12. Week 24 biopsy may be taken on a separate day from the other required assessments within the Week 24 study visit window.
- 13. Week 52 biopsy is optional. Trancriptomics will only be performed if biopsy is taken.
- 14. If test otherwise performed within 3 months prior to first dose of study treatment, testing at screening is not required.
- 15. Informed consent for optional substudies e.g., genetics must be obtained before collecting a sample.
- 16. If additional tests (e.g., pulmonary function tests, EMG, MRI) are required to complete ESSDAI assessment, these should be scheduled as close as possible to the stipulated study visit window.
- 17. From signing of consent until initiation of study treatment, only SAEs related to study participation will be collected.
- 18. From the end of general follow-up phase through the last contact (including the individualized safety follow-up phase), only designated AESIs (i.e., infections, malignancies, and depression/suicidality/self-injury), fatal SAEs, and SAEs assessed as related to the investigational product or to study participation will be collected.

## 11.3. Appendix 3: Treatment States and Phases

#### 11.3.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to study treatment, unless otherwise specified.

| Treatment Phase | Definition |
|-----------------|----------------------------------------------------|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Last Dose + 28 |
| Post-Treatment | Date > Last Dose + 28 |

#### 11.3.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the date of first and/or last dose of study treatment.

#### 11.3.2.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & up to 28 days after date of last dose. |
| | Study Treatment Start Date ≤ AE Start Date ≤ [Last Dose Study Treatment + 28] |
| Post-Treatment | If AE onset date is > 28 days after the last dose of study drug. |
| | AE Start Date >[ Last Dose Study Treatment + 28] |
| Onset Time | If Treatment Start Date > AE Onset Date = AE Onset Date - Treatment Start Date |
| Since 1st Dose | If Treatment Start Date ≤ AE Onset Date = AE Onset Date - Treatment Start Date +1 |
| (Days) | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on Inform/CRF OR value is missing. |

#### NOTES:

o If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

## 11.4. Appendix 4: Data Display Standards & Handling Conventions

#### 11.4.1. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently support to the currently su | The currently supported versions of SAS software will be used. |
| Reporting Area (Interim) | |
| HARP Server : US1SALX00259 | |
| HARP Area : \ARPROD\GSK1550188\MID201842\Interim_01 | |
| Reporting Area (Primary Analysis) | |
| HARP Server : US1SALX00259 | |
| HARP Area : \ARPROD\GSK1550188\MID201842\Primary_02 | |
| NOTE: | |
| <ul> <li>Primary_01 has</li> </ul> | been taken for previous CDISC reporting and hence not available |
| Reporting Area (En | d of Study Analysis) |
| HARP Server | : US1SALX00259 |
| HARP Area : \ARPROD\GSK1550188\MID201842\Final_02 | |
| Analysis Datasets | |
| Analysis datasets | Analysis datasets will be created according to IDSL standards |
| Generation of RTF I | Generation of RTF Files |
| RTF files will be g | generated at primary and end of study analysis |
| XML files in the format expected by DORS (Disclosure Obligation Reporting System) for | |

#### **Reporting Standards**

relevant displays

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected with a maximum of 4 DP presented.
- Numeric data will be reported at the precision collected on the eCRF.
   The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Reporting Standards**

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Data will be incorporated in figures, summaries and statistical analyses using the visit recorded in eCRF. No visit slotting is planned.

#### **Unscheduled Visits**

- Unscheduled visits will not be presented in summary tables or figures, with the exception of any time post baseline/worst toxicities where all data including unscheduled visits are used in derivations.
- All unscheduled visits will be included in listings.

| 7 Till drischeduled visits will be included in listings. | |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data | Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data N, n, frequency, % | |
| Reporting of Pharmacokinetic Concentration Data | |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Graphical Displays | |
| Refer to IDSL Sta | Refer to IDSL Statistical Principals 7.01 to 7.13. |
| • Include ref line (i | <ul> <li>Include ref line (i.e. y=0) for figures having negative values</li> </ul> |

## 11.5. Appendix 5: Derived and Transformed Data

#### 11.5.1. General

## **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target, then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from randomization date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomization Date → Study Day = Ref Date Randomization Date
  - Ref Data ≥ Randomization Date → Study Day = Ref Date (Randomization Date) + 1

#### **Data Cutt-off**

- The study data cut-off date of the primary analysis is September 9<sup>th</sup>, 2019. Data after September 9<sup>th</sup> will be removed from the extracted data after October 30<sup>th</sup> based on the algorithms detailed below.
- The data cut off will be applied on DMDATA before the generating of any analysis datasets and outputs.

| Datasets | Label | Algorithm |
|---|---|---|
| AE | ADVERSE EVENT | AESTDT <= CUTOFF DATE |
| BIOLINK | BIOMARKER SAMPLE | BIDT <= CUTOFF DATE |
| BIOMARK | BIOMARKER | BIDT <= CUTOFF DATE |
| BLIND | BLIND | BLDT <= CUTOFF DATE |
| CC | EULAR SJOGRENS SYNDROME DISEASE ACTIVITY INDEX | CCDT <= CUTOFF DATE |
| CE | CV CLINICAL EVENTS | CESTDT <= CUTOFF DATE |
| CHDPOT | PREGNANCY INFORMATION | IMPUTED CHDMNFD_, THEN THE IMPUTED DATE <= CUTOFF DATE |
| CONMEDS | CONCOMITANT MEDICATIONS | IMPUTED CMSTD_, THEN THE IMPUTED DATE <= CUTOFF DATE |
| CONV | LAB CONVERSION FACTOR | NOT CUT |
| CSSRSV4 | COLUMBIA SUICIDE SEVERITY RATING SCALE | ACTDT <= CUTOFF DATE |
| CVDXTEST | CEREBROVASCULAR EVENTS | DXDT <= CUTOFF DATE |
| DEMO | DEMOGRAPH | NOT CUT |
| DS | STUDY CONCLUSION | DSSTDT <= CUTOFF DATE |
| DTH | DEATH | DDDT <= CUTOFF DATE |
| DV1 | PROTOCOL DEVIATION | DVSTDT <= CUTOFF DATE |
| ECG | 12-LEAD ECG | EGDT <= CUTOFF DATE |
| EGCRIT | ECG REFERENCE DATA | NOT CUT |

| Datasets | Label | Algorithm |
|---|---|---|
| ELIG | ELIGIBILIT | NOT CUT |
| ENROL | INFORM ENROLLMENT | NOT CUT |
| ESSPRI | EULAR SJOGRENS SYNDROME<br>PATIENT REPORTED INDEX | ACTDT <= CUTOFF DATE |
| EVIDENCE | DEEP VEIN THROMBOSIS (DVT) /PULMONARY EMBOLISM (PE) | NOT CUT |
| EXPOSURE | STUDY TREATMENT | FIRST GET THE LARGEST VISITNUM FROM VISIT DATA WHERE VISITDT <= CUTOFF DATE; LEFT JOIN EXPOSURE WITH THE VISIT DATA BY SUBJID; VISITNUM FROM STATUS <= THE LARGEST VISITNUM FROM VISIT DATA WHERE EXSTDT IS MISSING OR EXSTDT <= CUTOFF DATE WHERE SSDT IS NOT MISSING. |
| FACE | NEUROLOGICAL SYMPTOMS QUESTIONNAIRE | FCEDT <= CUTOFF DATE |
| FACV | FINDING ABOUT CLINICAL EVENTS | NOT CUT |
| FADE | INVESTIGATIONAL PRODUCT DEVICE MALFUNCTION (DEV MALFUNCTION) | FDEDT <= CUTOFF DATE |
| FADTH | FINDINGS ABOUT DEATH | DDORRSDT <= CUTOFF DATE |
| FAMH | FINDING ABOUT METICAL<br>HISTORY | NOT CUT |
| FAMHIST | FAMILY HISTORY | NOT CUT |
| FAPR | UNSTIMULATED AND<br>STIMULATED SALIVARY FLOW | FPRDT <= CUTOFF DATE |
| GENPRO | PHARMACOGENETIC (PGx) RESEARCH CONSENT | GPSMPDT <= CUTOFF DATE |
| HRU | HOSPITALISATION | HUHOSTDT <= CUTOFF DATE |
| IMGEN | IMMUNOGENICITY | IGDT <= CUTOFF DATE |
| IMGLINK | IMMUNOGENICITY SAMPLING | IGDT <= CUTOFF DATE |
| INVESTIG | INVESTIGATOR SIGNATUR | NOT CUT |
| IPDISC | STUDY TREATMENT DISCONTINUATION | SDENDT <= CUTOFF DATE |
| LAB | LABORATORY TEST | LBDT < = CUTOFF DATE |
| LABCRIT | LAB REFERENCE DATA | NOT CUT |
| LBIOPSY | LIVER BIOPSY (BIOPSY) | LPDT < = CUTOFF DATE |
| LBTESTCD | LAB TEST CODES | NOT CUT |
| LEREPORT | LIVER MONITORING/STOPPING<br>EVENT REPORTING (LEREPORT) | LERSTDT < = CUTOFF DATE |
| LIMAGING | LIVER IMAGING (IMAGING) | LIDT <= CUTOFF DATE |
| MEDHIST | SJOGRENS SYNDROME SPECIFIC MEDICAL HISTORY | NOT CUT |
| MI | MICROSCOPIC FINDINGS | GET THE LARGEST VISITNUM FROM VISIT DATA WHERE VISITDT <= CUTOFF DATE; LEFT JOIN MI WITH THE VISIT DATA BY SUBJID; VISITNUM FROM MI < = THE LARGEST VISITNUM FROM VISIT DATA |
| MO | MORPHOLOGY | MODT <= CUTOFF DATE |
| NYHASCR | NYHA SCORE | NOT CUT |
| OCULAR | LACRIMAL FUNCTION (SCHIRMERS) TEST | XGDT <= CUTOFF DATE |
| OROCNRS | ORAL AND OCULAR DRYNESS NUMERIC RATING SCAL | ACTDT < = CUTOFF DATE |

| Datasets | Label | Algorithm |
|---|---|---|
| PFDSSISF | PROFILE OF FATIGUE AND DISCOMFORT - SICCA SYMPTOMS INVENTORY | ACTDT < = CUTOFF DATE |
| PHGA | PHYSICIAN GLOBAL ASSESSMENT OF DISEASE ACTIVITY | ACTDT < = CUTOFF DATE |
| PK | PK BLOOD SAMPLE COLLECTION;<br>PHARMACOKINETICS | PKSTDT < = CUTOFF DATE |
| PR | SCHIRMERS TEST SATURATION PROCEDURE | PRSTDT < = CUTOFF DATE |
| PSRAE | POSSIBLE SUICIDE RELATED ADVERSE EVENT QUESTION | AESTDT < = CUTOFF DATE |
| PSRAECO<br>M | POSSIBLE SUICIDE RELATED ADVERSE EVENT QUESTION COMMENT | NOT CUT |
| PTGA | PATIENT GLOBAL ASSESSMENT OF DISEASE ACTIVITY | ACTDT < = CUTOFF DATE |
| RACE | COLLECTED RACE | NOT CUT |
| RAND | RANDOMISATION | NOT CUT |
| RANDALL | RANDOMISED TREATMENT | NOT CUT |
| RISK | MEDICAL DEVICE | NOT CUT |
| RUCAM | LIVER EVENTS (LIVER EVENTS) | RUDT < = CUTOFF DATE |
| SS | SYMPTOMATIC THERAPY US | FIRST GET THE LARGEST VISITNUM FROM VISIT DATA WHERE VISITDT <= CUTOFF DATE; LEFT JOIN SS WITH THE VISIT DATA BY SUBJID; VISITNUM FROM STATUS <= THE LARGEST VIISTNUM FROM VISIT DATA WHERE SSDT IS MISSING OR SSDT <= CUTOFF DATE WHERE SSDT IS NOT MISSING. |
| STATUS | VISIT STATUS | GET THE LARGEST VISITNUM FROM VISIT DATA WHERE VISITDT <= CUTOFF DATE; LEFT JOIN STATUS WITH THE VISIT DATA BY SUBJID; VISITNUM FROM STATUS <= THE LARGEST VISITNUM FROM VISIT DATA |
| SUBUSE | HISTORY OF TOBACCO USE | NOT CUT |
| SURGERY | CEREBROVASCULAR SURGERY | SPDT < = CUTOFF DATE |
| TMSLICE | VISIT AND PERIOD | NOT CUT |
| VISIT | VISIT | VISITDT < = CUTOFF DATE |
| VITALS | VITAL SIGNS | VSDT < = CUTOFF DATE |
| VSCRIT | VITAL SIGNS REFERENCE DATA | NOT CUT |
| VIRAL | VIRAL LABORATORY RESULTS | LABDT < = CUTOFF DATE |

#### 11.5.2. Study Population

## Subject Disposition Status - Primary Analysis

## Study Completion Status at Week 68

A subject is considered **Completed** at Week 68 if **BOTH** of the following conditions are met:

- The study treatment is not stopped permanently before the scheduled end of the treatment period
- Subject completed Week 68 visit
- A subject is considered Ongoing at Week 68 if ALL of the following conditions are met:
  - The study treatment is not stopped permanently before the scheduled end of the treatment period subject has not completed Week 68 visit
  - Date of subject completion or withdrawal is missing
- A subject is considered **Withdrawn** at Week 68 if **EITHER** of the following conditions is met:
  - The study treatment is stopped permanently before the scheduled end of the treatment period
  - The study treatment is not stopped permanently before the scheduled end of the treatment period, but subject was withdrawn prior to Week 68

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - 1. Any subject with a missing day will have this imputed as day '15'.
  - 2. Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

#### **Extent of Exposure to Belimumab**

Number of days of exposure to belimumab will be calculated as:

## Duration of Exposure in Days = Date of Last Belimumab Injection – Date of First Belimumab Injection + 7

 Subjects who were randomized but did not report a treatment start date will be categorized as having zero days of exposure.

#### **Baseline Characteristics**

#### **Autoantibodies**

- SS-A positive subjects are defined as those who have screening SS-A ≥ 7 KU/L.
- SS-B positive subjects are defined as those who have screening SS-B ≥ 7 KU/L

#### **Extent of Exposure to Belimumab**

#### **Time Since Diagnosis**

Time since diagnosis of Primary Sjogren Syndrome is defined as:

• If treatment start date >= diagnosis date and then treatment start date - diagnosis date

- If the day and month of diagnosis is missing, this will be imputed as '30th June'
- If the year of diagnosis is missing, time since diagnosis will be set to missing

#### **Average Daily Prednisone Dose**

 At baseline, the average daily dose of prednisone is the sum of doses over 7 consecutive days up to, but not including Day 0 divided by 7: Days on which a subject does not have prednisone use recorded will be considered as 0 mg for the day in the calculation of average daily prednisone dose.

#### 11.5.3. Safety

#### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, unless otherwise specified the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - 1. Example 1: 2 Significant Digits = '< x' becomes x 0.01
  - 2. Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - 3. Example 3: 0 Significant Digits = '< x' becomes x − 1

Details of rules to apply for biomarker endpoints are covered in Section 11.5.6.

#### **Neurological Symptoms**

- Neurological systems are assessed based upon a questionnaire consisting of 7 questions with response of either yes or no.
- See Appendix 11 for further information.

#### Suicidal Risk Monitoring

## Columbia Suicidality Severity Rating Scale (C-SSRS)

- The C-SSRS is a measure of suicidal ideation and behavior.
- The following outcomes are C-SSRS categories and have binary responses (yes/no). The categories have been re-ordered from the actual scale in an increasing order of severity from 1 to 10 to facilitate the definitions of the comparative endpoints.
  - Category 1 CCI This sector indices, where the control of
  - Category 2 excluded.
  - Category 3 –
  - Category 4 –
  - Category 5 –
  - Category 6 –
  - Category 7 –
  - Category 8 –
  - Category 9 –
  - Category 10
- The following outcomes are numerical scores derived from the C-SSRS categories. The scores are created at each assessment for each patient.
  - Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C-SSRS) present at the assessment. Assign a score of 0 if no ideation is present.
  - Suicidal Behavior Score: The maximum suicidal behavior category (6-10 on the C-SSRS) present at the assessment. Assign a score of 0 if no behavior is present.
  - Suicidal Ideation or Behavior Score: The maximum suicidal ideation or behavior category (1-10 on the C-SSRS) present at the assessment. Assign a score of 0 if no ideation or behavior is present.
- See Appendix 11 for further details.

#### 11.5.3.1. **Adverse Events of Special Interest**

#### Handling Study specific AESI:

- GSK study statistician will generate cumulative spreadsheets in .csv format which is created by merging DMDATA.AE with MedDRA dictionary by preferred terms corresponding to study specific AESI SMQ's extracted from latest version of MedDRA, as specified in the below table.
- GSK study statistician will distribute spreadsheets via e-mail to the study team for clinical review.
- GSK study statistician will receive returned spreadsheets. A manual review will be performed so that any noted quality issues can be followed up.
  - GSK study statistician will create csv versions in the "Adjudicated" folder on arwork (\\us1salx00259.corpnet2.com\arenv\arwork\gsk1550188\refdata\aesi\Adjudication Results\MID201842\Adjudicated).

Study Specific Primary Analysis AESI specification to be capture in the process. For the End of Study Analyses, PTs related the MedDRA version at the time of database release will be used. If a new version of MedDRA is used, then a RAP amendment or addendum will be created to capture updated PTs.

## **End of Study Reporting**

MedDRA 23.0 PTs will be used. This is a major version release that includes changes to any level of the hierarchy and additionally includes COVID-19 related terminology. On this basis the RAP will not be updated, instead MedDRA V23.0 will be implemented. Same search Strategy will be applied to MedDRA V23.0.

| Category: Severe skin reaction per GSK Adjudication (Ten and Steven's Johnson Syndrome) | |
|---|---|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| Broad Search: Severe Cutaneous | Acquired epidermolysis bullosa |
| Adverse Reactions SMQ. | Blister |
| | Blister rupture |
| | Bullous impetigo |
| | Conjunctivitis |
| | Corneal exfoliation |
| | Drug eruption |
| | Epidermolysis |
| | Epidermolysis bullosa |
| | Fixed eruption |
| | Genital ulceration |
| | HLA-B*1502 assay positive |
| | HLA-B*5801 assay positive |
| | Hypopharyngeal synechiae |
| | Lip exfoliation |
| | Mouth ulceration |
| | Mucocutaneous ulceration |
| | Mucosa vesicle |
| | Mucosal erosion |
| | Mucosal exfoliation |
| | Mucosal necrosis |
| | Mucosal ulceration |
| | Nasal mucosal blistering |
| | Nikolsky's sign |
| | Noninfective conjunctivitis |
| | Oral mucosal blistering |
| | Oral mucosal exfoliation |
| | Oral papule |
| | Oropharyngeal blistering |
| | Pemphigoid |

| Category: Severe skin reaction per GSK Adjudication (Ten and Steven's Johnson Syndrome) | |
|---|---|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| | Pemphigus |
| | Penile exfoliation |
| | Skin erosion |
| | Skin exfoliation |
| | Staphylococcal scalded skin syndrome |
| | Stomatitis |
| | Symmetrical drug-related intertriginous and flexural exanthema |
| | Tongue exfoliation |
| | Vaginal exfoliation |
| | Vaginal ulceration |
| | Vulval ulceration |
| | Vulvovaginal rash |
| | Vulvovaginal ulceration |

| Category: Cardiac Disorders | |
|---|---|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| <b>Broad Search:</b> Cardiac Arrhythmias SMQ | Sub-Category: Arrhythmia related investigations, signs and |
| | symptoms (SMQ) |
| | Bezold-Jarisch reflex |
| | Bradycardia |
| | Cardiac arrest |
| | Cardiac death |
| | Cardiac telemetry abnormal |
| | Cardio-respiratory arrest |
| | Central bradycardia |
| | Electrocardiogram abnormal |
| | Electrocardiogram ambulatory abnormal |
| | Electrocardiogram change |
| | Heart rate abnormal |
| | Heart rate decreased |
| | Heart rate increased |
| | Loss of consciousness |
| | Palpitations |
| | Rebound tachycardia |
| | Respiratory sinus arrhythmia magnitude abnormal |
| | Respiratory sinus arrhythmia magnitude decreased |
| | Respiratory sinus arrhythmia magnitude increased |
| | Sudden death |
| | Syncope |
| | Tachycardia |

| Category: Cardiac Disorders | |
|---|---|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| | Tachycardia paroxysmal |
| | Sub-Category: Cardiac arrhythmia terms (incl bradyarrhythmias |
| | and tachyarrhythmias) (SMQ) -NIL- |
| | Sub-Category: Tachyarrhythmias (incl supraventricular and |
| | ventricular tachyarrhythmias) (SMQ) |
| | -NIL- |
| | Sub-Category: Supraventricular tachyarrhythmias (SMQ) |
| | ECG P wave inverted |
| | Electrocardiogram P wave abnormal |
| | Retrograde p-waves |
| Broad Search: Congenital and | Baseline foetal heart rate variability disorder |
| neonatal arrhythmias (SMQ) | Bradycardia foetal |
| | Bradycardia neonatal |
| | Cardiac arrest neonatal |
| | Cardio-respiratory arrest neonatal |
| | Foetal heart rate acceleration abnormality |
| | Foetal heart rate deceleration abnormality |
| | Neonatal sinus bradycardia |
| | Neonatal sinus tachycardia |
| | Neonatal tachycardia |
| | Nonreassuring foetal heart rate pattern |
| | Tachycardia foetal |
| | Nonreassuring foetal heart rate pattern |
| | Tachycardia foetal |
| Broad Search: Cardiac Failure SMQ | Artificial heart implant |
| | Atrial natriuretic peptide abnormal |
| | Atrial natriuretic peptide increased |
| | Bendopnoea |
| | Brain natriuretic peptide abnormal |
| | Brain natriuretic peptide increased |
| | Cardiac cirrhosis |
| | Cardiac contractility modulation therapy |
| | Cardiac device reprogramming |
| | Cardiac dysfunction |
| | Cardiac index decreased |
| | Cardiac output decreased |
| | Caralac output accircasca |
| | Cardiac resynchronisation therapy |
| | · |
| | Cardiac resynchronisation therapy |

| earch Strategy | MedDRA 22.0 PTs Included in SMQ |
|----------------|-----------------------------------------------------------|
| | Cardiomegaly |
| | Cardio-respiratory distress |
| | Cardiothoracic ratio increased |
| | Central venous pressure increased |
| | Diastolic dysfunction |
| | Dilatation ventricular |
| | Dyspnoea paroxysmal nocturnal |
| | Heart transplant |
| | Hepatic vein dilatation |
| | Implantable cardiac monitor replacement |
| | Intracardiac pressure increased |
| | Jugular vein distension |
| | Left ventricular diastolic collapse |
| | Left ventricular dilatation |
| | Left ventricular dysfunction |
| | Left ventricular enlargement |
| | Lower respiratory tract congestion |
| | Myocardial depression |
| | Nocturnal dyspnoea |
| | N-terminal prohormone brain natriuretic peptide abnormal |
| | N-terminal prohormone brain natriuretic peptide increased |
| | Oedema |
| | Oedema blister |
| | Oedema due to cardiac disease |
| | Oedema neonatal |
| | Oedema peripheral |
| | Orthopnoea |
| | Peripheral oedema neonatal |
| | Peripheral swelling |
| | Post cardiac arrest syndrome |
| | Prohormone brain natriuretic peptide abnormal |
| | Prohormone brain natriuretic peptide increased |
| | Pulmonary congestion |
| | Right ventricular diastolic collapse |
| | Right ventricular dilatation |
| | Right ventricular dysfunction |
| | Right ventricular enlargement |
| | Scan myocardial perfusion abnormal |
| | Stroke volume decreased |
| | Surgical ventricular restoration |

| Category: Cardiac Disorders | MadDDA 22 0 DTa Institute 4 to 2MO |
|------------------------------|-------------------------------------------|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| | Systolic dysfunction |
| | Venous pressure increased |
| | Venous pressure jugular abnormal |
| | Venous pressure jugular increased |
| | Ventricular assist device insertion |
| | Ventricular compliance decreased |
| | Ventricular dysfunction |
| | Ventricular dyssynchrony |
| | Wall motion score index abnormal |
| Broad Search: Cardiomyopathy | Abnormal precordial movement |
| SMQ | Acquired cardiac septal defect |
| | Acute left ventricular failure |
| | Alcohol septal ablation |
| | Arrhythmia |
| | Arrhythmia supraventricular |
| | Artificial heart implant |
| | Ascites |
| | Atrial enlargement |
| | Atrial hypertrophy |
| | Atrial pressure increased |
| | Autoimmune myocarditis |
| | Bendopnoea |
| | Blood pressure diastolic abnormal |
| | Blood pressure diastolic decreased |
| | Blood pressure diastolic increased |
| | Blood pressure fluctuation |
| | Blood pressure inadequately controlled |
| | Blood pressure systolic abnormal |
| | Blood pressure systolic decreased |
| | Blood pressure systolic increased |
| | Cardiac aneurysm |
| | Cardiac arrest |
| | Cardiac contractility modulation therapy |
| | Cardiac device reprogramming |
| | Cardiac dysfunction |
| | Cardiac electrophysiologic study abnormal |
| | Cardiac failure |
| | Cardiac failure acute |
| | Cardiac failure chronic |
| | Cardiac failure congestive |

| Category: Cardiac Disorde<br>Search Strategy | MedDRA 22.0 PTs Included in SMQ |
|---|---|
| · | Cardiac function test abnormal |
| | Cardiac imaging procedure abnormal |
| | Cardiac index abnormal |
| | Cardiac index decreased |
| | Cardiac index increased |
| | Cardiac monitoring abnormal |
| | Cardiac operation |
| | Cardiac output decreased |
| | Cardiac pseudoaneurysm |
| | Cardiac resynchronisation therapy |
| | Cardiac ventricular scarring |
| | Cardiac ventriculogram abnormal |
| | Cardiac ventriculogram left abnormal |
| | Cardiac ventriculogram right abnormal |
| | Cardiomegaly |
| | Cardiothoracic ratio increased |
| | Cardiovascular disorder |
| | Cardiovascular function test abnormal |
| | Chest pain |
| | Chest X-ray abnormal |
| | Computerised tomogram thorax abnormal |
| | Coxsackie carditis |
| | Coxsackie myocarditis |
| | Cytomegalovirus myocarditis |
| | Decreased ventricular preload |
| | Diastolic dysfunction |
| | Dilatation atrial |
| | Dilatation ventricular |
| | Directional Doppler flow tests abnormal |
| | Dyspnoea |
| | ECG signs of ventricular hypertrophy |
| | Echocardiogram abnormal |
| | Electrocardiogram abnormal |
| | Electrocardiogram change |
| | Electrocardiogram PR segment depression |
| | Electrocardiogram U wave inversion |
| | Endocardial fibroelastosis |
| | External counterpulsation |
| | Gonococcal heart disease |
| | Heart and lung transplant |

| Category: Cardiac Disorder<br>Search Strategy | MedDRA 22.0 PTs Included in SMQ |
|---|---|
| | Heart transplant |
| | Hepatomegaly |
| | Hyperdynamic left ventricle |
| | Hypersensitivity myocarditis |
| | Implantable cardiac monitor replacement |
| | Increased ventricular preload |
| | Intracardiac pressure increased |
| | Irregular breathing |
| | Labile blood pressure |
| | Left atrial dilatation |
| | Left atrial enlargement |
| | Left atrial volume abnormal |
| | Left atrial volume decreased |
| | Left atrial volume increased |
| | Left ventricular dilatation |
| | Left ventricular dysfunction |
| | Left ventricular end-diastolic pressure decreased |
| | Left ventricular enlargement |
| | Left ventricular failure |
| | Left ventricular heave |
| | Lupus myocarditis |
| | Lyme carditis |
| | Malarial myocarditis |
| | Mental status changes |
| | Multiple gated acquisition scan abnormal |
| | Myocardiac abscess |
| | Myocardial necrosis marker increased |
| | Myocarditis |
| | Myocarditis bacterial |
| | Myocarditis helminthic |
| | Myocarditis infectious |
| | Myocarditis meningococcal |
| | Myocarditis mycotic |
| | Myocarditis post infection |
| | Myocarditis septic |
| | Myocarditis syphilitic |
| | Myocarditis toxoplasmal |
| | Myoglobinaemia |
| | Myoglobinuria |
| | Nocturia |

| | | 201842 |
|---|---|---|
| Category: Cardiac Disorders | | |
| Search Strategy | MedDRA 22.0 PTs Included in SMQ | |
| Search Strategy | Nuclear magnetic resonance imaging thoracic abnormal | |
| | Oedema | |
| | Orthostatic hypotension | |
| | Palpitations | |
| | Papillary muscle disorder | |
| | Papillary muscle haemorrhage | |
| | Radiation myocarditis | |
| | Right atrial dilatation | |
| | Right atrial enlargement | |
| | Right atrial pressure increased | |
| | Right ventricle outflow tract obstruction | |
| | Right ventricular dilatation | |
| | Right ventricular enlargement | |
| | Right ventricular heave | |
| | Right ventricular systolic pressure decreased | |
| | Scan myocardial perfusion abnormal | |
| | Sudden cardiac death | |
| | Sudden death | |
| | Surgical ventricular restoration | |
| | Syncope | |
| | Systolic anterior motion of mitral valve | |
| | Systolic dysfunction | |
| | Ultrasound Doppler abnormal | |
| | Vascular resistance pulmonary increased | |
| | Ventricular arrhythmia | |
| | Ventricular assist device insertion | |
| | Ventricular dysfunction | |
| | Ventricular dyskinesia | |
| | Ventricular dyssynchrony | |
| | Ventricular enlargement | |
| | Ventricular hyperkinesia | |
| | Ventricular hypertrophy | |
| | Ventricular hypokinesia | |
| | Ventricular remodelling | |
| | Viral myocarditis | |
| | Wall motion score index abnormal | |
| | Wall motion score index abnormal | |
| Broad Search: Ischaemic heart | Sub-Category: Myocardial infarction (SMQ) | |
| disease SMQ | . , , | |
| | Blood creatine phosphokinase abnormal | |

Blood creatine phosphokinase abnormal Blood creatine phosphokinase increased

| Category: Cardiac Disorders | |
|---|---|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| | Cardiac ventricular scarring |
| | ECG electrically inactive area |
| | ECG signs of myocardial infarction |
| | Electrocardiogram Q wave abnormal |
| | Electrocardiogram ST segment abnormal |
| | Electrocardiogram ST segment elevation |
| | Electrocardiogram ST-T segment elevation |
| | Electrocardiogram U wave inversion |
| | Infarction |
| | Myocardial necrosis marker increased |
| | Scan myocardial perfusion abnormal |
| | Vascular graft occlusion |
| | Vascular stent occlusion |
| | Vascular stent thrombosis |
| | Sub-Category: Other ischaemic heart disease (SMQ) |
| | Arteriogram coronary abnormal |
| | Cardiac stress test abnormal |
| | Cardiopulmonary exercise test abnormal |
| | Cardiovascular event prophylaxis |
| | Computerised tomogram coronary artery abnormal |
| | Elastic vessel recoil complication |
| | Electrocardiogram PR segment depression |
| | Electrocardiogram ST segment depression |
| | Electrocardiogram ST-T segment abnormal |
| | Electrocardiogram ST-T segment depression |
| | Electrocardiogram T wave abnormal |
| | Electrocardiogram T wave inversion |
| | Electrocardiogram U wave inversion |
| | Exercise electrocardiogram abnormal |
| | Exercise test abnormal |
| | Post angioplasty restenosis |
| | Restenosis |
| | Stress echocardiogram abnormal |
| | Vascular stent stenosis |
| | Wall motion score index abnormal |

| Category: Posterior Reversible Encephalopathy Syndrome (PRES) | |
|---|---|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| Search using Preferred Term | Posterior Reversible Encephalopathy Syndrome |

| Category: PML | |
|-----------------------------|--------------------------------------------|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| Search using Preferred Term | Progressive Multifocal Leukoencephalopathy |

| Category: Biopsy Procedure | |
|---|---|
| Search Strategy | MedDRA 22.0 PTs Included in SMQ |
| Review all AE Preferred Term for biopsy related AESI | All AE terms will be included |

#### 11.5.3.2. Coronavirus Disease 2019 (COVID-19) Environment Onset Date

A COVID-19 environment onset date has been defined by GlaxoSmithKline for each Country as:

| Country | COVID-19) Environment Onset Date |
|----------------|----------------------------------|
| Argentina | 10 FEB 2020 |
| Canada | 10 MAR 2020 |
| France | 25 FEB 2020 |
| Germany | 10 FEB 2020 |
| Italy | 10 FEB 2020 |
| Netherlands | 10 FEB 2020 |
| Norway | 10 FEB 2020 |
| Spain | 10 FEB 2020 |
| Sweden | 10 FEB 2020 |
| United Kingdom | 24 FEB 2020 |

This represents the best estimate of the outbreak of COVID-19 within each country at this time.

## 11.5.4. **Efficacy**

# +++Efficacy+++ Calculation of ESSDAI/ClinESSDAI score

• The ESSDAI includes 12 domains (ie, organ systems: cutaneous, respiratory, renal, articular, muscular, peripheral nervous system, central nervous system, hematological, glandular, constitutional, lymphadenopathy and biological). Each domain has 3 or 4 possible activity levels (Table 8).
### +++Efficacv+++

### **Corrected ESSDAI score:**

- For each damage eligible domain
  - where damage is scored as present for 1st time after screening **THEN** corrected activity score = damage score for that domain for that visit and the activity score for all subsequent visits should be changed to equal the corresponding damage domain score
  - Except in rare cases where the activity score for the visit concerned is already equal to or greater than the damage score, in which case no change should be made.
- If damage is scored as present at screening AND if the damage score increases in level of
  involvement (low to moderate or moderate to high) after the screening visit then the activity
  score for that domain for that visit and all subsequent visits should be changed to equal the
  corresponding damage domain score
  - Except in rare cases where the activity score for the visit concerned is already equal to or greater than the damage score, in which case no change should be made.
- If damage is scored at screening and remains constant across visits, then no programmed correction can or should be made to the activity scores.
- The ClinESSDAI includes 11 of the 12 ESSDAI domains (biological domain is excluded).

Table 8 ESSDAI Domains

| Activity level | Response |
|---|---|
| CCI - This section containe<br>Assessment data collection<br>indices, which are protecte | n questionnaires or<br>ed by third party |
| copyright laws and therefor | re have been excluded. |

<sup>\*</sup>Refer to Appendix 11 for details of the domains which incorporate High Response

The Total ESSDAI and Total ClinESSDAI Scores are obtained by multiplying the level of activity(Table 8) by the domain weights (Table 9). There are differing weightings for the ESSDAI and ClinESSDAI, and the biological domain is excluded from the calculation of the ClinESSDAI. The ESSDAI total score can range between 0 and 123. The ClinESSDAI total score can range between 0 and 135.

- Missing domains:
  - If there are missing responses for ≥ 3 domains, the Total ESSDAI and Total ClinESSDAI scores will be set to missing.
  - o If <3 domains are missing, imputation of missing domain responses will be applied to enable derivation of total scores. The individual domain scores from the nearest prior assessment which is up to 28 days earlier (and post baseline) will be carried forward and used for computation of total score. If there is no prior assessment meeting this criteria, the total scores will be set to missing.

## +++Efficacy+++ Table 9 Weighting for Computation of ESSDAI and ClinESSDAI

| Domain | Wei | ght |
|---|---|---|
| | ESSDAI | ClinESSDAI |
| Constitutional | CCI - This section contained<br>Assessment data collection | |
| Lymphadenopathy and lymphoma | which are protected by third therefore have been exclude | party copyright laws and |
| Glandular | mererore have been exclude | eu. |
| Articular | | |
| Cutaneous | | |
| Pulmonary | | |
| Renal | | |
| Muscular | | |
| Peripheral nervous system | | |
| Central nervous system | | |
| Haematological | | |
| Biological | | |

### Calculation of ESSDAI Response (Corrected)

- Three ESSDAI response variables will be computed. Definitions for responders is specified below:
  - Responders 1 Subjects with a reduction in total ESSDAI of at least 5 points over baseline
  - Responders 2 Subjects with a reduction in total ESSDAI of at least 3 points over baseline
  - Responders 3 Subjects with a reduction in total ESSDAI of at least 3 points over baseline, and ESSDAI Total Score <5</li>
  - Responders 4 ESSDAI Total Score < 5</li>

### **Lacrimal Gland Function**

- Stirp length wet (mm/min) is calculated as length (mm) paper wet divided by time taken to wet (min) for the left and right eyes. The length of Schirmer's strip is 35mm so wet/min can be calculated accordingly if the entire paper was wet and the time was recorded.
  - If duration is given as 0 or Not Applicable it will be considered as 5 mins.

### 11.5.5. Health Outcomes

### +++Patient Reported Outcomes+++

### **Calculation of ESSPRI Total Score**

- The ESSPRI has 3 domains (dryness, fatigue and pain)
- The ESSPRI total score is the mean of the 3 domain scores, with each domain score being the response between CCI and and CCI which is provided in response to the below questions.
  - CCI This section contained Clinical Outcome Assessment data collection questionnaires or indices, which
    are protected by third party copyright laws and therefore have been excluded.
- If there are missing responses for >1 domain, the ESSPRI total is set to missing. If 1 domain is missing, the nearest prior assessment up to 28 days earlier (and post baseline) for this domain will be carried forward and used for computation of total ESSPRI score. If there is no prior assessment meeting this criteria, the total score will be set to missing.

### **Calculation of ESSPRI Response**

- Two ESSPRI Response will be calculated.
- **Definition 1** An ESSPRI response is defined as a decrease in the ESSPRI total score of at least one point or at least 15% compared to baseline.
- **Definition 2** An ESSPRI response is defined as a patient with baseline of ≥ 5 and ESSPRI score < 5.

### **Calculation of PROFAD-SSI-SF**

- Each of the 19 questions of the short form PROFAD-SSI-SF has a severity scores ranging from 0 to 7 indicating increasing severity.
- Eight domain scores are derived from the 19-item PROFAD-SSI-SF questionnaire by taking averages of available responses to the relevant questions. Where responses are available for less than 50% of the required questions at the specific visit, the domain score for that visit will be set to missing.

| Domain | Questions | Domain Score Set to Missing |
|---|---|---|
| Somatic fatigue | | ed Clinical Outcome Assessment data<br>or indices, which are protected by third party |
| Mental fatigue | copyright laws and therefo | |
| Arthralgia | | |
| Vascular | | |
| Cutaneous dryness | | |
| Vaginal dryness | | |
| Ocular dryness | | |
| Oral dryness | | |

PROF, PROFAD and SSI subscores are derived by summing the domain scores listed in Table 10. The SSI subscores will be derived for females only.

Table 10 PROFADSSI Domains

| PROF | PROFAD | SSI |
|-----------------|-----------------|-------------------|
| Somatic fatigue | Somatic fatigue | Cutaneous dryness |
| Mental fatigue | Mental fatigue | Vaginal dryness |
| | Arthralgia | Ocular dryness |
| | Vascular | Oral dryness |

### 11.5.6. Biomarkers

A list of Flow Cytometry Parameters and associated variable names in the Biomarker dataset (BIOMARK) which will be summarized are provided in Table 11.

If BIMETHCD=FLWTBNK AND IF BICATCD = CD19 AND BITESTCD=CONC AND BIORRES = '<5 'then BIORRESN (i.e. Table 11 Column = Low B cell Imputation = Yes) will be imputed by S&P to result of subset parameter in % \* 2.5.

Example calculation for subset parameter:

| Panel<br>[BIMETH<br>CD] | Parame<br>ter<br>[BICAT<br>CD] | Unit<br>[BITEST<br>CD] | Unit<br>[BIORRE<br>SU] | Result (Numerical)<br>[BIORRESN] | Result<br>[BIORR<br>ES] |
|---|---|---|---|---|---|
| FLWTBN<br>K | CD19 | CONC | CELLS/C<br>UMM | | < 5 |
| FLWPLS<br>M | CDX136 | CONC | CELLS/C<br>UMM | Imputation = 96/100 * 2.5 = 2.4 | |
| FLWPLS<br>M | CDX136 | PERCEN<br>T | % | 96 | |

IF BIORRES="UNABLE TO CALCULATE" THEN the standard values (BISTRESC and BISTRESN) will be the same as in original values (BIORRES, BIORRESU), do not apply any imputation (i.e. DO NOT set 0).

Any other parameter reported as < x will be imputed to  $\frac{1}{2}x$ 

**Table 11** Flow Cytometry Parameters

| Biomarker<br>Testing<br>Method<br>Code<br>(BIMETHC<br>D) | BICATC<br>D | Parameter | BITEST<br>CD | Source Data Units of Measureme nt (BIORRES U) | Conversi<br>on of<br>source<br>data to<br>Cells/mL<br>for<br>reporting | Low B<br>cell<br>Imputati<br>on | Label [1] |
|---|---|---|---|---|---|---|---|
| FLWTBNK | CDX03 | CD3+ CD4+ | CONC | CELLS/CU<br>MM | N | N | CD4+ T cells |
| FLWTBNK | CDX02 | CD3+ CD8+ | CONC | CELLS/CU<br>MM | N | N | CD8+ T cells |
| FLWTBNK | CD19 | CD19+ B Cell | CONC | CELLS/CU<br>MM | N | Imputed | CD19+ Total B cells |
| FLWPLSM | CDX136 | Naïve CD20+<br>CD27- (% of<br>CD19+ cells) | PERCEN<br>T | % | N | N | Naïve B cell<br>CD20+ CD27- (%<br>of CD19 cells) |
| FLWPLSM | CDX136 | Naïve CD20+<br>CD27- | CONC | CELLS/CU<br>MM | N | Y | Naïve B cell<br>CD20+ CD27- |
| FLWPLSM | CDX137 | Memory CD20+<br>CD27+ | CONC | CELLS/CU<br>MM | N | Y | Memory B cell<br>CD20+ CD27+ |
| FLWPLSM | CDX137 | Memory CD20+<br>CD27+<br>(% of CD19+<br>cells) | PERCEN<br>T | % | N | N | Memory B cell<br>CD20+ CD27+<br>(% of CD19+<br>cells) |
| FLWPLSM | CDX143 | CD20- CD138+ | CONC | CELLS/CU<br>MM | Y | Y | Plasmacell<br>CD20- CD138+ |
| FLWPLSM | CDX141 | Activated B Cell<br>CD20+ CD69+<br>(% of CD19+<br>cells) | PERCEN<br>T | % | | N | Activated Total B<br>Cells CD20+<br>CD69+ (% of<br>CD19+ cells) |
| FLWPLSM | CDX141 | Activated B Cell | CONC | CELLS/CU | Υ | Υ | Activated Total B |

| Biomarker<br>Testing<br>Method<br>Code<br>(BIMETHC<br>D) | BICATC<br>D | Parameter | BITEST<br>CD | Source Data Units of Measureme nt (BIORRES U) | Conversi<br>on of<br>source<br>data to<br>Cells/mL<br>for<br>reporting | Low B<br>cell<br>Imputati<br>on | Label [1] |
|---|---|---|---|---|---|---|---|
| | а | CD20+ CD69+ | | MM | | | Cells CD20+<br>CD69+ |
| FLWPLSM | CDX156 | Plasmablast All<br>CD27+CD38+CD<br>19+<br>(% of CD19+<br>cells) | PERCEN<br>T | % | N | N | Plasmablast All<br>CD27+CD38+CD<br>19+<br>(% of CD19+<br>cells) |
| FLWPLSM | CDX156 | Plasmablast All<br>CD27+CD38+CD<br>19+ | CONC | CELLS/CU<br>MM | Y | Y | Plasmablast All<br>CD27+CD38+CD<br>19+ |
| FLWPLSM | CDX493 | Plasmablast<br>CD20+ | CONC | CELLS/ML | NA | Y | Plasmablast<br>CD20+ |
| FLWPLSM | CDX494 | Plasmablast<br>CD20- | CONC | CELLS/ML | NA | Y | Plasmablast<br>CD20- |
| FLWPLSM | CDX145 | CD20+ CD138+ | CONC | CELLS/CU<br>MM | Y | Y | Plasmacells<br>CD20+CD138+ |
| FLWPLSM | CD20 | B cells CD20+ | CONC | CELLS/CU<br>MM | N | Y | B cells CD20+ |
| FLWTBNK | CDX04 | Natural Killer<br>CD16+ CD56+ | CONC | CELLS/CU<br>MM | N | N | Natural Killer<br>CD16+ CD56+ |
| FLWTRAN<br>S | CDX198 | Transitional T2<br>CD19+ CD24Int+<br>CD38Int+ CD27- | CONC | CELLS/CU<br>MM | Y | Y | Transitional T2<br>CD24Int+<br>CD38Int+ CD27- |
| FLWTRAN<br>S | CDX199 | Transitional<br>CD19+ CD24b+<br>CD38b+ CD27-<br>(% of CD19+<br>cells) | %CD19+ | % | N | N | Transitional<br>CD24b+ CD38b+<br>CD27-<br>(% of CD19+<br>cells) |
| FLWTRAN<br>S | CDX199 | Transitional<br>CD19+ CD24b+<br>CD38b+ CD27- | CONC | CELLS/CU<br>MM | Y | Y | Transitional<br>CD24b+ CD38b+<br>CD27- |
| FLWTRAN<br>S | CDX202 | Memory Breg<br>Phenotype<br>CD19+ CD24b+<br>CD27+ | CONC | CELLS/CU<br>MM | Y | Y | Memory B cells<br>CD24b CD27+ |
| FLWTRAN<br>S | CDX203 | Naïve IgD+<br>CD19+ CD27-<br>IgD+ | CONC | CELLS/CU<br>MM | N | Y | Naïve B cell IgD+ |
| FLWTRAN<br>S | CDX84 | Non-Switched<br>Memory<br>CD19+ CD27+<br>IgD+ | CONC | CELLS/CU<br>MM | N | Y | Non-Switched<br>Memory<br>CD27+ IgD+ |
| FLWTRAN<br>S | CDX86 | Switched Memory<br>CD19+ CD27+<br>IgD- | CONC | CELLS/CU<br>MM | N | Y | Switched Memory<br>CD27+ IgD- |
| FLWTRAN<br>S | CDX87 | Plasmablast<br>CD38br CD27br<br>CD19+ | CONC | CELLS/CU<br>MM | Y | Y | Plasmablast<br>CD38br CD27br<br>CD19+ |
| FLWPLSM | CDX154 | Short-lived<br>Plasma CD20- | CONC | CELLS/CU<br>MM | Y | Y | Short-lived<br>Plasma CD20- |

2020N437857\_00 201842

| Biomarker<br>Testing<br>Method<br>Code<br>(BIMETHC<br>D) | BICATC<br>D | Parameter | BITEST<br>CD | Source Data Units of Measureme nt (BIORRES U) | Conversi<br>on of<br>source<br>data to<br>Cells/mL<br>for<br>reporting | Low B<br>cell<br>Imputati<br>on | Label [1] |
|---|---|---|---|---|---|---|---|
| | | CD27br | | | | | CD27br |
| FLWTRAN<br>S | CDX197 | Transitional<br>CD24+ CD27-<br>CD19+ | CONC | CELLS/CU<br>MM | N | Y | Transitional<br>CD24+ CD27-<br>CD19+ |
| FLWTRAN<br>S | CDX205 | Naïve B cells<br>CD24- CD38br<br>CD19+ | CONC | CELLS/CU<br>MM | N | Y | Naïve B cell<br>CD24- CD38br<br>CD19+ |

<sup>[1]</sup> Label included for reference only

The cells/mL records will be derived from source data as required. Cells/mL = 1000 \* Cells/CUMM.

The reporting units and database information for serologic biomarkers, complement and serum chemokines are detailed in Table 12.

**Table 12 Additional Biomarkers** 

| Biomarker<br>Category | Biomarker | Dataset | Dataset Codes | Reporting<br>Unit | Notes |
|---|---|---|---|---|---|
| Serologic<br>Markers | SS-A | LAB | LBTESTCD =<br>ASSARO_PLQ | KU/L | Categories for summary: <7 7 - 10 >10 - 120 >120 - 240 >240 |
| | SS-B | LAB | LBTESTCD =<br>ASSBLA_PLQ | KU/L | Categories for summary: <10 10 – 80 >80 – 160 >160 – 320 >320 |
| | Rheumatoid<br>Factor | LAB | LBTESTCD =<br>RF_PLC | KU/L | Impute values <10 to 5 |
| | Lambda light chain protein | LAB | LBTESTCD =<br>LLCPRO_PLC | mg/L | |
| | Kappa light chain protein | LAB | LBTESTCD = KLCPRO_PLC | mg/L | |
| | kappa/lambda<br>ratio* | LAB | LABTESTCD = LKLC_PLQ | mg/L | Derived |
| | Beta 2<br>microglobulin | LAB | LBTESTCD =<br>B2M_PLC | NMOL/L=SI<br>or<br>original=mg/L | |
| Complement | CH50 | LAB | LBTESTCD =<br>CH50_PLC | U/ml<br>=original unit | Categories for summary: <10 10-30 >30-60 >60 |
| | C3 | BIOMARK | BICATCD=C3 | G/L | |
| | C4 | BIOMARK | BICATD=C4 | G/L | |
| Serum<br>cytokine | CXCL13 | BIOMARK | BICATCD=BLC = BICCAT= B- lymphocyte chemokine | NG/L | _ |

<sup>\*</sup> The parameter is derived as a ratio of Kappa light chain protein to Lambda light chain protein

A list of Minor Salivary Gland Parameters and associated variable names in the MI dataset which will be summarized are provided in Table 13.

Only baseline and Week 24 data will be reported for Primary Analysis reporting. Any parameter reported as 'No B-cells (CD20)' will be excluded from summary.

Table 13 Minor Salivary Gland Parameters

| Parameter | Units | MITESTCD | Replicate Results Databased defined by MIREFID2 (biopsy slices) [3] |
|---|---|---|---|
| [1] Lymphoma Risk | Negative/P ositive | AG001 | N |
| [2] Lymphocyte Focus Score | per 4 mm <sup>2</sup> | AG006 | Υ |
| <sup>[2]</sup> B cell (CD20) | count/mm <sup>2</sup> | AG007 | N |
| <sup>[2]</sup> B (CD20) / T (CD3) cell ratio | | AG008 | N |
| [2] Plasma cell (CD138+; both - CD20pos and CD20neg) | count/mm <sup>2</sup> | AG012 | N |
| T cell (CD3) | count/mm <sup>2</sup> | AE005 | N |
| Total aggregate area/total glandular area | ratio | AG004 | Υ |
| Average Focus size | mm <sup>2</sup> | AG005 | Υ |
| Percent Foci displaying Germinal centres* | % | AG010 | Υ |
| Percent Foci displaying follicular dendritic cells (CD21) | % | AG011 | Y |
| Percent Foci displaying CD3/CD20 segregation | % | AG009 | Υ |
| Plasma cell (CD138; both CD20+ and CD20-)/<br>B cell (CD20) | ratio | AG018 | N |
| Plasma cell (CD138+, CD20+) | count /mm <sup>2</sup> | AG020 | N |
| Plasma cell (CD138+, CD20-) | count /mm <sup>2</sup> | AG021 | N |
| Memory B Cell (CD20+CD27+) | count /mm <sup>2</sup> | AG022 | N |
| Follicular B cell (IgD+, CD20+) | count /mm <sup>2</sup> | AG017 | N |
| Non-switched Memory B cell (IgD+, CD20+, CD27+) | count /mm <sup>2</sup> | AG023 | N |
| Switched Memory B cell (IgD-, CD20+, CD27+) | count /mm <sup>2</sup> | AG024 | N |

<sup>[1]</sup> Lymphoma risk assessed at screening only and presented in baseline characteristics summary.

For the histology parameters where replicate results (i.e. from two different cutting levels) are provided (as indicated by 'Y'), average across all the replicates will be derived for analysis. If no replicate, then available value will be used for summary.

### 11.5.6.1. Immunogenicity

Anti-drug antibody (ADA) assays (Belimumab and Rituximab):

- 1. Binding assay: Tiered assay (Screening, confirmation, and titer) to assess the presence of ADA
  - Screening assessment is performed producing a result that is positive or negative. Negative samples in the screening assay are negative for the binding assay.
  - For samples with a positive screening assessment, a confirmation assay is carried out which produces a positive or negative result. A subject is confirmed as positive for the assessment at this step. Samples testing positive in the screening assay, but negative in the confirmation assay are

<sup>[2]</sup> Parameters reported at interim analysis

<sup>[3]</sup> For some assessments, sections from two different cutting levels are planned, and an additional section may be taken for analysis if discrepant results across cutting levels (difference >2 in focus score).

- negative; samples testing positive in both the binding assay and the confirmation assay are positive for the binding assay
- o For samples with a positive binding assay (positive in the screening and confirmation) result, a titer value is obtained to quantify the degree of binding in a titration assay step. The titer result is the inverse of the dilution at which the sample no longer tests positive in the screening assay.
- 2. Neutralizing assay (NAb) (only for Belimumab): Assay to determine if ADA present in a sample is neutralizing to the activity of the drug. Subjects who test positive for the binding assay may be further characterized by testing confirmed positive samples from the binding assay in the neutralizing assay, which produces a positive or negative result.

If a subject has a positive screening assessment from the binding assay, but the confirmatory assessment is missing, the immunogenicity response will be reported as "Unknown".

• **NOTE:** For subjects WD IP and immediately entering Week 68/FU, assess any impact if visits are not in chronological order, when categorizing Persistent Positive. Adjust if required.

### Reporting of Rituximab

The following definitions will be applied when summarizing the data.

### **Persistent Positive (PP)**

### Baseline (Week 8):

- 1. Baseline (Week 8) is the first-time immunogenicity is being tested and therefore cannot be PP
- 2. One exception is IF confirming = positive @ Baseline (Week 8) & subject WD from study prior to Week 24 THEN PP

### Post Baseline (Week 8):

Positive response that occurs at least 2 consecutive assessments or a single result at the final assessment (i.e. point 2 above)

### **Transient Positive (TP)**

• Single positive response that does not occur at the final assessment

NOTE: Both the screening and confirming test for the time point in question must be positive

Additional Programming Notes:

2020N437857\_00 201842

- IF your Positive @ Week 8 = TP AND IF the same subject @ Week 24 = Positive then will be classified as PP at Week 24 ONLY BUT cannot be retrospectively applied (i.e. being PP) to the same subject at Week 8
- IF the same subject @ Week 52 was negative then classified as negative at this timepoint (i.e. PP classification cannot be carried forward from previous timepoint)

## 11.6. Appendix 6: Reporting Standards for Missing Data

### 11.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as a subject who has completed the treatment and general follow up phase of the study including the Week 68 visit.</li> <li>Subjects may discontinue treatment and continue to complete remaining scheduled visits whilst off treatment or withdraw from study prior to Week 68.</li> <li>All available data from subjects who discontinue treatment or are withdrawn from the study will be included in analysis, summary tables and figures, unless otherwise specified.</li> </ul> |

## 11.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank<br/>fields on the collection instrument:</li> </ul> |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing<br/>displays. Unless all data for a specific visit are missing in which case the<br/>data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | <ul> <li>Any subjects excluded from the summaries and/or statistical analyses will be<br/>documented along with the reason for exclusion in the clinical study report.</li> </ul> |

## 11.6.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> </li> </ul> |

## 11.6.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be<br/>imputed using the following convention:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | <ul> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the<br/>full date cannot be ascertained, the following assumptions will be made:</li> </ul> |
| | <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will<br/>be used for the month.</li> </ul> |
| | <ul> <li>However, if these results in a date prior to Week 1 Day 1 and the event<br/>could possibly have occurred during treatment from the partial information,<br/>then the Week 1 Day 1 date will be assumed to be the start date.</li> </ul> |
| | <ul> <li>The AE will then be considered to start on-treatment (worst case).</li> </ul> |
| | <ul> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day<br/>(dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> |
| | <ul> <li>The recorded partial date will be displayed in listings.</li> </ul> |

## 11.6.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Appendix 5 details imputations that will applied to obtain total scores for<br/>ESSDAI, ClinESSDAI and ESSPRI where sufficient partial data are collected.<br/>An MMRM approach is planned for the key efficacy readouts.</li> </ul> |

## 11.7. Appendix 7: Values of Potential Clinical Importance

## 11.7.1. Laboratory Values

| Hematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Lymphocytes | GI/L | | 0.8 | |
| Neutrophil Count | GI/L | | 1.5 | |
| Platelet Count | GI/L | | 100 | 550 |
| While Blood Cell Count (WBC) | GI/L | | 3 | 20 |
| Monocytes | GI/L | | 1.8 | 8 |
| Eosinophils | GI/L | | 0.05 | 0.55 |
| Basophils | GI/L | | 0 | 0.2 |
| Red Blood Cell Count (RBC) | TI/L | | 3.6 | 5.1 |
| Hemoglobin | G/L | | 71 | 199 |
| Hematocrit | I | | 0.201 | 0.599 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| <b>Laboratory Parameter</b> | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | G/L | | 32 | 50 |
| Creatinine | umol/L | | 53 | 104.3 |
| Glucose | mmol/L | | 3.9 | 6.9 |
| Potassium | mmol/L | | 3.5 | 5.3 |
| Sodium | mmol/L | | 135 | 146 |
| Chloride | mmol/L | | 95 | 108 |
| Urea/BUN | mmol/L | | 2.5 | 9 |
| Creatinine Kinase | IU/L | | 0 | 190 |
| Uric Acid | umol/L | | 150 | 450 |

| Liver Function | | | |
|----------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |

2020N437857\_00 201842

| Laboratory Parameter | Units | Normal Ranges | |
|----------------------|-------|----------------|----------------|
| | | Low Flag (< x) | High Flag (>x) |
| IgG | G/L | 6.94 | 16.18 |
| IgM | G/L | 0.48 | 2.71 |
| IgA | G/L | 0.81 | 4.63 |

## 11.7.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|----------|
| (Change from Baseline) | | Decrease | Increase |
| Systolic Blood Pressure | mmHg | ≥ 30 | ≥ 30 |
| Diastolic Blood Pressure | mmHg | ≥ 20 | ≥ 20 |
| Heart Rate | bpm | ≥ 30 | ≥ 30 |

# 11.8. Appendix 8: Laboratory Parameters & Toxicity Grading Tables

## 11.8.1. Laboratory Parameters

| | | Other |
|---|---|---|
| Hematology | Urinalysis | <b>Screening Tests</b> |
| CBC: WBC Count | Specific gravity | HIV, Hepatitis B<br>(HBsAg) and HbcAb |
| Hemoglobin Hematocrit | pH, glucose, protein,<br>blood and ketones by | Hepatitis C (Hep C antibody) |
| Platelet Count | dipstick | FSH and estradiol |
| RBC Indices: | | Serum or urine hCG |
| RBC Count | | Pregnancy |
| • MCV | | |
| • MCH | | |
| WBC Differential: | | |
| Neutrophils | | |
| Lymphocytes | | |
| Monocytes | | |
| Eosinophils | | |
| Basophils | | |
| Biological Markers | Immunogenicity | PK |
| TBNK panel: | Rituximab | Rituximab PK |
| CD16+CD56+ (Natural Killer Cell) Count (counts/ml) | immunogenicity | |
| % CD16+CD56+ (Natural Killer Cell) (as a proportion of tot | | Belimumab PK |
| lymphocytes) | Belimumab | |
| CD3+CD4+ (Helper T Cell) Count | immunogenicity | |
| CD3+CD8+ (Cytotoxic T Cell) Count | | |
| Serologic Markers | | |
| Concentration SS-A and SS-B | | |
| Concentration Rheumatoid factor | | |
| Concentration Lambda and kappa free light chains | | |
| Concentration Beta 2 microglobulins | | |
| Complement Factors: | | |
| Concentration C3 | | |
| Concentration C4 | | |
| Concentration CH50 | | |
| <u>Immunoglobulins</u> | | |
| • IgG, IgA, IgM | | |
| Core 6-colour B cell assay ('plasma B cell panel'): | | |
| • B cell (CD19+) | | |
| Naïve B cell (CD19+CD20+CD27-) (absolute count) | | |

2020N437857\_00 201842

| <ul> <li>Naïve B cell (CD19+CD20+CD27-) (percentage of CD19</li> </ul> |
|------------------------------------------------------------------------|
|------------------------------------------------------------------------|

- Memory B cell (CD19+CD20+CD27+) (absolute count)
- Memory B cell (CD19+CD20+CD27+) (percentage of CD19+)
- Plasmablast All (CD19+CD27+CD38+) (absolute count)
- Plasmablast All (CD19+CD27+CD38+) (percentage of CD19+)
- Plasmablast CD20+ (CD19+CD20+CD27br+CD38br+) (absolute count)
- Plasmablast CD20- (CD19+CD20-CD27br+CD38br+) (absolute count)

### Exploratory 6-colour B cell assay ('plasma B cell panel'):

- Activated B cells (CD19+CD20+CD69+) (absolute count)
- Activated B cells (CD19+CD20+CD69+) (percentage of CD19+)
- Plasmacell (CD20- CD138+) (absolute count)

### Listings only 6-colour B cell assay ('plasma B cell panel'):

- Plasmacells CD20+ (CD20+CD138+) (absolute count)
- B cells CD20+ (CD19+CD20+)(absolute count)

### Core CD24w/Plasma B cell assay ('Transitional B cell Panel'):

- Transitional T2 (CD19+ CD24Int+CD38Int+CD27-) (absolute count)
- Transitional (CD19+CD24br+CD38br+CD27-) (percentage of CD19+)
- Transitional (CD19+CD24br+CD38br+CD27-) (absolute count)
- Non-switched memory (CD19+CD27+lgD+) (absolute counts)
- Switched memory (CD19+CD27+lgD-) (absolute counts)

## Exploratory CD24w/Plasma B cell assay ('Translational B cell Panel'):

- Memory 'Breg phenotype' (CD19+CD24br+CD27+) (absolute count)
- Naïve lgD+ (CD19+CD27-lgD+) (absolute count)

## <u>Listings only CD24w/Plasma B cell assay ('Transitional B cell Panel')</u>

- Plasmablasts (CD38br CD27br CD20+) (absolute count)
- Short-lived Plasma (CD20- CD27br) (absolute count)
- Transitional (CD24+ CD27-) (absolute count)
- Naïve B cells (CD24-CD38br+) (absolute count)

### Concentration C-Reactive Protein

### Concentration free BLyS \*

#### Core Minor Salivary Gland histology assessments:

- Lymphocyte Focus Score (in 4mm²)
- B cell (CD20) count/mm<sup>2</sup>
- B (CD20) / T (CD3) cell ratio

| Plasma cell (CD138+; both - CD20pos and CD20neg) count/mm <sup>2</sup> |
|------------------------------------------------------------------------|
| Memory B Cell (CD20+CD27+) count/mm <sup>2†</sup> |
| Exploratory Minor Salivary Gland Histology Assessments |
| T (CD3) cell /mm² |
| Total aggregate area/total glandular area (ratio) |
| Average Focus size (mm²) |
| % Foci displaying Germinal centres |
| % Foci displaying follicular dendritic cells (CD21) |
| % Foci displaying CD3/CD20 segregation |
| Plasma cell (CD138; both CD20+ and CD20-)/ B cell (CD20) ratio |
| Plasma cell (CD138+, CD20+) count /mm² |
| Plasma cell (CD138+, CD20-) count /mm² |
| Lymphoma risk - Assessed as Yes or No |
| End of Study: Additional parameters maybe reported, if available: |
| Follicular B cell (IgD+, CD20+) |
| Non-switched Memory B cells (IgD+, CD20+, CD27+) |
| Switched Memory B cells (IgD-, CD20+, CD27+) |
| Serum cytokines and chemokines: |

<sup>†</sup>Will be reported for End of Study

Concentration CXCL13

## 11.8.2. Toxicity Grading Tables

Modified version of <u>DMID</u> is used for the toxicity grading with the exception of IgG (values taken from scientific literature) and lymphocytes (values taken from CTCAE V4).

| HEMATOLOGY | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| Hemoglobin | 9.6-11 G/DL | 8.1-9.5 G/DL | 6.5-8 G/DL | 0-6.4 G/DL |
| | 96-110 G/L | 81-95 G/L | 65-80 G/L | 0-64 G/L |
| Leukocytes | 3-3.9 THOU/MCL | 2-2.9 THOU/MCL | 1-1.9 THOU/MCL | 0-0.9 THOU/MCL |
| | 3-3.9 GI/L | 2-2.9 GI/L | 1-1.9 GI/L | 0-0.9 GI/L |
| Absolute Neutrophils | 1.5-1.99 THOU/MCL | 1-1.49 THOU/MCL | 0.5-0.99 THOU/MCL | 0-0.49 THOU/MCL |
| WATER BACK TO CAPE CONTROL | 1.5-1.99 GVL | 1-1.49 GI/L | 0.5-0.99 GI/L | 0-0.49 GI/L |
| Platelets | 75,000-99,999 PER CUMM | 50,000-74,999 PER CUMM | 25,000-49,999 PER CUMM | 0-24,999 PER CUMM |
| | 75-99 GI/L | 50-74 GI/L | 25-49 GI/L | 0-24 GI/L |

<sup>\*</sup>Total BLyS concentrations only for End of Study analysis

## 2020N437857\_00 201842

| CHEMISTRIES | | GRADE 0<br>(QUEST DB<br>REQUIREMENT) | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|---|---|
| THE STREET | | AL QUITE HEIT | 2006 1 | - IVILLA | MINE V | SIGNE 3 |
| Sodium (step-wise grading for | | | | | | |
| Hyponatremia and Hyperna-<br>tremia combined) | | 138-145 MEQ/L | 130-150 MEQ/L | 123-157 MEQ/L | 116-165 MEQ/L | 0-99,999 MEQ/L |
| | | 136-145 MMOL/L | 130-150 MMOL/L | 123-157 MMOL/L | 118-165 MMOL/L | 0-99.999 MMOL/L |
| Hyponatremia | | 100000000000000000000000000000000000000 | 130-135 MEQ/L | 123-129 MEQ/L | 116-122 MEQ/L | <116 MEQ/L |
| Hypematremia | | | 146-150 MEQ/L | 151-157 MEQ/L | 158-165 MEQ/L | >165 MEQ/L |
| Potassium (step-wise grading | | | | | | |
| for Hypokalemia and Hyper-<br>kalemia combined) | | 3.5-5.5 MEQ/L | 3-6 MEQ/L | 2.5-6.5 MEQ/L | 2-7 MEQ/L | 0-9.999.9 MEQ/L |
| naiema comunecy | | 3.5-5.5 MMOL/L | 3-6 MMOL/L | 2.5-6.5 MMOL/L | 2-7 MMOL/L | 0-9,999.9 MMOL/L |
| Hypokalemia | | o.c o.c minocic | 3.0-3.4 MEQ/L | 2.5-2.9 MEQ/L | 2.0-2.4 MEQ/L | <2.0 MEQ/L |
| Hperkalemia | | | 5.6-6.0 MEQ/L | 6.1-6.5 | 6.6-7.0 MEQ/L | >7.0 MEQ/L |
| Phosphate | | | | | | |
| (analyte not within chem.<br>panel for this protocol so will | | | | | | |
| flag) | | | 2-2.4 MG/DL | 1.5-1.9 MG/DL | 1-1.4 MG/DL | 0-0.9 MG/DL |
| | | | 0.65-0.75 MMOL/L | 0.5-0.64 MMOL/L | 0.3-0.49 MMOL/L | 0-0.29 MMOL/L |
| Calcium (corrected for Albu-<br>min) | | | | | | |
| (step-wise grading for Hypo- | | | | | | |
| calcemia and Hypercalcemia<br>combined) | | 8.5-10.5 MG/DL | 7.8-11.5 MG/DL | 7-12.5 MG/DL | 6.1-13.5 MG/DL | 0-9.999.9 MG/DL |
| oundired) | | 5.5-10.5 MG/DL | 7.0-11.5 MG/DL | 1-12.5 MOIDE | 0. 1-13.5 MO/DL | 0-8,888.8 MOIDL |
| | | To the world the same | | | | |
| | | 2.12-2.62 MMOL/L | 1.94-2.86 MMOL/L | 1.74-3.12 MMOL/L | 1.52-3.36 MMOL/L | 1.52-9,999.99 MMOL/L |
| Hypocalcemia | | | 7.8-8.4 mg/dL | 7.0-7.7 mg/dL | 6.4-6.9 mg/dL | <6.1 mg/dL |
| Hypercalcemia<br>Magnesium | | | 10.6-11.5 mg/dL | 11.6-12.5 mg/dL | 12.6-13.5 mg/dL | >13.5 mg/dL |
| (analyte not within chem. | | | | | | |
| panel for this protocol so will | | | 1.2-1.4 MEQ/L | 0.9-1.1 MEQ/L | 0.6-0.8 MEQ/L | 0-0.5 MEQ/L |
| flag) | | | 0.6-0.7 MMOL/L | 0.46-0.59 MMOL/L | 0.3-0.45 MMOL/L | 0-0.29 MMOL/L |
| Albumin | | | 3-3.4 G/DL | 2.5-2.9 G/DL | 2-2.4 G/DL | 0-1.9 G/DL |
| | | | 30-34 G/L | 25-29 G/L | 20-24 G/L | 0-19 G/L |
| Bilirubin (Total) | | | 1.4-1.9 MG/DL | 2.0-3.2 MG/DL | 3.3-6.5 MG/DL | 6.6-9,999.9 MG/DL |
| | | | 23-33 UMOL/L | 34-55 UMOL/L | 56-110 UMOL/L | 111-9,999.9 UMOL/L |
| | | | > 1.0-1.5 x ULN | > 1.2-2.5 x ULN | > 2.5-5 x ULN | >5 x ULN |
| Glucose<br>(step-wise grading for Hypo- | | | | | | |
| glycemia and Hyperglycemia combined) | | 65-115 MG/DL | 55-160 MG/DL | 40-250 MG/DL | 30-500 MG/DL | 0-99.999 MG/DL |
| combined) | | 3.6-6.4 MMOL/L | 3.1-8.9 MMOL/L | 2.2-13.9 MMOL/L | 1.7-27.8 MMOL/L | 0-99999 MMOL/L |
| Hypoglycemia | | J.J-U.H MIMOLIL | 55-94 mg/dL | 40-54 mg/dL | 30-39 mg/dL | <30 mg/dL |
| Hyperglycemia | | | 116-160 mg/dL | 161-250 mg/dL | 251-500 mg/dL | >500 251-500 mg/dL |
| Creatinine | | Ref Range MG/DL | | | MG/DL | TOTAL TOTAL STATE OF THE STATE |
| | M 18-<br>19y | 0.67-1.26 | 1.27 - 1.89 | 1.90 - 3.78 | 3.79 - 7.58 | >7.56 |
| | F 18-19y | 0.67-1.26 | 1.02 - 1.51 | 1.52 - 3.03 | 3.04 - 6.08 | >6.08 |
| | M 20- | 0.80-1.30 | | | | >7.80 |
| | 29y | 0.80-1.30 | 1.31 - 1.95 | 1.96 - 3.90 | 3.91 - 7.80 | |
| | F 20-29y<br>M 30-39y | 0.57-1.03 | 0.58 - 1.54<br>1.34 - 1.99 | 1.54 - 3.09<br>2.00 - 3.99 | 3.10 - 6.18<br>4.00 - 7.98 | >6.18<br>>7.98 |
| | M 30-39y<br>F 30-39y | 0.79-1.33 | 1.07 - 1.59 | 1.60 - 3.18 | 3.19 - 6.38 | >7.98 |
| | M 40-49y | 0.78-1.34 | 1.35 - 2.01 | 2.02 - 4.02 | 4.03 - 8.04 | >8.04 |
| | F 40-49y | 0.59-1.07 | 1.08 - 1.60 | 160 - 3.21 | 3.22 - 6.42 | >6.04 |
| | M 50-59v | 0.76-1.46 | 1.47 - 2.19 | 2.20 - 4.38 | 4.39 - 8.76 | >8.76 |
| | F 50-59y | 0.60-1.10 | 1.11 - 1.65 | 1.66 - 3.30 | 3.31 - 6.60 | >6.60 |
| | M 60-69v | 0.76-1.46 | 1.47 - 2.19 | 2.20 - 4.38 | 4.39 - 8.76 | >8.76 |
| | | | | The second second | en selven se se se | |
| | F 60-69y | 0.60-1.18 | 1.19 - 1.77 | 1.78 - 3.54 | 3.55 - 7.08 | >7.08 |
| | M >69y | 0.67-1.54 | 1.55 - 2.31 | 2.32 - 4.62 | 4.63 - 9.24 | >9.24 |
| | F>69y | 0.63-1.22 | 1.23 - 1.83 | 1.84 - 3.66 | 3.67 - 7.32 | >7.32 |
| | | Ref Range UMOL/L | | | UMOLAL | |

## 201842 | Statistical Analysis Plan EoS RAP 15 Sep 2020 | TMF-2108787 | 4.0

## CONFIDENTIAL

## 2020N437857\_00 201842

| | M 18-19y | 59.2-111.4 | 111.5 - 167.1 | 167.2 - 334.2 | 334 3 - 668 4 | >668 4 |
|---|---|---|---|---|---|---|
| | F 18-19y | 42.4-89.3 | 89.4 - 133.9 | 134.0 - 267.9 | 268.0 - 535.8 | >535.8 |
| | M 20-29v | 70.7-114.9 | | | | |
| | F 20-29v | 50.4-91.1 | 115.0 - 172.3 | 172.4 - 344.7 | 344.8 - 689.4 | >689.4 |
| | | | 91.2 - 136.6 | 136.7 - 273.3 | 273.4 - 546.6 | >548.8 |
| | M 30-39y | 69.8-117.6 | 117.7 - 176.4 | 176.5 - 352.8 | 352.9 - 705.6 | >705.6 |
| | F 30-39y | 51.3-93.7 | 93.8 - 140.5 | 140.6 - 281.1 | 281.2 - 562.2 | >562.2 |
| | M 40-49y | 69.0-118.5 | 118.6 - 177.7 | 177.8 - 355.5 | 355.6 - 711.0 | >711.0 |
| | F 40-49y | 52.2-94.6 | 94.7 - 141.9 | 142 - 283.8 | 283.9 - 567.6 | >587.6 |
| | M 50-59y | 67.2-129.1 | 129.2 - 193.6 | 193.7 - 387.3 | 387.4 - 774.6 | >774.6 |
| | F 50-59y | 53.0-97.2 | 97.3 - 145.8 | 145.9 - 291.6 | 291.7 - 583.2 | >583.2 |
| | M 60-69y | 67.2-129.1 | 129.2 - 193.6 | 193.7 - 387.3 | 387.4 - 774.6 | >774.6 |
| | F 60-69y | 53.0-104.3 | 104.4 - 156.4 | 158.5 - 312.9 | 313.0 - 625.8 | >625.8 |
| | M >69y | 59.2-136.1 | 136.2 - 204.1 | 204.2 - 408.3 | 408.4 - 816.6 | >816.6 |
| | F>69y | 55.7-107.8 | 107.9 - 161.7 | 161.8 - 323.4 | 323.5 - 646.8 | >646.8 |
| | 200000 | | >1.0-1.5 x ULN | >1.5-3 x ULN | >3.0-6.0 x ULN | >6.0 x ULN |
| Uric Acid | | | 7.5-10 MG/DL | 10.1-12 MG/DL | 12.1-15 MG/DL | 15.1-9,999.9 MG/DL |
| -accidend | | | 450-590 UMOL/L | 591-710 UMOL/L | 711-890 UMOL/L | 891-99,999 UMOL/L |
| AST | 0-64y | | 53-105 U/L | 106-210 U/L | 211-420 U/L | 421-99,999 U/L |
| | 65-199y | | 69-137U/L | 138-275 U/L | 276-550 U/L | 551-99,999 U/L |
| | | | 1.25-2.5 x ULN | >2.5-5.0 x ULN | >5.0-10.0 x ULN | >10.0 x ULN |
| ALT | | | 60-120 U/L | 121-240 U/L | 241-480 U/L | 481-99,999 U/L |
| | | | 1.25-2.5 x ULN | >2.5-5.0 x ULN | >5.0-10.0 x ULN | >10.0 x ULN |
| GGT<br>(analyte not within chem.<br>panel for this protocol so will | | | | | | |
| flag) | M 0-64y | | 82-162 U/L | 163-325 U/L | 326-650 U/L | 651-99,999 U/L |
| | F 0-64y | | 57-112 U/L | 113-225 U/L | 228-450 U/L | 451-9,999 U/L |
| | 65-199y | | 94-187 U/L | 188-375 U/L | 376-750 U/L | 751-99,999 U/L |
| | | | 1.25-2.5 x ULN | >2.5-5.0 x ULN | >5.0-10.0 x ULN | >10.0 x ULN |
| Alkaline Phosphatase | M 16-<br>19y | | 282-562 U/L | 563-1,125 U/L | 1,126-2,250 U/L | 2,251-99,999 U/L |
| entres com Grandstate & Carter to Sec. of | F 16-19y | | 207-412 U/L | 413-825 U/L | 826-1,650 U/L | 1,651-99,999 U/L |
| | 20-199y | | 157-312 U/L | 313-625 U/L | 626-1,250 U/L | 1,251-99,999 U/L |
| | | | 1.25-2.5 x ULN | → 2.5-5.0 x ULN | >5.0-10.0 x ULN | >10.0 x ULN |

| IMMUNOGLOBULINS | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| IgG (Immunoglobulins) | 550-700 MG/DL | 400-549 MG/DL | 250-399 MG/DL | 0-249 MG/DL |
| | 5.5-7 G/L | 4-5.49 G/L | 2.5-3.99 G/L | 0-2.49 G/L |

| GRADE 0 | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| | 1++ | 2++, 3++ | 4++ | n/a |
| 0-1, 1-3 | 3-5 | 5-10, 6-10, 10+, 10-15, 10-20,<br>15-25, 20-40,<br>20+, 25-50, 50-100, | CLUMPING, CLUMPED, | n/a |
| | GRADE 0<br>0-1, 1-3 | 1++ | 1++ 2++, 3++<br>5-10, 6-10, 10+, 10-15, 10-20,<br>0-1, 1-3 3-5 15-25, 20-40, | 1++ 2++, 3++ 4++ 5-10, 6-10, 10+, 10-15, 10-20, 15-25, 20-40, 20+, 25-50, 50-100, CLUMPING, CLUMPED, |

| PROTEIN/CREATININE<br>RATIO | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| Protein/Creatinine Ratio | 0.2-1 MG/MG | 1.001-2 MG/MG | 2,001-3.5 MG/MG | 3.501-999.999 MG/MG |

| Lymphopenia | GRADE 1 | GRADE 2 | GRADE 3 | GRADE 4 |
|---|---|---|---|---|
| Lymphocyte count | <lln -="" 800="" mm3;<br=""><lln -="" 0.8<br="">x 10e9 /L</lln></lln> | <800 - 500/mm3;<br><0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3;<br><0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10e9<br>/L |

# 11.9. Appendix 9: Model Checking and Diagnostics for Statistical Analyses

### 11.9.1. Statistical Analysis Assumptions

### 11.9.1.1. Continuous Endpoints

| Endpoint(s) | Change from Baseline in ESSDAI Score |
|-------------|-------------------------------------------------------------|
| | Change from Baseline in ClinESSDAI Score |
| | Change from Baseline in Stimulated salivary Flow |
| | Change from Baseline in Oral Dryness Numeric Response Scale |
| Analysis | • MMRM |

- Model assumptions will be applied, but appropriate adjustments may be made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.
- Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure.
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
- Distributional assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted
  values (i.e. checking the normality assumption and constant variance assumption of the model
  respectively) to gain confidence that the model assumptions are reasonable.
- If there are any serious departures from the distributional assumptions, nonparametric rank
  Hodges-Lehmann's confidence intervals will be provided in order to assess the robustness of
  the parametric analysis. This will be carried out in addition to the parametric analyses.

| Endpoint(s) | • | Change from Baseline in ESSDAI Score |
|-------------|---|--------------------------------------|
| | • | Change from Baseline in ESSPRI Score |
| Analysis | • | Bayesian |

### **General Considerations for Bayesian Analysis:**

Convergence for all the parameters in the model will be verified

### **Initial Values:**

- Unless otherwise specified, initial parameter values of 0.5 will be used for the fixed effect parameters.
- If convergence of the Markov chain Monte Carlo (MCMC) algorithm is problematic, then alternative estimates may be used (for example, these could be based on maximum likelihood estimates).

### **Convergence Diagnostics:**

To be able to perform Bayesian inference using MCMC simulations the samples for all the
parameters in the model need to be obtained from the corresponding target posterior
distribution. To ensure that this is the case the following is a list of convergence diagnostics
that can be applied for each parameter:

### Comparing MCSE vs posterior standard deviation:

- The Monte Carlo Standard Errors (MCSE) should be compared with the standard deviation of the posterior distribution (SD) to ensure that only a fraction of the posterior variability is due to the simulation, i.e., the ratio MCSE/SD should be as small as possible, typically close to 0.01.
- Adequate values for the number of MCMC samples / thinning / number of burn-in samples should be chosen to ensure that the ratio MCSE/SD for all the parameters in the model is approximately 0.01.
- In addition, if possible, the number of tuning units and maximum number of tuning iterations
  may be increased to find a better proposal distribution for the model parameters, which in turn
  may reduce the MCSE/SD ratio.
- Where possible the code should be written to allow the SAS compiler to identify and make use
  of conjugacy, since this can greatly reduce the corresponding MCSE/SD ratio

### Diagnostic plots and visual inspection:

- Trace plots of samples versus the simulation index can used to assess some aspects of
  convergence. The centre of the chain should appear stable with very small fluctuations, i.e.,
  the distribution of points should not change as the chain progresses and the posterior mean
  and variance are relatively constant.
- Autocorrelation plots can be used to assess degree of autocorrelation (should decline rapidly and show no oscillation patterns).
- The posterior density should look reasonable for each parameter (e.g. for posterior parameters expected to follow a normal distribution, the density plot should not appear bi-modal, but for parameters acting as binary flags, then bi-modal is acceptable).
- Examination of correlation structures between relevant posterior parameters should be used to
  provide information about what potential issues may be and also what corrective action(s) may
  be worthwhile attempting.

2020N437857\_00 201842

### 11.9.1.2. Binary Endpoints

| Endpoint(s) | • | Binary Endpoints as described in Section 8.1.2 |
|-------------|---|------------------------------------------------|
| Analysis | • | Generalised Estimating Equations (GEE) |

- For the GEE analyses, model assumptions will be applied, but appropriate adjustments may be made based on the data.
- An unstructured working correlation structure will be assumed and standard errors will be calculated based on the empirical sandwich covariance estimate (default setting for PROC GENMOD in SAS)
- An unstructured correlation structure will be used by specifying 'type=UN' on the REPEATED line.
  - o In the event that this model fails to converge, alternative correlation structures may be considered such as Independent, CS or AR(1).
  - Quasilikelihood under the Independence Model Criteria (QIC) will be used to assist with the selection of covariance structure.

## 11.10. Appendix 10 – Abbreviations & Trade Marks

## **Abbreviations**

| , |
|------------------------------------------------------------------------|
| Description |
| Analysis Data Model |
| Adverse Event |
| Akaike's Information Criteria |
| Analysis and Reporting |
| Clinical Data Interchange Standards Consortium |
| Confidence Interval |
| Clinical Pharmacology Modeling & Simulation |
| Clinical Statistics |
| Clinical Study Report |
| Common Terminology Criteria for Adverse Events |
| Clinical Trial Register |
| Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| Division of Microbiology and Infectious Diseases |
| Date of Birth |
| Decimal Places |
| Electronic Case Record Form |
| End of Study |
| Eular Sjögren's Syndrome Disease Activity Index |
| Clinical Eular Sjögren's Syndrome Disease Activity Index |
| Eular Sjögren's Syndrome Patient Reported Index |
| GlaxoSmithKline |
| Interim Analysis |
| International Conference on Harmonization |
| Independent Data Monitoring Committee |
| Integrated Data Standards Library |
| Individualized Follow Up |
| International Modules Management System |
| Investigational Product |
| Safety Review Committee |
| Intent-To-Treat |
| Last Observation Carries Forward |
| Mixed Model Repeated Measures |
| Potential Clinical Importance |
| Pharmacodynamic |
| Protocol Deviation Management Plan |
| Physicians Global Assessment |
| Pharmacokinetic |
| Per Protocol |
| Program Safety Analysis Plan |
| Primary Sjogren's Syndrome |
| Patient Global Assessment |

## 2020N437857\_00

## CONFIDENTIAL

| _ | - | _ | _ | - | _ | _ | 1 |
|---|---|----|----|----|----|---|---|
| | _ | _ | | | | | |
| | つ | U. | 18 | ₹∠ | 12 | | |

| Abbreviation | Description |
|--------------|---------------------------------------------------------|
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |
| SAC | Statistical Analysis Complete |
| SAE | Serious Adverse Event |
| SE | Standard Error |
| SD | Standard Deviation |
| SOP | Standard Operation Procedure |
| SRDP | Study Results Dissemination Plan |
| SRT | Safety Review Team |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |
| VEO-PCO | Value, Evidence and Outcomes, Patient Centred Outcomes. |

## Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| BENLYSTA |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| MabThera |
| MedDRA |
| Rituxan |
| SAS |
| WinNonlin |

## 11.11.1. Columbia Suicide severity rate scale (CSSRS) post baseline

## COLUMBIA SUICIDE-SEVERITY RATING SCALE (C-SSRS)

| SUICIDAL IDEATION | |
|---|---|
| sk questions 1 and 2. If both are negative, proceed to "Suicida<br>the answer to question 2 is "yes," ask questions 3, 4 and 5. If t<br>nd/or 2 is "yes", complete "Intensity of Ideation" section. | the answer to question 1 Visit |
| CI - This section contained Clinical Outcome Assessment data contected by third party copyright laws and therefore have been except the content of the conte | ollection questionnaires or indices, which are cluded. |

| SUICIDAL IDEATION | | |
|---|---|---|
| | | Since Last<br>Visit |
| CCI - This section contained Clinical Outcome Assessment data or<br>protected by third party copyright laws and therefore have been ex | | dices, which are |
| | | - |
| US:ENG (United States/English) | IDSL Version 01.01 - 11 AUG 11 | [CSSRSV4.1 Since Last Visit] |

| Ideation Type | Type # (1-5) | Description of Ideation | Since Last<br>Visit |
|---|---|---|---|
| ost Severe Ideation | | | VISIT |
| - This section contained | Clinical Outcome Asses | sment data collection questionnaires or inc | dices, which are protect |
| nird party copyright laws | and therefore have been | 1 excluded. | |

| 1 71 | |
|---|---|
| INTENSITY OF IDEATION (Continued) | |
| | Since Last<br>Visit |
| | Most Severe |
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indiby third party copyright laws and therefore have been excluded. | ces, which are protected |
| by third party copyright laws and therefore have been excluded. | |
| US:ENG (United States/English) IDSL Version 01.01 - 11 AUG 11 INTENSITY OF IDEATION (Continued) | CSSRSV4.1 Since Last Visit |
| INVENSITY OF IDEATION (Continuous) | |
| | Since Last<br>Visit |
| | Most Severe |
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or ind protected by third party copyright laws and therefore have been excluded. | ices, which are |







### 11.11.2. Columbia Suicide severity rate scale (CSSRS) at baseline

### COLUMBIA SUICIDE-SEVERITY RATING SCALE (C-SSRS)



COLUMBIA SUICIDE-SEVERITY RATING SCALE (C-SSRS) (Continued) SUICIDAL IDEATION Lifetime: Current: Time He/She Felt Within Last Most Suicidal 6 Months US:ENG (United States/English) IDSL Version 01.00 - 20 MAY 11 [CSSRSV4.1 Baseline]

| SUICIDAL IDEATION | | |
|---|---|---|
| | Lifetime:<br>Time He/She Felt<br>Most Suicidal | Current:<br>Within Last<br>6 Months |
| CCI - This section contained Clinical Outcome Assessment data collection protected by third party copyright laws and therefore have been excluded | | es, which are |
| US:ENG (United States/English) | SL Version 01.00 - 20 MAY 11 | [CSSRSV4.1 Baseline] |

| INTENSITY OF IDEATION | | |
|---|---|---|
| CCI - This section contained Clinical Outcome Assessment data collect protected by third party copyright laws and therefore have been excluded. | tion questionnaires or indicaled. | es, which are |
| US:ENG (United States/English) | IDSL Version 01.00 - 20 MAY 11 | [CSSRSV4 1 Baseline] |

2020N437857\_00 201842

| | | - |
|---|---|---|
| INTENSITY OF IDEATION (Continued) | | |
| | Most Severe:<br>Lifetime | Most Severe:<br>Current |
| CCI - This section contained Clinical Outcome Assessment data collection que protected by third party copyright laws and therefore have been excluded. | estionnaires or indic | ces, which are |
| protected by third party copyright laws and therefore have been excluded. | | |
| US:ENG (United States/English) IDSL Versi | on 01.00 - 20 MAY 11 | TCSSPSV4 1 Receline |
| oo.eno (omeo omesengasi) | 20 1101 | [occitor III baseline |
| INTENSITY OF IDEATION (Continued) | | - |
| | Most Severe: | Most Severe: |
| CCL. This section contained Clinical Outcome Assessment data collection que | Lifetime | Current |
| CCI - This section contained Clinical Outcome Assessment data collection ques<br>protected by third party copyright laws and therefore have been excluded. | stiormanes or mulce | es, willcit are |
| IS:ENG (United States/English) IDSI Versin | on 01 00 - 20 MAV 11 | |


## COLUMBIA SUICIDE-SEVERITY RATING SCALE (C-SSRS) (Continued)



COLUMBIA SUICIDE-SEVERITY RATING SCALE (C-SSRS) (Continued)

| SUICIDAL BEHAVIOR (Continued) | | | Lifetime |
|---|---|---|---|
| CCI - This section contained Clinical Outcome Asses | sment data collection qu | estionnaires or in | dices, which are |
| protected by third party copyright laws and therefore | have been excluded. | | |
| JS:ENG (United States/English) | IDSI Vare | ion 01 00 - 20 MAV 11 | [CSSRSV4.1 Baseline |
| o.Erro (orned ordes/English) | IDOL VEIS | 01101.00 - 20 MAT 11 | (COOKOV4.1 Daseline |

| Answer for Actual Attempts Only | Most Recent<br>Attempt | Most Lethal<br>Attempt | Initial/First<br>Attempt |
|---|---|---|---|
| | - Accompt | Attompt | Attompt |
| Date: → | Day Month Year | Day Month Year | Day Month Year |
| CCI - This section contained Clinical Outcome Assessme<br>protected by third party copyright laws and therefore have | nt data collection que been excluded. | uestionnaires or in | dices, which are |
| , , , , , , , | | | |
| | | | - |
| US:ENG (United States/English) | IDSL Versi | on 01.00 - 20 MAY 11 | [CSSRSV4.1 Baseline] |

## 11.11.3. Eular Sjögren's syndrome disease activity index (ESSDAI)

## EULAR SJÖGREN'S SYNDROME DISEASE ACTIVITY INDEX (ESSDAI)\_Modified

| (LOODAI)_MOUNT | | | |
|---|---|---|---|
| Domain | Activity Level | Description | Abnormality currently<br>present and stable for<br>>12 months and due to<br>damage rather than<br>activity? If yes, indicate<br>level of involvement |
| Constitutional Exclusion of fever of infectious origin and voluntary weight loss | CCI - This section of collection questions party copyright laws | contained Clinical Outcome Assessment data<br>naires or indices, which are protected by third<br>s and therefore have been excluded. | |
| 2. Lymphadenopathy and lymphoma Exclusion of infection | | | |
| 3. Glandular Exclusion of stone or infection | | | |
| Articular Exclusion of osteoarthritis US:ENG (United States/English) | | IDCI Marries D4 00 | - 05 JAN 16 [ESSDAI_Modified] |

## EULAR SJÖGREN'S SYNDROME DISEASE ACTIVITY INDEX (ESSDAI)\_Modified (Continued)

| S. Cutaneous Rate as 'Wo activity' stable long-lasting features related to damage 6. Pulmonary Rate as 'No activity' stable long-lasting features related to damage, or respiratory involvement not related to the disease (tobacco use, etc.) COL - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. | Domain | Activity Level | Description | Abnormality currently present and stable for >12 months and due to damage rather than activity? If yes, indicate level of involvement |
|---|---|---|---|---|
| Rate as 'No activity' stable long-lasting features related to damage, or respiratory involvement not related to the disease | Rate as 'No activity'<br>stable long-lasting<br>features related to | or indices, which are | ontained Clinical Outcome Assessment data a protected by third party copyright laws and the protected by the protect | collection questionnaires<br>therefore have been |
| | Rate as 'No activity' stable long-lasting features related to damage, or respiratory involvement not related to the disease | | | |

2020N437857\_00 201842

# EULAR SJOGREN'S SYNDROME DISEASE ACTIVITY INDEX (ESSDAI)\_Modified (Continued)

| 7. Renal Rate as 'No activity' stable long-lasting features related to damage and renal involvement not related to the disease. If bigosy has been performed, please rate activity based on histological features first 8. Muscular Exclusion of weakness due to corticosteroids | Domain | Activity Level | Description | Abnormality currently |
|---|---|---|---|---|
| Rate as 'No activity' stable long-lasting features related to damage and renal involvement not related to the disease. If biopsy has been performed, please rate activity based on histological features first 8. Muscular Exclusion of weakness due to | | | | >12 months and due to<br>damage rather than<br>activity? If yes, indicate |
| Exclusion of weakness due to | Rate as 'No activity' stable long-lasting features related to damage and renal involvement not related to the disease. If biopsy has been performed, please rate activity based on histological features | CCI - This section of or indices, which are excluded. | ontained Clinical Outcome Assessment data a protected by third party copyright laws and | collection questionnaires therefore have been |
| US:ENG (United States/English) IDSL Version 01.00 - 05 JAN 16 [ESSDAI_Modified] | Exclusion of<br>weakness due to | | | |

2020N437857\_00 201842

## EULAR SJOGREN'S SYNDROME DISEASE ACTIVITY INDEX (ESSDAI)\_Modified (Continued)

| Domain | Activity Level | Description | Abnormality currently |
|---|---|---|---|
| | | | present and stable for |
| | | | >12 months and due to |
| | | | damage rather than<br>activity? If yes, indicate |
| | | | level of involvement |
| 9. PNS | CCI - This section co | ontained Clinical Outcome Assessment data | |
| Rate as 'No activity' | or indices, which are | ontained Clinical Outcome Assessment data<br>e protected by third party copyright laws and | I therefore have been |
| stable long-lasting | excluded. | | |
| features related to | | | |
| damage or PNS<br>involvement not | | | |
| related to the disease | | | |
| 10. CNS | | | |
| Rate as 'No activity'<br>stable long-lasting | | | |
| features related to | | | |
| damage or CNS | | | |
| involvement not | | | |
| related to the disease | | | |
| US:ENG (United States/English) | | IDSI Verries 04 00 | - 05 JAN 16 [ESSDAI_Modified] |
| US.ENG (United States/English) | | IDSL Version 01.00 | - 00 JAN 10 [ESSDAI_MODITED] |

2020N437857\_00 201842

## EULAR SJOGREN'S SYNDROME DISEASE ACTIVITY INDEX (ESSDAI)\_Modified (Continued)

| Domain | Activity Level | Description | Abnormality currently present and stable for >12 months and due to damage rather than activity? If yes, indicate level of involvement |
|---|---|---|---|
| 11. Haematological For anaemia, neutropenia, and thrombopenia, only autoimmune cytopenia must be considered Exclusion of vitamin or iron deficiency, drug-induced cytopenia | data collection que | contained Clinical Outcome Assessment estionnaires or indices, which are protected right laws and therefore have been | |
| 12. Biological US:ENG (United States/English) | | IDSL Version 01.00 | - 05 JAN 16 (ESSDAI_Modified) |

2020N437857\_00 201842

## 11.11.4. Neurological Symptoms

| | YES | NO |
|---|---|---|
| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. | | |

If any of the above are answered "Yes" at any visit, the investigator will contact the medical monitor.

Any neurological symptom that cannot be attributed to a concurrent medical condition or concomitant medication must be referred to a neurologist.

#### 11.11.5. Oral and Ocular dryness

### ORAL AND OCULAR DRYNESS SCALES



#### 11.11.6. Physician global assessment of disease activity (PGA)

#### PHYSICIAN GLOBAL ASSESSMENT OF DISEASE ACTIVITY



UK:ENG (United Kingdom/English)

Non-Standard [Physician Global Assessment of Disease Activity]

2020N437857 00 201842

### CONFIDENTIAL

#### 11.11.7. Eular Sjögren's syndrome patient reported index (ESSPRI)

## **EULAR SJÖGREN'S SYNDROME PATIENT REPORTED INDEX (ESSPRI)**



US:ENG (United States/English)

IDSL Version 01.00 - 22 APR 15 [ESSPRI]

## 11.11.8. Profile of fatigue and discomfort - SICCA symptoms inventory short form (PROFAD-SSI-SF)

## PROFILE OF FATIGUE AND DISCOMFORT - SICCA SYMPTOMS INVENTORY - SHORT FORM - 19 ITEM (PROFAD-SSI-SF)



PROFILE OF FATIGUE AND DISCOMFORT - SICCA SYMPTOMS INVENTORY - SHORT FORM - 19 ITEM (PROFAD-SSI-SF) (Continued)



2020N437857\_00 201842

IDSL Version 01.00 - 29 APR 15 [PROFAD-SSI-SF]

UK:ENG (United Kingdom/English)

### 11.11.9. Patient global assessment of disease activity (PtGA)

## PATIENT GLOBAL ASSESSMENT OF DISEASE ACTIVITY (PtGA)

Considering all of the ways your symptoms related to your Sjögren's syndrome (your dryness, your fatigue, your pain and your mental fatigue) are affecting you, how do you rate the severity of your Sjogren's syndrome now? (Select one number)

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

UK:ENG (United Kingdom/English)

Non-Standard [Patient Global Assessment of Disease Activity (PtGA)]

### 11.11.10. Sjogren's Allowable Medication Categories

| Medication Category | Rule |
|---|---|
| Anti-malarials | Set to "ANTIMALARIALS" if the preferred term begins with |
| | "QUINACRINE", "QUININE", "HYDROXYCHLOROQUINE", |
| | "MEPACRINE", or "CHLOROQUINE", "NOVOCHLOROQUINE" |
| | AND |
| | the route of administration is "ORAL" |
| Steroids | Set to 'STEROIDS' if at least one associated ATC code (ATCCD1 – |
| | ATCCD6) begins with 'H02' |
| | AND |
| | Route of administration is "ORAL" |
| Muscarinic agonists | Refer to Table 14 |

Table 14 Muscarinic agonists terms

| Term Name | Term Code |
|---|---|
| CARBACHOL + HYPROMELLOSE | 01175401 |
| PHENYLEPHRINE + PILOCARPINE | 00906001 |
| ACETYLCHOLINE | 00611301 |
| METIPRANOLOL HYDROCHLORIDE + PILOCARPINE HYDROCHLORIDE | 01482401 |
| PHENYLEPHRINE + PILOCARPINE NITRATE | 01309901 |
| PHENYLEPHRINE HYDROCHLORIDE + PILOCARPINE HYDROCHLORIDE | 00597501 |
| BORIC ACID + PILOCARPINE HYDROCHLORIDE + THIAMINE | 00937701 |
| HYDROCHLORIDE | |
| XANOMELINE | 01302901 |
| CARTEOLOL HYDROCHLORIDE + PILOCARPINE HYDROCHLORIDE | 40521001 |
| XANOMELINE TARTRATE | 01302902 |
| PILOCARPINE BORATE | 00043504 |
| METHACHOLINE | 00978001 |
| METHACHOLINE CHLORIDE | 00978002 |
| PILOCARPINE HYDROCHLORIDE + TIMOLOL MALEATE | 00971201 |
| CARBACHOL | 00060901 |
| EUPHRASIA EXTRACT + PILOCARPINE HYDROCHLORIDE + POTASSIUM | 01200001 |
| IODIDE | |
| ACECLIDINE HYDROCHLORIDE | 00189502 |
| ACETYLCHOLINE CHLORIDE | 00611302 |
| NAPHAZOLINE HYDROCHLORIDE + PILOCARPINE BORATE | 00981301 |
| NAPHAZOLINE HYDROCHLORIDE + NEOSTIGMINE BROMIDE + PILOCARPINE | 00280001 |
| HYDROCHLORIDE | |
| BETHANECHOL HYDROCHLORIDE | 00115903 |
| PILOCARPINE | 00043501 |
| PILOCARPINE HYDROCHLORIDE | 00043503 |
| EPINEPHRINE BITARTRATE + PILOCARPINE HYDROCHLORIDE | 00458001 |
| ACECLIDINE | 00189501 |
| NAPHAZOLINE HYDROCHLORIDE + PILOCARPINE BORATE + PILOCARPINE | 00981401 |
| HYDROCHLORIDE | 00570004 |
| PHYSOSTIGMINE SALICYLATE + PILOCARPINE HYDROCHLORIDE | 00578301 |
| PILOCARPINE NITRATE | 00043502 |
| BETHANECHOL CHLORIDE | 00115902 |
| BETHANECHOL HYDROCHLORIDE | 54486501 |
| BENZALKONIUM CHLORIDE + HYPROMELLOSE + PHENYLMERCURIC | 00221601 |
| NITRATE + PILOCARPINE HYDROCHLORIDE | 01017201 |
| PHYSOSTIGMINE + PILOCARPINE | 01017301 |
| BETHANECHOL | 00115901 |
| DIPIVEFRINE HYDROCHLORIDE + PILOCARPINE HYDROCHLORIDE | 53176901 |
| CEVIMELINE DIPLOMENTAL LINE DIPLOMENTAL | 01435201 |
| BENZALKONIUM CHLORIDE + DIPIVEFRINE HYDROCHLORIDE + | 01318101 |

| Term Name | Term Code |
|---------------------------|-----------|
| PILOCARPINE HYDROCHLORIDE | |
| CEVIMELINE HYDROCHLORIDE | 52131601 |

#### 11.11.11. Prednisone Conversion Factors

A concomitant medication is identified as a steroid if at least one associated ATC code (ATCCD1 – ATCCD6) begins with 'H02.'

The following routes are considered to provide systemic exposure: oral, subcutaneous, intramuscular, intradermal, and intravenous. Topical routes of administration are excluded (e.g., topical, conjunctival, intranasal).

At data base release all preferred terms identified with an ATC code beginning with 'H02' will be reviewed to ensure a conversion factor and dosing frequency exist for all terms with a systemic route of administration.

Similarly, all routes of administration for preferred terms with an ATC code beginning with 'H02' will be reviewed to ensure all systemic routes have been identified in the list above.

In order to be converted, the frequency and dose of the steroid must be present with the unit dose in milligrams (mg).

Reported dose for systemic steroid is converted to prednisone equivalent dose using conversion factor for each particular medication (refer to online calculator http://www.globalrph.com/corticocalc.htm).

Daily Prednisone Equivalent Dose (mg) = Collected Dose (mg) x Conversion Factor x Frequency Factor

| Preferred term | Conversion factor for converting to a prednisone-equivalent dose |
|---|---|
| BETAMETHASONE | 8.333 |
| BETAMETHASONE DIPROPIONATE | 8.333 |
| BETAMETHASONE SODIUM PHOSPHATE | 8.333 |
| BETAMETHASONE VAL | 8.333 |
| BETROSPAM | 8.333 |
| BUDESONIDE | 0.333 |
| CELESTONA BIFAS | 8.333 |
| CORTISONE | 0.2 |
| CORTISONE ACETATE | 0.2 |
| CRONOLEVEL | 8.333 |
| DEFLAZACORT | 0.8333 |
| DEPO-MEDROL MED LIDOKAIN | 1.25 |
| DEXAMETHASONE | 6.667 |
| DEXAMETHASONE ACETATE | 6.667 |
| DEXAMETHASONE SODIUM PHOSPHATE | 6.667 |

| FLUOCORTOLONE | 3 |
|---|---|
| HYDROCORTISONE | 0.25 |
| Preferred term | Conversion factor for converting to a prednisone-equivalent dose |
| HYDROCORTISONE ACETATE | 0.25 |
| HYDROCORTISONE SODIUM SUCCINATE | 0.25 |
| MEPREDNISONE | 1.25 |
| METHYLPREDNISOLONE | 1.25 |
| METHYLPREDNISOLONE ACEP | 1.25 |
| METHYLPREDNISOLONE ACETATE | 1.25 |
| METHYLPREDNISOLONE SODIUM SUCCINATE | 1.25 |
| PARAMETHASONE | 2.5 |
| PREDNISOLONE | 1 |
| PREDNISOLONE SODIUM PHOSPHATE | 1 |
| PREDNISOLONE SODIUM SUCCINATE | 1 |
| PREDNISONE | 1 |
| PREDNISONE ACETATE | 1 |
| TRIAMCINOLONE | 1.25 |
| TRIAMCINOLONE ACETATE | 1.25 |
| TRIAMCINOLONE ACETONIDE | 1.25 |

| Frequency Factors | |
|-------------------|--------|
| Frequency | Factor |
| BID | 2 |
| BIW | 2/7 |
| OAM | 1/30 |
| Once | 1 |
| One | 1 |
| OD | 1 |
| PRN | null |
| Q2H | 12 |
| Q2W | 1/14 |
| Q3H | 8 |
| Q3MO | 1/84 |
| Q3w | 1/21 |
| Q4H | 6 |
| Q4W | 1/28 |
| Q6H | 4 |
| Q8H | 3 |
| Q12H | 2 |
| QAM | 1 |
| QD | 1 |
| QH | 24 |
| QHS | 1 |

| Frequency Factors | |
|-------------------|------|
| QID | 4 |
| QM | 1 |
| QOD | 1/2 |
| QPM | 1 |
| QW | 1/7 |
| QWK | 1/7 |
| TID | 3 |
| TIW | 3/7 |
| UNK | Null |
| 2 TIMES PER WEEK | 2/7 |
| 3 TIMES PER WEEK | 3/7 |
| 4 TIMES PER WEEK | 4/7 |
| 5 TIMES PER WEEK | 5/7 |
| 5XWK | 5/7 |
| 5 TIMES PER DAY | 5 |
| EVERY 2 WEEKS | 1/14 |
| EVERY 3 WEEKS | 1/21 |
| EVERY 4 WEEKS | 1/28 |
| EVERY WEEK | 1/7 |

#### 11.11.12. Exit Interview

#### Instructions for Interviewer:

- At the beginning of the interview, please confirm the patient's study number.
- Text written in **bold** is to be read verbatim to each subject.
- Text written in [italics] is an instruction to the interviewer.
- Probes are to be used as needed to encourage the subject to provide full responses to each of the
  questions. They should be used if the subject gives an incomplete or unclear response or
  explanation with the initial question.
- Actively listen during the interview and take notes as necessary.

#### INTRODUCTION:

Hello, my name is [state first name] and I will be asking you some questions about your experience with medications in this study. The interview will be recorded and a transcript will be developed. In order to protect your confidentiality, only your study number will be included in the transcript. You are free to stop the interview at any time if you decide you no longer wish to participate.

The following questions have been developed to provide information on patient experiences with medications. It is important that you give your best answers, so please listen carefully to each question before you respond.

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by hird party copyright laws and therefore have been excluded. | |
|---|---|
| The party sopyright tares and anothers have been excluded. | |
| | _ |

| CCI - This section contained Clinical Outcome Assessment data collect<br>third party copyright laws and therefore have been excluded. | tion questionnaires or indices, which are protected by |
|---|---|
| third party copyright laws and therefore have been excluded. | |

| CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indic party copyright laws and therefore have been excluded. | ces, which are protected by third |
|---|---|

## 11.12. Appendix 12: Headline Results

## 11.12.1. Headline Results Output

The following tables will be included as headline results:

Table 15 Headline Results Output

| Table | Title |
|---|---|
| 1.1 | Summary of Subject Status and Reason for Study Withdrawal |
| 1.8 | Summary of Demographic Characteristics |
| 1.20 | Summary of Baseline Disease Activity |
| 2.11 | Summary of Statistical Analysis Results of Change from Baseline: ESSDAI Total Score (Corrected) |
| 2.19 | Summary of Responders on Total ESSDAI |
| 2.29 | Summary of Statistical Analysis Results of Change from Baseline: Stimulated Salivary Flow |
| 2.33 | Summary of Statistical Analysis Results of Change from Baseline: Oral Dryness Numeric Response Scale |
| 2.37 | Summary of Statistical Analysis Results of Percentage Change from Baseline in Core Salivary Gland Histology at Week 24 [1] |
| 2.38 | Summary of Bayesian Posterior Probabilities: ESSDAI Total Score (Corrected) [2] |
| 3.2 | Summary of All Adverse Events by System Organ Class and Preferred Term |
| 3.9 | Adverse Events of Special Interest by Category |
| 3.29 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) |
| 6.2 | Summary Statistics of Change from Baseline: ESSPRI Total Score and Domains |
| 6.4 | Summary of ESSPRI Responders |
| 6.11 | Summary of Bayesian Posterior Probabilities: ESSPRI Total Score [2] |
| 7.10 | Summary Statistics of Percentage Change from Baseline: Flow Cytometry Parameters [1] |
| | ummarize B cell (CD20)/mm2 in Salivary Gland<br>permits (generated by GSK) |

## 11.13. Appendix 13: List of Data Displays

### 11.13.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|---|---|---|
| Study Population | 1.1 to 1.22(EOS: 1.1001 to 1.1023) | N/A |
| Efficacy | 2.1 to 2.39 | to 2.12 |
| | 2.2 (EOS: 2.1001 to 2.1043) | (EOS: 2.1001 to 2.1011) |
| Safety | 3.1 to 3.62 | 3.1 to 3.4 |
| | (EOS: 3.1002 to 3.1062) | (EOS: 3.1001 to 3.1004) |
| Pharmacokinetic | 4.1 to 4.4 | 4.1 to 4.5 |
| | | (EOS: 4.1001 to 4.1002) |
| Pharmacokinetic/ | N/A 5.1 | |
| Pharmacodynamic | | |
| Health Outcomes | 6.1 to 6.14 | 6.1 to 6.3 |
| | (EOS: 6.1001 to 6.1015) | (EOS: 6.1001 to 6.1002) |
| Exploratory/Biomarker | 7.1 to 7.22 | 7.1 to 7.9 |
| | (EOS: 7.1001 to 7.1023) | (EOS: 7.1001 to 7.1009) |
| Section | Listings | |
| ICH Listings | 1 to 31 (EOS: 1002 to 1030) | |
| Other Listings | 32 to 58 (EOS: 1032 to 1061) | |

NOTE: For the End of Study Analysis reporting, selected Primary Analysis displays have been identified and will be generated. All displays generated for the End of Study Analysis will have unique numbering, and their display numbers have been indicated in parentheses in the list of displays.

#### 11.13.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and mock up displays are presented separately.

| Section | Figure | Table | Listing |
|---------------------------------|---------|---------|---------|
| Study Population | N/A | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | N/A | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic/Pharmacodynamic | PKPD_Fn | N/A | N/A |
| Exploratory/Biomarker | PD_Fn | | |

#### 11.13.3. Deliverables

| Delivery [Priority] | Description |
|---------------------|---------------------------------------------|
| HL[1] | Primary Analyses (Week 52) Headline Results |
| SAC_WK52 [2] | Primary Analysis (Week 52) SAC |
| SAC_EOS [3] | End of Study (Week 104) SAC |

#### NOTES:

• Unless otherwise specified in the Programming Notes, displays will be generated by Quanticate.

For the End of Study Analysis reporting, selected Primary Analysis displays have been identified and will be generated, using the final data. The displays will be updated (as required) to capture the additional visits and to reflect the final data. If further details are required, a RAP amendment or addendum will be generated to specify the changes. If' Per Protocol Population" not run, then no data will be reported".

This RAP details the planned analysis for both database freezes (Primary Analysis and End of Study Analysis), with the expectation of an observed treatment benefit being observed following the Primary Analysis.

In the event that the Primary Analysis reporting does not identify treatment benefit an abridged set of analysis may be conducted for the end of study analysis, which will be detailed in a RAP amendment or addendum.

2020N437857\_00 201842

## 11.13.4. Study Population Tables

| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Subject Dispos | ition | | | | • |
| 1.1.(1.1001) | Safety | POP_T1 | Summary of Subject Status and Reason for Study<br>Withdrawal | ICH E3, FDAAA, EudraCT EoS : Refer to mock shell POP_T1.1 | HL [1]<br>SAC_WK52 [2]<br>SAC_EOS [3] |
| 1.2.(1.1002) | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 Add Total column (if feasible) NOTE: Align with eCRF Footnote: Note: Treatment status with respective to Week 52 [1] Subjects may have only one primary reason. | SAC_WK52 [2]<br>SAC_EOS [3] |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements NOTE: Align with eCRF | SAC_WK52 [2] |
| 1.4. | Enrolled | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | EudraCT/Clinical Operations | SAC_WK52 [2] |
| Protocol Deviat | ion | | ' | <u>'</u> | • |
| 1.5. (1.1005) | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC_WK52 [2]<br>SAC_EOS [3] |

| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Population Ana | lysed | | | 1 | |
| 1.6. (1.006) | Safety | SP1 | Summary of Study Populations | IDSL | SAC_WK52 [2]<br>SAC_EoS [3] |
| 1.7. | Safety | SP2 | Summary of Exclusions from Per Protocol Population | | SAC_WK52 [2] |
| Demographics | | l | | | |
| 1.8. | Safety | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | HL [1]<br>SAC_WK52 [2] |
| 1.9. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | SAC_WK52 [2] |
| 1.10. | Safety | DM5 | Summary of Race and Racial Combinations | | SAC_WK52 [2] |
| 1.11. | Safety | FH1 | Summary of Family History of Cardiovascular Risk Factors | Footnote: Women <65 years or men < 55 years. Half siblings are considered first degree relatives | SAC_WK52 [2] |
| 1.12. | Safety | SU1 | Summary of Substance Use | | SAC_WK52 [2] |
| Medical Conditi | on & Con Med | ls | | | |
| 1.13. | Safety | MH4 | Summary of Medical Conditions (Sjögren Specific) | ISRC version with all medical conditions Ref eCRF and align | SAC_WK52 [2] |
| 1.14. | Safety | MH4 | Summary of Medical Conditions (non-Sjögren Specific) | | SAC_WK52 [2] |
| 1.15.(1.1015) | Safety | CM1 | Summary of Concomitant Medications | ICH E3 Add Total column (if feasible) | SAC_WK52 [2]<br>SAC_EOS [3] |

| Study Population Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 1.16.(1.1016) | Safety | CM1 | Summary of Most Frequently used Concomitant Medications by Generic Term | Footnote: Includes concomitant medications taken by >= 5% subjects Add Total column (if feasible) | SAC_WK52 [2]<br>SAC_EOS [3] |
| 1.17. | Safety | POP_T2 | Summary of Permitted pSS Medication Usage at Baseline | Add Total column (if feasible) | SAC_WK52 [2] |
| 1.18. | Safety | POP_T3 | Summary of Steroids, Anti-malarial and Muscarinic Agonists Use at Baseline | Add Total column (if feasible) | SAC_WK52 [2] |
| Disease History | ! | | | | |
| 1.19. | Safety | POP_T4 | Summary of AECG Classification Criteria Reported for Subjects at Baseline | Add Total column (if feasible) | SAC_WK52 [2] |
| 1.20. | Safety | POP_T5 | Summary of Baseline Disease Activity | Add Total column (if feasible) | HL [1]<br>SAC_WK52 [2] |
| 1.21. | Safety | POP_T6 | Summary of Autoantibody, Immunoglobulin, Complement, and Other Biomarker Measurements at Baseline | Add Total column (if feasible) | SAC_WK52 [2] |
| Other | | | | | |
| 1.22.(1.1022) | Safety | POP_T7 | Cumulative Study Withdrawal by Study Week | | SAC_WK52 [2]<br>SAC_EOS [3] |
| 1.1023. | Safety | POP_T8 | Summary of Overall Subject Status | | SAC_EOS [3] |

2020N437857\_00 201842

## 11.13.5. Efficacy Tables

| Efficacy: Tables | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ESSDAI Score | | | | | |
| 2.1.(2.1001) | Safety | EFF_T1 | Summary Statistics of ESSDAI Total Score (Uncorrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.2.(2.1002) | Per<br>Protocol | EFF_T1 | Summary Statistics of ESSDAI Total Score (Uncorrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.3. (2.1003) | Safety | EFF_T1 | Summary Statistics of ESSDAI Total Score (Corrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.4. (2.1004) | Per<br>Protocol | EFF_T1 | Summary Statistics of ESSDAI Total Score (Corrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.5. (2.1005) | Safety | EFF_T1 | Summary Statistics of Change from Baseline: ESSDAI Total Score (Uncorrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.6. (2.1006) | Per<br>Protocol | EFF_T1 | Summary Statistics of Change from Baseline: ESSDAI Total Score (Uncorrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.7.(2.1007) | Safety | EFF_T1 | Summary Statistics of Change from Baseline: ESSDAI Total Score (Corrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.8. (2.1008) | Per<br>Protocol | EFF_T1 | Summary Statistics of Change from Baseline: ESSDAI Total Score (Corrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.9. | Safety | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: ESSDAI Total Score (Uncorrected) | All visits to wk 52 entered to MMRM model. Note: Add the final model parameters | SAC_WK52 [2] |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10. | Per<br>Protocol | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: ESSDAI Total Score (Uncorrected) | All visits to wk 52 entered to MMRM model. Note: Add the final model parameters | SAC_WK52 [2] |
| 2.11. | Safety | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: ESSDAI Total Score (Corrected) | All visits to wk 52 entered to MMRM model. Note: Add the final model parameters | HL [1]<br>SAC_WK52 [2] |
| 2.12. | Per<br>Protocol | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: ESSDAI Total Score (Corrected) | All visits to wk 52 entered to MMRM model. Note: Add the final model parameters | SAC_WK52 [2] |
| 2.13.(2.1013) | Safety | EFF_T3 | Summary of ESSDAI Domain Activity (Uncorrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.14.(2.1014) | Per<br>Protocol | EFF_T3 | Summary of ESSDAI Domain Activity (Uncorrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2] |
| 2.15.(2.1015) | Safety | EFF_T3 | Summary of ESSDAI Domain Activity (Corrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.16.(2.1016) | Per<br>Protocol | EFF_T3 | Summary of ESSDAI Domain Activity (Corrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.17.(2.1017) | Safety | EFF_T4 | ESSDAI Improvement (At Least 1 Category on Domain Score) by Domain Among Subjects with Domain Involvement at Baseline (Corrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.18.(2.1018) | Safety | EFF_T5 | ESSDAI Worsening (At Least 1 Category on Domain Score) by Domain (Corrected) | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.19.(2.1019) | Safety | EFF_T6 | Summary of Responders on Total ESSDAI Score (Corrected) | Corrected ESSDAI score will be used.<br>Include all visits up to Week 68 | HL [1]<br>SAC_WK52 [2] |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | EoS: Include all scheduled visits Footnote: Responders are defined as below: Responder 1: ≥5 point reduction in ESSDAI Total vs baseline Responder 2: ≥3 point reduction in ESSDAI Total vs baseline Responder 3: ≥3 point reduction in ESSDAI Total vs baseline and Total Score < 5 Responder 4: Total score < 5 | SAC_EOS [3] |
| 2.20.(2.1020) | Per<br>Protocol | EFF_T6 | Summary of Responders on Total ESSDAI Score (Corrected) | Corrected ESSDAI score will be used. Include all visits up to Week 68 EoS: Include all scheduled visits Footnote: Responders are defined as below: Responder 1: ≥5 point reduction in ESSDAI Total vs baseline Responder 2: ≥3 point reduction in ESSDAI Total vs baseline Responder 3: ≥3 point reduction in ESSDAI Total vs baseline Responder 4: Total Score < 5 Responder 4: Total Score < 5 Footnote to include model parameter as per mock table | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.21. | Safety | EFF_T7 | Summary of Statistical Analysis of Responder on Total ESSDAI Score (Corrected) | Footnote: Responder definition and include footnotes as per EFF_T7 Note: Add the final model parameters | SAC_WK52 [2] |

| Efficacy: Tables | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.22.(2.1022) | Safety | EFF_T8 | Proportion of Subjects with Damage by Domain | Additional Supplementary to ESSDAI for 5 domains EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| ClinESSDAI Sco | ore | | | | |
| 2.23.(2.1023) | Safety | EFF_T1 | Summary Statistics: ClinESSDAI Total Score (Corrected) | Corrected ESSDAI score will be used. Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.24.(2.1024) | Safety | EFF_T1 | Summary Statistics of Change from Baseline:<br>ClinESSDAI Total Score (Corrected) | Corrected ESSDAI score will be used. Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.25.(2.1025) | Safety | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: ClinESSDAI Total Score (Corrected) | Corrected ESSDAI score will be used. All visits to wk 52 entered to MMRM model. Note: Add the final model parameters | SAC_WK52 [2] |
| 2.26.(2.1026) | Safety | EFF_T6 | Summary of ClinESSDAI Responders (Corrected) | Corrected ESSDAI score will be used. Including just one section with Responder Criteria: Reduction from baseline ≥3 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| Stimulated and | Unstimulated | Salivary Flow | r | | |
| 2.27.(2.1027) | Safety | EFF_T1 | Summary Statistics of Stimulated and Unstimulated Salivary Flow | Include all visits up to Week 68 EoS: Include all scheduled visits Page by parameter – stimulated and unstimulated flow | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.28.(2.1028) | Safety | EFF_T1 | Summary Statistics of Change from Baseline:<br>Stimulated and Unstimulated Salivary Flow | Include all visits up to Week 68 EoS: Include all scheduled visits by parameter | SAC_WK52 [2]<br>SAC_EOS [3] |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | Page by parameter – stimulated and unstimulated flow | |
| 2.29. | Safety | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: Stimulated Salivary Flow | All visits to wk 52 entered to MMRM model. Note: Add the final model parameters | HL [1]<br>SAC_WK52 [2] |
| 2.30. | Per<br>Protocol | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: Stimulated Salivary Flow | All visits to wk 52 entered to MMRM model. Note: Add the final model parameters | SAC_WK52 [2] |
| Oral Dryness | | | | | |
| 2.31.(2.1031) | Safety | EFF_T1 | Summary Statistics of Oral Dryness Numeric Response Scale | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.32.(2.1032) | Safety | EFF_T1 | Summary Statistics of Change from Baseline: Oral Dryness Numeric Response Scale | Include all visits up to Week 68 EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.33. | Safety | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: Oral Dryness Numeric Response Scale | All visits to wk 52 entered to MMRM model<br>Note: Add the final model parameters | HL [1]<br>SAC_WK52 [2] |
| 2.34. | Per<br>Protocol | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: Oral Dryness Numeric Response Scale | All visits to wk 52 entered to MMRM model. Note: Add the final model parameters | SAC_WK52 [2] |

| Efficacy: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Salivary Gland | Histology | • | | | |
| 2.35.(2.1035) | Safety | EFF_T9 | Summary Statistics for Salivary Gland Histology<br>Assessments | Includes baseline and Week 24 only Include all parameters as specified in RAP Table 13 Note: Include Week 52 for EoS reporting | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.36.(2.1036) | Safety | EFF_T9 | Summary Statistics of Percentage Change from Baseline: Salivary Gland Histology Assessments EOS: Summary Statistics of Change from Baseline: Salivary Gland Histology Assessments | Includes only Week 24 data Include all parameters as specified in RAP Table 13 Note: Include Week 52 for EoS reporting | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.37.(2.1037) | Safety | EFF_T10 | Summary of Statistical Analysis Results of Percentage<br>Change from Baseline in Core Salivary Gland Histology<br>at Week 24 EOS: Summary of Statistical Analysis Results of Change<br>from Baseline in Core Salivary Gland Histology at<br>Week 24 | Parameters to be included in the analysis are B cell (CD20) count/mm² Lymphocyte Focus Score (per 4mm²) B (CD20) / T (CD3) cell ratio Plasma cell (CD138+; both - CD20pos and CD20neg) count/mm² Note: Exclude Week 52 for EoS reporting (i.e. only n=6 samples). | HL [1]<br>SAC_WK52 [2]<br>SAC_EOS [3] |
| Further Efficacy | / Evaluation | <u>'</u> | | | |
| 2.38. | Safety | EFF_T11 | Summary of Bayesian Posterior Probabilities: ESSDAI Total Score (Corrected) | Add appropriate footnotes based on final out To be generated by GSK | HL [1]<br>SAC_WK52 [2] |

| Efficacy: Tables | 5 | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| <b>Further Evaluat</b> | ion | | | | |
| 2.39.(2.1039) | Safety | N/A | Summary of Responders on Total ESSDAI Score | EoS: Include all scheduled visits % responders calculated using n for each visit EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| (2.1040) | Completer | EFF_T1 | Summary Statistics of ESSDAI Total Score (Corrected) – Completer | Include all scheduled visits Add footnote: Note: Completer is defined as "Subjects who completed the 52 Week treatment visits AND general follow up phase of the study including the visit at Week 68" | SAC_EOS [3] |
| (2.1041) | Completer | EFF_T2 | Summary of Statistical Analysis Results of Change from Baseline: ESSDAI Total Score (Corrected) - Completer | Include visits upto and including Week 68/FU Add footnote: As T2.1040 | SAC_EOS [3] |
| (2.1042) | Completer | EFF_T1 | Summary Statistics of Stimulated and Unstimulated Salivary Flow - Completer | Include all scheduled visits Page by parameter – stimulated and unstimulated flow Add footnote: As T2.1040 | SAC_EOS [3] |
| (2.1043) | Completer | EFF_T1 | Summary Statistics of Oral Dryness Numeric Response<br>Scale - Completer | Include all scheduled visits Add footnote: As T2.1040 | SAC_EOS [3] |

2020N437857\_00 201842

## 11.13.6. Efficacy Figures

| Efficacy: Figure | es | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ESSDAI | l. | • | | ' | |
| 2.1.(2.1001) | Safety | EFF_F1 | Mean (± SE) of ESSDAI Total Score (Uncorrected) | All scheduled visits Legend: Treatment EoS: Include all visits up to Week 68/FU. X-axis: Add line break between Week 52 and Week 68/FU with no joining lines. | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.2.(2.1002) | Safety | EFF_F1 | Mean (± SE) of ESSDAI Total Score (Corrected) | All scheduled visits<br>Legend: Treatment<br>EoS: As F2.1001 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.3. (2.1003) | Safety | EFF_F1 | Mean (± SE) of Change from Baseline in ESSDAI Total Score (Uncorrected) | All scheduled visits<br>Legend: Treatment<br>EoS: As F2.1001 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.4. (2.1004) | Safety | EFF_F1 | Mean (± SE) of Change from Baseline in ESSDAI Total Score (Corrected) | All scheduled visits<br>Legend: Treatment<br>EoS: As F2.1001 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.5. | Safety | EFF_F1 | Adjusted Mean (95% CI) Change from Baseline: ESSDAI Total Score (Uncorrected) | Panel: Rows = 1 by Cols = 1 for parameter X-Axis: Visit: Continuous Scale Y-Axis: ESSDAI total Score and scaled accordingly Legend: Treatment Include all visits to Week 52 Note: Add the final model parameters | SAC_WK52 [2] |
| 2.6. | Safety | EFF_F1 | Adjusted Mean (95% CI) Change from Baseline: ESSDAI Total Score (Corrected) | Panel: Rows = 1 by Cols = 1 for parameter X-Axis: Visit: Continuous Scale Y-Axis: ESSDAI total Score and scaled | SAC_WK52 [2]<br>SAC_EOS [3] |

| Efficacy: Figure | es | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | | accordingly Legend: Treatment Include all visits to Week 52 Note: Add the final model parameters | |
| 2.7. (2.1007) | Safety | EFF_F2 | ESSDAI Activity by Domain | Page By: Domain Panel: Visit (Include only Baseline, Week 24 and Week 52) EoS: Panel: Visit (Include only Baseline, Week 24 & Week 52) X-Axis = Treatment Y-Axis = Percentage of Subjects Stacked bar chart SAS colors for the categories are No Activity - CXDCDCDC Low Activity - CX9370DB Moderate Activity - CX7FFF00 High Activity - CXFF8C00 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.8. (2.1008) | Safety | EFF_F3 | ESSDAI Responders Bar Chart by Treatment and Visit (Corrected) | EoS: Include all scheduled visits except IFU, EW & W68/FU Footnote: Responders are defined as below: Responder 1: ≥5 point reduction in ESSDAI Total vs baseline Responder 2: ≥3 point reduction in ESSDAI Total vs baseline Responder 3: ≥3 point reduction in ESSDAI Total vs baseline and Total Score < 5 Responder 4: Total Score < 5 | SAC_WK52 [2]<br>SAC_EOS [3] |
| Efficacy: Figure | es | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Stimulated & U | nstimulated Sa | alivary Flow | | | |
| 2.9. (2.1009) | Safety | EFF_F1 | Mean (+/- SE) of Change from Baseline in Stimulated Salivary Flow | EoS: As F2.1001 Panel: Rows = 1 by Cols = 1 for parameter X-Axis: Visit: Continuous Scale Legend: Treatment | SAC_WK52 [2]<br>SAC_EOS [3] |
| 2.10.(2.1010) | Safety | EFF_F1 | Mean (+/- SE) of Change from Baseline in Unstimulated Salivary Flow | As F2.1001<br>Legend: Treatment | SAC_WK52 [2]<br>SAC_EOS [3] |
| Oral Dryness | | • | | | |
| 2.11.(2.1011) | Safety | EFF_F1 | Mean (+/- SE) of Change from Baseline in Oral Dryness<br>Numeric Response | EoS: As F2.1001 Panel: Rows = 1 by Cols = 1 for parameter X-Axis: Visit: Continuous Scale Y-Axis: Oral dryness numeric response and scaled accordingly Legend: Treatment | SAC_WK52 [2]<br>SAC_EOS [3] |
| Salivary Gland | Histology | | | | |
| 2.12.<br>(2.1012) | Safety | EFF_F4 | Median (+/- IQR) of Percentage Change from Baseline in Salivary Gland Core Parameters EoS: Median (+/- IQR) of Change from Baseline in Salivary Gland Core Parameters | Percentage change (Primary) and change (EoS) to wk 24 for B cell (CD20) count/mm2 Lymphocyte Focus Score (in 4mm²) B (CD20) / T (CD3) cell ratio Plasma cell (CD138+; both - CD20pos and CD20neg) count/mm² X-Axis: Week 24 visit only Legend: Treatment NOTE: Limited sample at WK52 (i.e. n=6), hence Week 52 not required for EoS. | SAC_WK52 [2]<br>SAC_EOS [3] |

| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Exploratory ( | Correlation Evalu | uation | | | |
| 2.13. | Safety | PD_F1 | ESSDAI and ClinESSDAI Bland-Altman Plot at Week 24 (Corrected) | Panel: Rows = 1 by Cols = 1 for parameter X-Axis: Average of Change from baseline to Wk24 Total ClinESSDAI and Change from baseline to wk 24 Total ESSDAI Y-Axis: Difference of Change from baseline to Wk24 Total ESSDAI and Change from baseline to wk 24 Clin ESSDAI Legend: Treatment Note: Add footnotes as required Note: For SAC_EOS [3]: Include other timepoints and add identifies | SAC_WK52 [2] |
| 2.14. | Safety | PD_F2 | Scatter Plot of Wk 24 Changes for Total ESSDAI Score vs<br>Salivary Gland B Cells | Panel: Rows = 1 by Cols = 1 for parameter X-Axis: Percentage Change from baseline to Wk24 Salivary Gland B Cells Y-Axis: Change from baseline to Wk24 Total ESSDAI Legend: Treatment | SAC_WK52 [2] |
| 2.15. | Safety | PD_F3 | Median Free Blys Vs Median CD19+ B cell by Treatment | Panel per Treatment. Legend: Visit X-axis: CD19+ B cells Y-axis: Free Blys B Cell measured by flow cytometry | SAC_WK52 [2] |

2020N437857\_00 201842

## 11.13.7. Safety Tables

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Exposure | 1 | | | | |
| 3.1. | Safety | SAFE_T15 | Summary of Extent of Exposure | | SAC_WK52 [2] |
| Adverse Events | s (AEs) | | | , | |
| 3.2. (3.1002) | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 Footnote: Note: Subjects are counted only once per SOC/PT EoS: Include visits upto W68/FU EoS Footnote: Note: Includes Treatment & General Follow Up periods only. | HL [1]<br>SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.3. (3.1003) | Safety | AE1 | Summary of All Adverse Events by System Organ Class | Excludes Preferred Term breakdown Footnote: Note: Subjects are counted only once per SOC EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.4. (3.1004) | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | ICH E3 EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.5. (3.1005) | Safety | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events | ICH E3 | SAC_WK52 [2] |

| Safety: Tables | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | | | by Overall Frequency | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_EOS [3] |

| No. | Population | IDSL / TST | Title | Programming Notes | Deliverable |
|---|---|---|---|---|---|
| | | Example<br>Shell | | | [Priority] |
| 3.6. (3.1006) | Safety | AE1 | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.7. (3.1007) | Safety | AE15 | Summary of Common (>=5%) Non Serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Participant and Occurrences) | FDAAA EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.8. (3.1008) | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4<br>Adverse Events by Overall Frequency | ICH E3 EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.9. (3.1009) | Safety | SAFE_T7 | Adverse Events of Special Interest by Category | Includes events defined in Belimumab PSAP and study specific special interest events EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | HL [1]<br>SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.10. (3.1010) | Safety | SAFE_T8 | Malignant Neoplasm Adverse Events of Special Interest by Category and PT | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.11. (3.1011) | Safety | SAFE_T9 | Post-Administration Systemic Reaction Adverse Events of Special Interest by Category and PT | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.12. (3.1012) | Safety | SAFE_T9 | Serious Post-Administration Systemic Reaction Adverse Events of Special Interest by Category and PT | Change title and content so only Serious PASR's are summarized EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.13. | Safety | SAFE_T10 | Post-Injection Systemic Reactions per Anaphylactic Reactions CMQ Broad search by PT, in First Six Doses of Belimumab/Placebo | All infusion column would include the overall study treatment | SAC_WK52 [2] |
| 3.14. | Safety | SAFE_T10 | Serious Post-Injection Systemic Reactions per<br>Anaphylactic Reactions CMQ Broad search by PT, in<br>First Six Doses of Belimumab/Placebo | All infusion column would include the overall study treatment | SAC_WK52 [2] |
| 3.15. | Safety | SAFE_T10 | Serious Acute Post-Injection Systemic Reactions per<br>GSK Adjudication by PT, in First Six Doses of<br>Belimumab/Placebo | All infusion column would include the overall study treatment | SAC_WK52 [2] |
| 3.16. | Safety | SAFE_T10 | Serious Delayed Acute Post-Injection Systemic<br>Reactions per GSK Adjudication by PT, in First Six Doses<br>of Belimumab/Placebo | All infusion column would include the overall study treatment | SAC_WK52 [2] |
| 3.17. | Safety | SAFE_T10 | Serious Delayed Non-Acute Post-Injection Systemic<br>Reactions per GSK Adjudication by PT, in First Six Doses<br>of Belimumab/Placebo | All infusion column would include the overall study treatment | SAC_WK52 [2] |
| 3.18. (3.1018) | Safety | SAFE_T11 | Infection Adverse Events of Special Interest by Category and PT | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.19. (3.1019) | Safety | SAFE_T11 | Infection Adverse Events of Special Interest Leading to Study Agent Discontinuation by Category and PT by Category and PT | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.20. (3.1020) | Safety | SAFE_T12 | Depression/Suicide/Self-injury Adverse Events of Special Interest by Category and PT | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.21. (3.1021) | Safety | SAFE_T13 | Severe Skin Reactions Adverse Events of Special Interest by Preferred Term | Study specific AESI EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.22. (3.1022) | Safety | SAFE_T13 | Cardiac Disorders Adverse Events of Special Interest by Preferred Term | Study specific AESI EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.23. (3.1023) | Safety | SAFE_T13 | Posterior Reversible Encephalopathy Syndrome (PRES)<br>Adverse Events of Special Interest by Preferred Term | Study specific AESI EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.24. (3.1024) | Safety | SAFE_T13 | Progressive Multifocal Leukocephalopathy (PML) Adverse Events of Special Interest by Preferred Term | Study specific AESI EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.25. (3.1025) | Safety | SAFE_T13 | Biopsy Adverse Events of Special Interest by Preferred Term | Study specific AESI EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.26. (3.1026) | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class and Preferred Term | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.27. (3.1027) | Safety | AE1 | Summary of Serious Adverse Events by System Organ Class | No preferred term breakdown EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.28. (3.1028) | Safety | AE1 | Summary of Adverse Events Leading to Discontinuation of Study Treatment or Withdrawal from Study by System Organ Class and Preferred Term | EACTRCD and AEWD EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.29. (3.1029) | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | FDAAA, EudraCT EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | HL [1]<br>SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.30. (3.1030) | Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by<br>System Organ Class and Preferred Term | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.31. (3.1031) | Safety | AE1 | Summary of Fatal Adverse Events by System Organ Class and Preferred Term | EoS: Include visits upto W68/FU EoS Footnote: Add as T3.1002 | SAC_WK52 [2]<br>SAC_EOS [3] |
| Labs | | | | | |
| 3.32. (3.1032) | Safety | LB1 | Summary of Hematology Laboratory Values | EoS: Include all scheduled visits Add footnote: Basophils% = % of leukocytes; Eosinophils% = % of leukocytes | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.33. (3.1033) | Safety | LB1 | Summary of Hematology Changes from Baseline | EoS: Include all scheduled visits ICH E3 Includes baseline values. Add footnote: Basophils% = % of leukocytes; Eosinophils% = % of leukocytes | SAC_WK52 [2]<br>SAC_EOS [3] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.34. (3.1034) | Safety | SAFE_T5 | Laboratory Reference Range Shifts from Baseline: Hematology | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.35. (3.1035) | Safety | SAFE_T1 | Worst Laboratory Toxicity Grade: Hematology | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.36. (3.1036) | Safety | SAFE_T2 | Laboratory Toxicity Grade Worsening of at Least 2 Grades from Baseline: Hematology | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.37. (3.1037) | Safety | LB1 | Summary of Clinical Chemistry Laboratory Values | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.38. (3.1038) | Safety | LB1 | Summary of Changes from Baseline: Clinical Chemistry Laboratory Values | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.39. (3.1039) | Safety | SAFE_T1 | Worst Laboratory Toxicity Grade: Clinical Chemistry | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.40. (3.1040) | Safety | SAFE_T2 | Laboratory Toxicity Grade Worsening of at Least 2<br>Grades from Baseline: Clinical Chemistry | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.41. (3.1041) | Safety | SAFE_T6 | Summary of Liver Assessments | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.42. (3.1042) | Safety | UR3 | Summary of Urinalysis Dipstick Results | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |

| Safety: Tables | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.43. (3.1043) | Safety | LB1 | Summary of Protein/Creatinine Ratio | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.44. (3.1044) | Safety | LB1 | Summary of Immunoglobulins by Visit | EoS: Include all scheduled visits Page by parameter: IgG, IgA, IgM, | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.45. (3.1045) | Safety | LB1 | Summary of Change from Baseline in Immunoglobulins by Visit | EoS: Include all scheduled visits Page by parameter: IgG, IgA, IgM, | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.46. (3.1046) | Safety | SAFE_T1 | Worst Laboratory Toxicity Grade: Immunoglobulin | EoS: Include all scheduled visits Includes IgG only Include footnote for baseline | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.47. (3.1047) | Safety | SAFE_T2 | Laboratory Toxicity Grade Worsening of at Least 2<br>Grades from Baseline: Immunoglobulin | EoS: Include all scheduled visits Includes IgG only Include footnote for baseline | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.48. (3.1048) | Safety | SAFE_T4 | Immunoglobulins below LLN | EoS: Include all scheduled visits Page by parameter: IgG, IgA, IgM, | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.49. (3.1049) | Safety | SAFE_T4 | Immunoglobulins above ULN | EoS: Include all scheduled visits Page by parameter: IgG, IgA, IgM, | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.50. (3.1050) | Safety | LB1 | Summary of C-Reactive Protein | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.51. (3.1051) | Safety | LB1 | Summary of Changes from Baseline in C-Reactive Protein | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Signs | | | | | • |
| 3.52. (3.1052) | Safety | VS1 | Summary of Vital Signs | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.53. (3.1053) | Safety | VS1 | Summary of Change from Baseline for Vital Signs | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| ECG | | | | | |
| 3.54. | Safety | EG1 | Summary of ECG Findings | Screening Visit Only | SAC_WK52 [2] |
| 3.55. | Safety | EG2 | Summary of Screening ECG | Include all intervals | SAC_WK52 [2] |
| TBNK | | | | | |
| 3.56. (3.1056) | Safety | LB1 | Summary of CD4 and CD8 | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.57. (3.1057) | Safety | LB1 | Summary of Changes from Baseline in CD4 and CD8 | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |

| Safety: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Neurological Sy | mptoms | | | | |
| 3.58. (3.1058) | Safety | SAFE_T3 | Summary of Neurological Symptoms | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| Columbia-Suici | de Severity Ra | ating Scale | | | |
| 3.59. (3.1059) | Safety | ECSSRS1 | Summary of C-SSRS Suicidal Ideation or Behaviour During Treatment | EoS: Include all scheduled visits Include summaries for both lifetime and current state. | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.60. (3.1060) | Safety | ECSSRS2 | Summary of Treatment-Emergent C-SSRS Suicidal Ideation or Behaviour Relative to Pre-treatment | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.61. (3.1061) | Safety | ECSSRS3 | Shift Table of Changes in C-SSRS Categories from Pre-<br>Treatment to On-Treatment | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| Immunogenicity | / | | | | • |
| 3.62. (3.1062) | Safety | SAFE_T14 | Summary of Immunogenic Response by Visit | EoS: Include all scheduled visits Belimumab antibodies Rituximab antibodies EoS Footnote: For anti-Rituximab, baseline is Week 8 | SAC_WK52 [2]<br>SAC_EOS [3] |
| Further Analyse | es | | | | |
| 3.1063 | Safety | SAFE_10 | Post-IV Systemic Reactions per Anaphylactic Reactions CMQ Broad search by PT, in First Two 2 Infusions of Rituximab/Placebo | All infusion column would include the overall study treatment | SAC_EOS [3] |

2020N437857\_00 201842

# 11.13.8. Safety Figures

| Safety: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Lab | | | | | • |
| 3.1 (3.1001) | Safety | EFF_F1 | Mean (+/- SE) of Hematology | EoS: As F2.1001 Parameters for SAC: WBC count, Neutrophil counts, Haemoglobin, Platelets, Lymphocytes, Hematocrit, Monocytes, Eosinophils, Basophils All visits contained with the summary source table, with Day 0 being included as part of the plot | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.2 (3.1002) | Safety | EFF_F4 | Median (+/- IQR) of Immunoglobulins | EoS: As F2.1001 x-axis is visit, line per treatment group. | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.3 (3.1003) | Safety | EFF_F4 | Median (+/- IQR) of Change from baseline of Immunoglobulins | EoS: As F2.1001<br>x-axis is visit, panel per treatment group.<br>Include IgG, IgA and IgM. | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3.4 (3.1004) | Safety | EFF_F1 | Median (+/- IQR) of Absolute Values of CD4 and CD8 | EoS: As F2.1001 x-axis is visit, line per treatment group. | SAC_WK52 [2]<br>SAC_EOS [3] |

2020N437857\_00 201842

## 11.13.9. Pharmacokinetic Tables

| Pharmacokine | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Concentra | tion Data | | | | |
| 4.1. | PK-B | PK01 | Summary of Plasma Belimumab Pharmacokinetic Concentration-Time Data (ng/mL) | Include 3 columns: Combination, Belimumab, Total | SAC_WK52 [2] |
| 4.2. | PK-B | PK01 | Summary of Plasma Belimumab Pharmacokinetic<br>Concentration-Time Data (µg/mL) by Baseline Body Weight<br>Quartiles | Include 3 columns: Combination, Belimumab, Total | SAC_WK52 [2] |
| 4.3. | PK-R | PK01 | Summary of Plasma Rituximab Pharmacokinetic Concentration-Time Data (ng/mL) | Include 3 columns: Combination, Rituximab, Total | SAC_WK52 [2] |
| 4.4. | PK-B | PK01 | Summary of Plasma Belimumab Pharmacokinetic<br>Concentration-Time Data (µg/mL) by Belimumab<br>Immunogenicity Status | Include 3 columns: Combination, Belimumab, Total Produce if ≥6 subjects in total have positive belimumab immunogenicity. | SAC_WK52 [2] |

2020N437857\_00 201842

# 11.13.10. Pharmacokinetic Figures

| Pharmacokinetic: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>TST ID /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individual Plots | | | | | |
| 4.1. (4.1001) | PK-B | PKCF1P | Individual Belimumab Plasma Concentration-Time Plot by Treatment (Linear and Semi-Log) | Paginate by Treatment Combo and Bel Arms NOTE: Ensure treatment legends can be differentiated | SAC_EOS [3] |
| 4.2. (4.1002) | PK-R | PKCF1P | Individual Rituximab Plasma Concentration-Time Plot by Treatment (Linear and Semi-Log) | Paginate by Treatment Combo and Ritux Arms NOTE: Ensure treatment legends can be differentiated | SAC_EOS [3] |
| Median Plots | 1 | <u> </u> | | | |
| 4.3. | PK-B | PKCF3 | Median Plasma Belimumab Concentration-Time Plots by Treatment (Linear and Semi-log) | Combo and Bel Arms | SAC_WK52 [2] |
| 4.4. | PK-B | PKCF3 | Median Plasma Belimumab Concentration-Time Plots by Body Weight Quartile (Linear and Semi-log) | Combo and Bel Arms | SAC_WK52 [2] |
| 4.5. | PK-R | PKCF3 | Median Plasma Rituximab Concentration-Time Plots by Treatment (Linear and Semi-log) | Combo and Ritux Arms | SAC_WK52 [2] |

2020N437857\_00 201842

## 11.13.11. Pharmacokinetic / Pharmacodynamic Figures

| Pharmacokineti | Pharmacokinetic / Pharmacodynamic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 5.1. | Safety | PKPD_F1 | Scatterplot of CD19+ B cells Versus Belimumab Concentration | 2 panels: combo and bel Individual subject data y-axis=CD19+ B cells (from TBNK panel CONC record) x-axis=Belimumab concentration | SAC_WK52 [2] |

2020N437857\_00 201842

### 11.13.12. Health Outcomes Tables

| Health Outcome | Health Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ESSPRI Score | | | | · | |
| 6.1. (6.1001) | Safety | EFF_T1 | Summary Statistics of ESSPRI Total Score and Domains | EoS: Include all scheduled visits Summarize for both the overall score and 3 domains (dryness, fatigue and pain) | SAC_WK52 [2]<br>SAC_EOS [3] |
| 6.2. (6.1002) | Safety | EFF_T1 | Summary Statistics of Change from Baseline:<br>ESSPRI Total Score and Domains | EoS: Include all scheduled visits Summarized for both the overall score and 3 domains (dryness, fatigue and pain) | HL [1]<br>SAC_WK52 [2]<br>SAC_EOS [3] |
| 6.3. (6.1003) | Per<br>Protocol | EFF_T1 | Summary Statistics of Change from Baseline:<br>ESSPRI Total Score and Domains | EoS: Include all scheduled visits Summarized for both the overall score and 3 domains (dryness, fatigue and pain) | SAC_WK52 [2]<br>SAC_EOS [3] |
| 6.4. (6.1004) | Safety | EFF_T4 | Summary of ESSPRI Responders | EoS: Include all scheduled visits Footnote: Responder 1: Decrease in the ESSPRI total score of at least one point or at least 15% compared to baseline | HL [1]<br>SAC_WK52 [2]<br>SAC_EOS [3] |
| 6.5. (6.1005) | Per<br>Protocol | EFF_T4 | Summary of ESSPRI Responders | EoS: Include all scheduled visits Footnote: Responder 1: Decrease in the ESSPRI total score of at least one point or at least 15% compared to baseline | SAC_WK52 [2]<br>SAC_EOS [3] |

| Health Outcome | Health Outcomes: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.6. | Safety | EFF_T7 | Summary of Statistical Analysis of Responders on ESSPRI | Footnote: Responder 1: Decrease in the ESSPRI total score of at least one point or at least 15% compared to baseline Responder 2: Subjects with baseline score of >= 5 and Total ESSPRI score of < 5. The denominator for percentages at each visit are the subjects who had a score >= 5 at baseline. Note: Add the final model parameters | SAC_WK52 [2] |
| PROFAD SSI SF | = | | | | |
| 6.7. | Safety | EFF_T1 | Summary Statistics of PROFAD SSI SF Subscores | Summarize for the 3 subscores (PROF, PROFAD, SSI) Footnote (if feasible): 1. PROF is calculated as the sum of domains Somatic fatigue and Mental fatigue 2. PROFAD is calculated as the sum of domains Somatic fatigue, Mental fatigue, Arthralgia and Vascular 3. SSI is calculated as the sum of domains Cutaneous dryness, Vaginal dryness, Ocular dryness and Oral dryness. The SSI subscore is derived for females only. | SAC_WK52 [2] |

| Health Outcom | es: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.8. | Safety | EFF_T1 | Summary Statistics of Change from Baseline in PROFAD SSI SF Subscores | Summarize for the 3 subscores (PROF, PROFAD, SSI) Footnote (if feasible): 1. PROF is calculated as the sum of domains Somatic fatigue and Mental fatigue 2. PROFAD is calculated as the sum of domains Somatic fatigue, Mental fatigue, Arthralgia and Vascular 3. SSI is calculated as the sum of domains Cutaneous dryness, Vaginal dryness, Ocular dryness and Oral dryness. The SSI subscore is derived for females only. | SAC_WK52 [2] |
| PtGA | | | | | |
| 6.9. | Safety | EFF_T1 | Summary Statistics of PtGA | | SAC_WK52 [2] |
| 6.10. | Safety | EFF_T1 | Summary Statistics of Change from Baseline: PtGA | | SAC_WK52 [2] |
| Further Health | Outcomes Ana | alyses | | | |
| 6.11. | Safety | EFF_T11 | Summary of Bayesian Posterior Probabilities: ESSPRI Total Score | To be generated by GSK Add appropriate footnotes based on final output | SAC_WK52 [2] |

| Health Outcomes: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.14. (6.1014) | Safety | EFF_T4 | Summary of ESSPRI Responders | EoS: Include all scheduled visits Footnote: Responder 1: Decrease in the ESSPRI total score of at least one point or at least 15% compared to baseline Responder 2: Subjects with baseline score of >= 5 and Total ESSPRI score of < 5. The denominator for percentages at each visit are the subjects who had a score >= 5 at baseline. | SAC_WK52 [2]<br>SAC_EOS [3] |
| (6.1015) | Completer | EFF_T1 | Summary Statistics of ESSPRI Total Score and Domains – Completer | Include all scheduled visits Summarize for both the overall score and 3 domains (dryness, fatigue and pain) Add footnote: Note: Completer is defined as "Subjects who completed the 52 Week treatment visits AND general follow up phase of the study including the visit at Week 68" | SAC_EOS [3] |

2020N437857\_00 201842

## 11.13.13. Health Outcomes Figures

| Health Outcomes: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ESSPRI Score | | | | | |
| 6.1. (6.1001) | Safety | EFF_F1 | Mean (+/-± SE) of Change from Baseline of ESSPRI<br>Total Score and Domains | EoS: As F2.1 Intervals with compose of arithmetic mean ± SE. All visits. Legend: Treatment | SAC_WK52 [2]<br>SAC_EOS [3] |
| 6.2. (6.1002) | Safety | EFF_F3 | Proportion of Subjects with an ESSPRI Response | EoS: Include all scheduled visits Footnote: Responder 1: Decrease in the ESSPRI total score of at least one point or at least 15% compared to baseline Responder 2: Subjects with baseline score of ≥ 5 and Total ESSPRI score of < 5 at each visit. The denominator for percentages are the subjects who had a score >=5 at baseline at each visit. | SAC_WK52 [2]<br>SAC_EOS [3] |
| PROFAD SSI SI | | | | | |
| 6.3. | Safety | EFF_F1 | Mean (+/-± SE) of Change from Baseline PROFAD SSI SF Subscores | Parameter by: Subscores Intervals with compose of arithmetic mean ± SE. All visits. Legend: Treatment | SAC_WK52 [2] |

2020N437857\_00 201842

## 11.13.14. Exploratory Tables

| Exploratory: Tabl | Exploratory: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Ocular Dryness | | | | | |
| 7.1. (7.1001) | Safety | EFF_T1 | Summary Statistics of Ocular Dryness Score | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.2. (7.1002) | Safety | EFF_T1 | Summary Statistics of Change from Baseline:<br>Ocular Dryness Score | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| Lacrimal Gland F | unction | | | | |
| 7.3. | Safety | EFF_T1 | Summary Statistics: Lacrimal Gland Function (Schirmer's test) | Page by: Laterality Parameter: Strip length wet (mm/min) Footnote: Note: Unit = mm/min | SAC_WK52 [2] |
| 7.4. | Safety | EFF_T1 | Summary Statistics of Change from Baseline:<br>Lacrimal Gland Function (Schirmer's test) | Page by: Laterality Parameter: Strip length wet (mm/min) Footnote: Note: Unit = mm/min | SAC_WK52 [2] |
| PGA | | | | | |
| 7.5. | Safety | EFF_T1 | Summary Statistics of PGA | | SAC_WK52 [2] |
| 7.6. | Safety | EFF_T1 | Summary Statistics of Change from Baseline: PGA | | SAC_WK52 [2] |

| Exploratory: Tabl | Exploratory: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Serologic Marker | s | | | | |
| 7.7. (7.1007) | Safety | EFF_T1 | Summary Statistics of Serologic Markers | Page by marker Include all visits up to Week 68 EoS: Include all scheduled visits Lambda and Kappa Light Chains Ratio of Kappa / Lambda Beta 2 Microglobulin Rheumatoid Factor | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.8. (7.1008) | Safety | EFF_T9 | Summary Statistics Percentage Change from Baseline: Serologic Markers | Page by marker Include all visits up to Week 68 EoS: Include all scheduled visits Ratio of Kappa /Lambda Light Chains Beta 2 Microglobulin Rheumatoid Factor | SAC_WK52 [2]<br>SAC_EOS [3] |
| Flow Cytometry F | Parameters | | | | |
| 7.9. (7.1009) | Safety | EFF_T9 | Summary Statistics of Flow Cytometry Flow Parameters | Include all parameters specified in RAP Table 11 except for: Plasmablasts (CD38br CD27br CD20+) Plasmacells CD20+ (CD20+ CD138+) Short-lived Plasma (CD20- CD27br) Transitional (CD24+ CD27-) Naïve B cells (CD24-CD38br+) B cells CD20+ (CD19+CD20+) | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.10. (7.1010) | Safety | EFF_T9 | Summary Statistics of Percentage Change from Baseline: Flow Cytometry Parameters | Include all parameters specified in RAP Table 11 for the Final Analysis except for: Plasmablasts (CD38br CD27br CD20+) | HL [1] SAC_WK52 [2]<br>SAC_EOS [3] |

| Exploratory: Tabl | Exploratory: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| | | | | Plasmacells CD20+ (CD20+ CD138+) Short-lived Plasma (CD20- CD27br) Transitional (CD24+ CD27-) Naïve B cells (CD24-CD38br+) B cells CD20+ (CD19+CD20+) | |
| 7.11. (7.1011) | Safety | EFF_T10 | Summary of Statistical Analysis Results of Percentage Change from Baseline in: Flow Cytometry Parameters at Week 24 EOS: Summary of Statistical Analysis Results of Change from Baseline in: Flow Cytometry Parameters at Week 24 | Include only the below parameters for analysis CD19+ B cell (CD3-CD19+) Naïve B cell (CD19+CD20+CD27-) Memory B cell (CD19+CD20+CD27+) Activated B Cell (CD20+ CD69+) Plasmablast All (CD19+CD27+CD38+) Plasmablast (CD20+) Plasmablast (CD20-) Transitional B cells (CD19+CD24bCD38+CD27-) Footnote: Analysis performed using Hodges-Lehmann estimator based on Wilcoxon rank test for 2 sample populations. | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.12. | Per<br>Protocol | EFF_T10 | Summary of Statistical Analysis Results of Percentage Change from Baseline in: Flow Cytometry Parameters at Week 24 | Include only the below parameters for analysis CD19+ B cell (CD3-CD19+) Naïve B cell (CD19+CD20+CD27-) Memory B cell (CD19+CD20+CD27+) Activated B Cell (CD20+CD69+) Plasmablast All | SAC_WK52 [2] |

| xploratory: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 7.13.<br>(7.1013) | Safety | Example Shell EFF_T10 | Summary of Statistical Analysis Results of Percentage Change from Baseline in: Flow Cytometry Parameters at Week 52 EoS Summary of Statistical Analysis Results of Change from Baseline in: Flow Cytometry Parameters at Week 52 | (CD19+CD27+CD38+) Plasmablast (CD20+) Plasmablast (CD20-) Transitional B cells (CD19+CD24bCD38+CD27-) Footnote: Analysis performed using Hodges-Lehmann estimator based on Wilcoxon rank test for 2 sample populations. Include only the below parameters for analysis CD19+ B cell (CD3-CD19+) Naïve B cell (CD19+CD20+CD27-) Memory B cell (CD19+CD20+CD27+) Activated B Cell (CD20+CD69+) Plasmablast All (CD19+CD27+CD38+) Transitional B cells (CD19+CD24bCD38+CD27-) Plasmablast (CD20+) | SAC_WK52 [2]<br>SAC_EOS [3] |
| | | | | Plasmablast (CD20-) Footnote: Analysis performed using Hodges-Lehmann estimator based on Wilcoxon rank test for 2 sample populations. | |

| Exploratory: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| BLyS | | | | | |
| 7.14. (7.1014) | Safety | EFF_T9 | Summary Statistics of Free BLyS Levels in Blood EoS: Summary Statistics of Free and Total BLyS Levels in Blood | EoS: Include all scheduled visits Subset BICATCD = "TNF13BPF" | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.15. (7.1015) | Safety | EFF_T9 | Summary Statistics of Percentage Change from Baseline: Free BLyS Levels in Blood EoS: Summary Statistics of Free and Total BLyS Levels in Blood | EoS: Include all scheduled visits Subset BICATCD = "TNF13BPF" | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.16. (7.1016) | Per<br>Protocol | EFF_T9 | Summary Statistics of Percentage Change from<br>Baseline: Free BLyS Levels in Blood<br>EoS<br>Summary Statistics of Free and Total BLyS<br>Levels in Blood | EoS: Include all scheduled visits Subset BICATCD = "TNF13BPF" | SAC_WK52 [2]<br>SAC_EOS [3] |
| Complement Fact | ors | | | | |
| 7.17. (7.1017) | Safety | EFF_T9 | Summary Statistics of Complement Factors | EoS: Include all scheduled visits To be run on C3, C4 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.18. (7.1018) | Safety | EFF_T9 | Summary Statistics of Percentage Change from Baseline: Complement Factors | EoS: Include all scheduled visits To be run on C3, C4 Note: For SAC_EOS [3] - Include protocol defined Serological biomarkers | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.19. (7.1019) | Safety | PD_T1 | Summary of CH50 by Visit | Frequency count | SAC_WK52 [2] |

| Exploratory: Tabl | Exploratory: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| | | | | | SAC_EOS [3] |
| Serum Cytokines | and Chemoki | nes | | | |
| 7.20. (7.1020) | Safety | EFF_T9 | Summary Statistics of Serum Cytokines and Chemokines | EoS: Include all scheduled visits CXCL13 NOTE: BICATCD=BLC = BICAT = B- lymphocyte chemokine Add footnote: Note: B-lymphocyte Chemokine = CXCL13 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7.21. (7.1021) | Safety | EFF_T9 | Summary Statistics of Percentage Change from Baseline: Serum Cytokines and Chemokines | EoS: Include all scheduled visits CXCL13 NOTE: BICATCD=BLC = BICAT = B- lymphocyte chemokine Add footnote: Note: B-lymphocyte Chemokine = CXCL13 | SAC_WK52 [2]<br>SAC_EOS [3] |

| Exploratory: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| SS-A and SS-B | • | | | | |
| 7.22. (7.1022) | Safety | PD_T2 | Summary of Autoantibodies by Visit | EoS: Include all scheduled visits Frequency count of SS-A and SS-B at final | SAC_WK52 [2]<br>SAC_EOS [3] |
| Further Evaluatio | n | | | | |
| (7.1023) | Completer | EFF_T9 | Summary Statistics of Flow Cytometry Flow Parameters – Completer | Include all parameters specified in RAP Table 11 except for: Plasmablasts (CD38br CD27br CD20+) Plasmacells CD20+ (CD20+ CD138+) Short-lived Plasma (CD20- CD27br) Transitional (CD24+ CD27-) Naïve B cells (CD24-CD38br+) B cells CD20+ (CD19+CD20+) Add footnote: Note: Completer is defined as "Subjects who completed the 52 Week treatment visits AND general follow up phase of the study including the visit at Week 68" | SAC_EOS [3] |

2020N437857\_00 201842

# 11.13.15. Exploratory Figures

| Exploratory: Fi | igures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Ocular Drynes | s NRS | , | | | |
| 7.1. (7.1001) | Safety | EFF_F1 | Mean (+/- SE) of Change from Baseline in Ocular Dryness NRS | All scheduled visits<br>Legend: Treatment<br>EoS: As F2.1001 | SAC_WK52 [2]<br>SAC_EOS [3] |
| Lacrimal Gland | f Function | | | | |
| 7.2. | Safety | EFF_F1 | Mean (+/- SE) of Change from Baseline in Lacrimal Gland Function (Schirmers Test) | All scheduled visits<br>Legend: Treatment<br>EoS: As F2.1001 | SAC_WK52 [2] |
| PGA | | | | | |
| 7.3. | Safety | EFF_F1 | Mean (+/- SE) of Change from Baseline in PGA | All scheduled visits<br>Legend: Treatment | SAC_WK52 [2] |
| Flow Cytometr | у | | | - | |
| 7.4. (7.1004) | Safety | EFF_F4 | Median (+/- IQR) of Absolute Values of Flow<br>Cytometry | EoS: As F2.1001 Include only the following parameters (Page by) CD19+ B cell (CD3-CD19+) Naïve B cell (CD19+CD20+CD27-) Memory B cell (CD19+CD20+CD27+) Activated B Cell (CD20+CD69+) Plasmablast All (CD19+CD27+CD38+) Transitional B cells (CD19+CD27+CD38+) Transitional B cells (CD19+CD27-) Plasmablast CD20+ Plasmablast CD20- x-axis is visit, y-axis in absolute values of the parameters. Panel per treatment group. | SAC_WK52 [2]<br>SAC_EOS [3] |

| Exploratory: Fi | | IDOL / TOT ID / | T:0 | | D |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 7.5. (7.1005) | Safety | EFF_F4 | Median (+/- IQR) for Percentage Change from Baseline in Flow Cytometry | EoS: As F2.1001 CD19+ B cell (CD3-CD19+) Naïve B cell (CD19+CD20+CD27-) Memory B cell (CD19+CD20+CD27+) Activated B Cell (CD20+CD69+) Plasmablast All (CD19+CD27+CD38+) Transitional B cells (CD19+CD24bCD38+CD27-) Plasmablast CD20+ Plasmablast CD20- x-axis is visit, y-axis in percentage change from baseline of the parameters. Panel per treatment group. | SAC_WK52 [2]<br>SAC_EOS [3] |
| Blys | | | | | |
| 7.6. (7.1006) | Safety | EFF_F4 | Median (+/- IQR) for Percentage Change from<br>Baseline in Free Blys<br>EoS<br>Median (+/- IQR) for Percentage Change from<br>Baseline in Free and Total Blys | EoS: EoS: As F2.1001 x-axis is visit, panel by parameter (Free & Total BLyS). | SAC_WK52 [2]<br>SAC_EOS [3] |
| Serologic Biom | narkers | | | | |
| 7.7. (7.1007) | Safety | EFF_F4 | Median (+/- IQR) for Percentage Change from Baseline in Serological Biomarkers | EoS: EoS: As F2.1001 Include Rheumatoid Factor, Lambda light chain protein, Kappa light chain protein, Kappa/Lambda ratio, Beta 2 microglobulin | SAC_WK52 [2]<br>SAC_EOS [3] |
| Complement Fa | actors | | | | |
| 7.8. (7.1008) | Safety | EFF_F4 | Median (+/- IQR) for Percentage Change from Baseline in Complement Factors | EoS: EoS: As F2.1001<br>Include C3 and C4 | SAC_WK52 [2]<br>SAC_EOS [3] |

| Exploratory: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Serum Chemol | kines | | | | |
| 7.9. (7.1009) | Safety | EFF_F4 | Median (+/- IQR) for Percentage Change from Baseline in CXCL13 | EoS: EoS: As F2.1001 NOTE: BICATCD=BLC = BICAT = B- lymphocyte chemokine | SAC_WK52 [2]<br>SAC_EOS [3] |

2020N437857\_00 201842

## 11.13.16. ICH Listings

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study Populati | on | | | | |
| 1. | Safety | TA1 | Listing of Randomized and Actual Treatments | | SAC_WK52 [2] |
| 2. (1002) | Safety | ES2 | Listing of Reasons for Study Withdrawal | | SAC_WK52 [2]<br>SAC_EOS [3] |
| 3. | Safety | POP_L1 | Listing of Reasons for Permanent Study Treatment Discontinuation | | SAC_WK52 [2] |
| 4. | Screened | ES7 | Listing of Reasons for Screening Failure | | SAC_WK52 [2] |
| 5. (1005) | Safety | SP3 | Listing of Subjects Excluded from Any Populations | | SAC_WK52 [2]<br>SAC_EOS [3] |
| 6. (1006) | Safety | DV2 | Listing of Important Protocol Deviations | | SAC_WK52 [2]<br>SAC_EOS [3] |
| 7. | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC_WK52 [2] |
| Demographics | | | | | |
| 8. | Safety | DM2 | Listing of Demographic Characteristics | | SAC_WK52 [2] |
| 9. | Safety | DM9 | Listing of Race | | SAC_WK52 [2] |
| 10. (1010) | Safety | POP_L2 | Listing of Physical Exam | | SAC_WK52 [2]<br>SAC_EOS [3] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Medical Condit | ion & Concomitant | Medications | | | |
| 11. | Safety | MH2 | Listing of Medical Conditions (Sjögren specific) | iSRC version has all medical conditions | SAC_WK52 [2] |
| 12. | Safety | MH2 | Listing of Medical Conditions (non-Sjögren specific) | | SAC_WK52 [2] |
| 13. (1013) | Safety | CP_CM3 | Listing of Concomitant Medications | | SAC_WK52 [2]<br>SAC_EOS [3] |
| Disease Histor | у | | | | |
| 14. | Safety | POP_L3 | Listing of Disease Characteristics (AECG Criteria) | | SAC_WK52 [2] |
| Exposure | | | | | |
| 15. | Safety | OEX3a | Listing of Exposure | | SAC_WK52 [2] |
| Adverse Event | S | | | | |
| 16. (1016) | Safety | AE7 | Listings of Subject Numbers for Individual Adverse Events | EoS: Include visits upto W68/FU EoS Footnote: Note: Includes Treatment & General Follow Up periods only. | SAC_WK52 [2]<br>SAC_EOS [3] |
| 17. (1017) | Safety | AE8 | Listing of All Adverse Events | EoS: Include visits upto W68/FU EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 18. (1018) | Safety | AE8 | Listing of Post Treatment Adverse Events | EoS: Include visits upto W68/FU EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 19. (1019) | Safety | SAFE_L3 | Listing of Adverse Events of Special Interest | EoS: Include visits upto W68/FU EoS Footnote: As Listing 1016 Include all AESI, including study specific | SAC_WK52 [2]<br>SAC_EOS [3] |
| 20. (1020) | Safety | AE8 | Listing of Fatal Serious Adverse Events | EoS: Include visits upto W68/FU EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 21. (1021) | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | EoS: Include visits upto W68/FU EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 22. (1022) | Safety | AE14 | Listing of Reasons for Considering as a Serious<br>Adverse Event | EoS: Include visits upto W68/FU EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 23. (1023) | Safety | AE8 | Listing of Adverse Events Leading to Discontinuation of Treatment or Withdrawal from Study | EoS: Include visits upto W68/FU EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 24. (1024) | Safety | AE2 | Listing of Relationship between System Organ<br>Class and Verbatim Text | EoS: Include visits upto W68/FU EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laboratory | | | | | |
| 25. (1025) | Safety | LB5 | Listing of Hematology Laboratory Data | EoS: Include all scheduled visits EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 26. (1026) | Safety | LB5 | Listing of Clinical Chemistry Laboratory Data | EoS: Include all scheduled visits EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 27. (1027) | Safety | LB5 | Listing of Liver Function Laboratory Data | EoS: Include all scheduled visits EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 28. (1028) | Safety | UR2a | Listing of Urinalysis Data | EoS: Include all scheduled visits EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 29. (1029) | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | EoS: Include all scheduled visits EoS Footnote: As Listing 1016 | SAC_WK52 [2]<br>SAC_EOS [3] |
| Vital Signs | | | | | • |
| 30. (1030) | Safety | VS4 | Listing of Vital Signs | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| ECGs | | | | | |
| 31. | Safety | EG5 | Listing of Abnormal ECG Findings | | SAC_WK52 [2] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Other | | | | | |
| (1061) | Safety | DV2 | Listing of Protocol Deviations Related to Covid-19 | Include only subjects with related Covid-19 PD's. Subset standard text 'COVID-19'. | SAC_EOS [3] |

2020N437857\_00 201842

# 11.13.17. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | | | | | |
| 32. (1032) | Safety | SAFE_L1 | Listing of Neurological Symptoms | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 33. (1033) | Safety | ECSSRS4 | Listing of C-SSRS Suicidal Ideation and Behavior Data | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 34. (1034) | Safety | ECSSRS5 | Listing of C-SSRS Suicidal Behavior Details | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 35. (1035) | Safety | SAFE_L2 | Grade 3 or Grade 4 Laboratory Toxicity Results: Hematology | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 36. (1036) | Safety | SAFE_L2 | Grade 3 or Grade 4 Laboratory Toxicity Results:<br>Clinical Chemistry | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| 37. (1037) | Safety | SAFE_L2 | Grade 3 or Grade 4 Laboratory Toxicity Results: Immunoglobulin | EoS: Include all scheduled visits IgG only | SAC_WK52 [2]<br>SAC_EOS [3] |
| 38. | Safety | SAFE_L4 | Listing of Positive Results for Other Screening<br>Tests | Include HIV, Hepatitis B (HBsAg), HbcAb, Hepatitis C (Hep C antibody), FSH, estradiol and serum or urine hCG pregnancy test. | SAC_WK52 [2] |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 39. (1039) | Safety | IMM2 | Listing of Positive Immunogenicity Results | Primary Belimumab EoS Belimumab & Rituximab Results All antibody and assay data Footnote: For anti-Rituximab, baseline is Week 8 | SAC_WK52 [2]<br>SAC_EOS [3] |
| 40. (1040) | Safety | LB5 | Listing of Immunoglobulins | Define flags "I" "N" "U" etc in the footnotes | SAC_WK52 [2]<br>SAC_EOS [3] |
| 41. (1041) | Safety | LB5 | Listing of CD4 and CD8 | EoS: Include all scheduled visits | SAC_WK52 [2]<br>SAC_EOS [3] |
| Efficacy | | | | | |
| 42. (1042) | Safety | EFF_L1 | Listing of ESSDAI Responses | EoS: Include all scheduled visits At SAC Include Total ESSDAI, ClinESSDAI and individual domains | SAC_WK52 [2]<br>SAC_EOS [3] |
| 43. (1043) | Safety | EFF_L2 | Listing of Damage Scoring for Subjects with Damage | EoS: Include all scheduled visits For each subject with damage. All timepoints, but only in domain which has any damage reported. | SAC_WK52 [2]<br>SAC_EOS [3] |
| 44. (1044) | Safety | EFF_L3 | Listing of Change from Baseline of Clinical Efficacy Endpoints and Number of B cells (CD20/mm2) in salivary gland. | EoS: Include all scheduled visits To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 45. (1045) | Safety | EFF_L4 | Listing of Stimulated and Unstimulated Salivary Flow | EoS: Include all scheduled visits To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |
| 46. (1046) | Safety | EFF_L5 | Listing of Oral and Ocular Dryness NRS | EoS: Include all scheduled visits To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |
| 47. | Safety | EFF_L6 | Listing of Lacrimal Function (Schirmer's) Test | To be generated by GSK | SAC_WK52 [2] |
| 48. | Safety | EFF_L7 | Listing of PROFAD-SSI-SF Subscores | To be generated by GSK | SAC_WK52 [2] |
| 49. | Safety | EFF_L8 | Listing of Patient Global Assessment (PtGA) | To be generated by GSK | SAC_WK52 [2] |
| 50. | Safety | EFF_L9 | Listing of Physicians Global Assessment (PGA) | To be generated by GSK | SAC_WK52 [2] |
| 51. (1051) | Safety | EFF_L10 | Listing of Free and Total BLyS Levels | EoS: Include all scheduled visits To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |
| 52. (1052) | Safety | EFF_L11 | Listing of Flow Cytometry Parameters | EoS: Include all scheduled visits Include all parameters Page by: Parameters To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |
| 53. (1053) | Safety | EFF_L11 | Listing of Serologic Markers | EoS: Include all scheduled visits Include all parameters Page by: Parameters To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID<br>/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 54. | Safety | EFF_L11 | Listing of Salivary Gland Assessment | Include all parameters Page by: Parameters To be generated by GSK | SAC_WK52 [2] |
| 55. (1056) | Safety | EFF_L12 | Listing of ESSPRI Score | EoS: Include all scheduled visits To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |
| 541 (1057) | Safety | EFF_L11 | Listing of Complement Factors (CH50) | EoS: Include all scheduled visits To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |
| 542 (1058) | Safety | EFF_L11 | Listing of Complement Factors (Biomarkers) | EoS: Include all scheduled visits To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |
| 1059. | Safety | POP_L4 | Listing of Overall Subject Status | EoS: Include all scheduled visits To be generated by GSK | SAC_EOS [3] |
| 411 (1411) | Safety | SAFE_L4 | Listing of All Adverse Events Post Week 68 during the Individualized Follow Up Period | Primary: Blinded listing EoS: Unblinded listing To be generated by GSK | SAC_WK52 [2]<br>SAC_EOS [3] |

201842 | Statistical Analysis Plan EoS RAP 15 Sep 2020 | TMF-2108787 | 4.0

CONFIDENTIAL

2020N437857\_00 201842

### 11.14. Appendix 14: Example Mock Ups

Data Display Specification are presented in a separate document.